| Official Protocol Title: | A Phase III Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-1439A Once-Daily Versus ATRIPLA <sup>TM</sup> Once-Daily in Treatment-Naïve HIV-1 Infected Subjects |
|---|---|
| NCT number: | NCT02403674 |
| <b>Document Date:</b> | 02-Nov-2022 |

**Protocol/Amendment No.:** 021-09

THIS PROTOCOL AMENDMENT AND ALL OF THE INFORMATION RELATING TO IT ARE CONFIDENTIAL AND PROPRIETARY PROPERTY OF MERCK SHARP & DOHME LLC, RAHWAY, NJ, USA (MSD).

This protocol amendment is applicable only to Colombia, Guatemala, Honduras, Mexico, Peru, Australia, New Zealand, Russia, South Africa, Thailand, Portugal, Spain.

#### **SPONSOR:**

Merck Sharp & Dohme LLC (hereafter referred to as the Sponsor or MSD) 126 East Lincoln Avenue P.O. Box 2000 Rahway, NJ 07065 USA

Protocol-specific Sponsor Contact information can be found in the Investigator Trial File Binder (or equivalent).

#### TITLE:

A Phase III Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-1439A Once-Daily Versus ATRIPLA<sup>TM</sup> Once-Daily in Treatment-Naïve HIV-1 Infected Subjects

**IND NUMBER:** 124997

**EudraCT NUMBER: 2014-003382-17** 

**Protocol/Amendment No.:** 021-09

## **TABLE OF CONTENTS**

| DOCU | ME | NT I | HISTORY | 10 |
|---|---|---|---|---|
| SUMN | IAR | Y Ol | F CHANGES | 15 |
| 1.0 | TRI | IAL S | SUMMARY | 16 |
| 2.0 | TRI | | DESIGN | <b>17</b> |
| 2.1 | T | rial ] | Design | <b>17</b> |
| 2.2 | T | rial ] | Diagram | 19 |
| 3.0 | OB | JEC. | ΓΙVE(S) & HYPOTHESIS(ES) | <b>21</b> |
| 3.1 | P | rima | ry Objective(s) & Hypothesis(es) | <b>21</b> |
| 3. | 1.1 | Base | e Study | 21 |
| 3.2 | S | econ | dary Objective(s) & Hypothesis(es) | <b>22</b> |
| 3.2 | 2.1 | Base | e Study | 22 |
| 3.3 | E | xplo | ratory Objectives | <b>24</b> |
| 3 | 3.1 | Base | e Study | 24 |
| 3 | 3.2 | Stuc | ly Extension 1 | 24 |
| 4.0 | BAG | CKG | ROUND & RATIONALE | 24 |
| 4.1 | В | ackg | ground | 24 |
| 4. | 1.1 | Pha | rmaceutical and Therapeutic Background | 24 |
| 4.2 | R | atio | nale | <b>26</b> |
| 4.2 | 2.1 | Rati | onale for the Trial and Selected Subject Population | 26 |
| 4.2 | 2.2 | Rati | onale for Dose Selection/Regimen | 26 |
| 4.2 | 2.3 | Rati | onale for Endpoints | 28 |
| | 4.2. | 3.1 | Efficacy Endpoints | 28 |
| | 4.2.3 | 3.2 | Safety Endpoints | 29 |
| | 4.2.3 | 3.3 | Pharmacokinetic Endpoints | 30 |
| | 4.2.3 | 3.4 | Patient-Reported Outcome Endpoints | 30 |
| | 4.2. | 3.5 | Planned Exploratory Biomarker | 30 |
| | 4.2.3 | 3.6 | Future Biomedical Research | 31 |
| 4.2 | 2.4 | Rati | onale for Study Extensions. | 31 |
| 4.3 | В | enef | it/Risk | 31 |

| 5.0 | M | ETHODOL | OGY | 32 |
|---|---|---|---|---|
| 5. | 1 | <b>Entry Crite</b> | ria | 32 |
| | 5.1.1 | Diagnosis | /Condition for Entry into the Trial | 32 |
| | 5.1.2 | Subject In | clusion Criteria | 32 |
| | 5.1.3 | Subject Ex | xclusion Criteria | 36 |
| 5.2 | 2 | Trial Treati | ment(s) | 37 |
| | 5.2.1 | Dose Sele | ction | 38 |
| | 5.2 | 2.1.1 Dose | Selection (Preparation) | 38 |
| | 5.2 | 2.1.2 Dose | Modification/Interruption (Base Study or the Study Extensions) | 39 |
| | 5.2.2 | Timing of | Dose Administration | 39 |
| | 5.2 | 2.2.1 Base | Study | 39 |
| | 5.2 | 2.2.2 Study | Extensions | 39 |
| | 5.2.3 | Trial Blin | ding/Masking | 40 |
| 5 | 3 | Randomiza | tion or Treatment Allocation | 40 |
| 5.4 | 4 | Stratificatio | n | 40 |
| 5. | 5 | Concomitar | t Medications/Vaccinations (Allowed & Prohibited) | 41 |
| 5.0 | 6 | Rescue Med | lications & Supportive Care | 44 |
| 5. | 7 | Diet/Activit | y/Other Considerations | 44 |
| 5. | 8 | Subject Wit | hdrawal/Discontinuation Criteria | 44 |
| 5.9 | 9 | Subject Rep | lacement Strategy | 46 |
| 5. | 10 | Beginning a | nd End of the Trial | 46 |
| 5. | 11 | Clinical Cri | teria for Early Trial Termination | 47 |
| 6.0 | TI | RIAL FLOV | V CHART | 48 |
| 7.0 | TI | RIAL PROC | CEDURES | 55 |
| 7. | 1 | Trial Proce | dures | 55 |
| | 7.1.1 | Administr | ative Procedures | 55 |
| | 7. | .1.1 Inform | ned Consent | 55 |
| | | 7.1.1.1.1 C | Seneral Informed Consent | 55 |
| | | | Consent and Collection of Specimens for Future Biomedical desearch | |
| | 7.1 | .1.2 Inclus | sion/Exclusion Criteria | 56 |
| | 7.1 | .1.3 Subje | ct Identification Card | 56 |

| 7.1.1.4 | Medical History | 56 |
|---|---|---|
| 7.1.1.5 | Prior and Concomitant Medications Review | 56 |
| 7.1.1. | 5.1 Prior Medications | 56 |
| 7.1.1. | 5.2 Concomitant Medications | 57 |
| 7.1.1.6 | Assignment of Screening Number | 57 |
| 7.1.1.7 | Assignment of Randomization Number | 57 |
| 7.1.1.8 | Trial Compliance (Medication/Diet/Activity/Other) | 57 |
| 7.1.1.9 | Patient-Reported Outcomes | 58 |
| 7.1.2 Cli | nical Procedures/Assessments | 58 |
| 7.1.2.1 | Physical Examination | 58 |
| 7.1.2.2 | Height Assessment | 59 |
| 7.1.2.3 | Vital Signs and Weight | 59 |
| 7.1.2.4 | 12-Lead ECG (performed locally) | 59 |
| 7.1.2.5 | Adverse Events | 60 |
| 7.1.2.6 | Toxicity Management | 60 |
| 7.1.2.7 | Birth Control Confirmation. | 60 |
| 7.1.3 Lat | poratory Procedures/Assessments | 61 |
| 7.1.3.1 | Serum /Urine Pregnancy Test | 61 |
| 7.1.3.2 | Laboratory Safety Evaluations (Hematology, Chemistry and Others) | 61 |
| 7.1.3.3 | HIV/ Hepatitis Screening | 62 |
| 7.1.3.4 | Virology Test | 62 |
| 7.1.3.5 | Viral Resistance Testing | 62 |
| 7.1.3.6 | CD4 Cell Counts | 63 |
| 7.1.3.7 | Pharmacokinetic/Pharmacodynamic Evaluations | 63 |
| 7.1.3.8 | Future Biomedical Research | 64 |
| 7.1.4 Oth | ner Procedures | 64 |
| 7.1.4.1 | Withdrawal/Discontinuation | 64 |
| 7.1.4. | 1.1 Withdrawal From Future Biomedical Research | 64 |
| 7.1.4.2 | Blinding/Unblinding | 65 |
| 7.1.4.3 | Calibration of Equipment. | 66 |
| 7.1.5 Vis | it Requirements | 66 |
| 7.1.5.1 | Screening | 66 |

| 7.1 | 1.5.2 | Treatment Visits in Base Study (Visit 2 to 12) | . 67 |
|---|---|---|---|
| 7.1 | 1.5.3 | Treatment Visits in Study Extension 1 (Visit 13 to Visit 19) | . 69 |
| 7.1 | 7.1.5.4 Treatment Visits in Study Extension 2 (Visit 20 to Visit 25) | | |
| 7.2 | 7.1.5.5 Treatment Visits in Study Extension 3 (Visit 26 to Visit 31) | | |
| 7.1 | 1.5.6 | Virologic Failure Confirmation Visit - Base Study and Study Extension 1 | |
| 7.1 | 1.5.7 | Early Discontinuation Visit - Base Study, Study Extension 1, Study Extension 2, and Study Extension 3 | |
| 7.1 | 1.5.8 | Post-Trial (Base Study and Study Extensions) | . 72 |
| 7.2 | Asses | sing and Recording Adverse Events | . 72 |
| 7.2.1 | | finition of an Overdose for This Protocol and Reporting of Overdose to Sponsor | . 73 |
| 7.2.2 | Rep | porting of Pregnancy and Lactation to the Sponsor | . 73 |
| 7.2.3 | Imr | mediate Reporting of Adverse Events to the Sponsor | . 74 |
| 7.2 | 2.3.1 | Serious Adverse Events | . 74 |
| 7.2 | 2.3.2 | Events of Clinical Interest | . 75 |
| 7.2.4 | Eva | aluating Adverse Events | . 75 |
| 7.2.5 | Spo | onsor Responsibility for Reporting Adverse Events | . 78 |
| 7.3 | TRIA | L GOVERNANCE AND OVERSIGHT | . 78 |
| 7.3.1 | Sci | entific Advisory Committee | . 78 |
| 7.3.2 | Exe | ecutive Oversight Committee | . 78 |
| 7.3.3 | Dat | a Monitoring Committee | . 78 |
| 8.0 ST | TATIS | STICAL ANALYSIS PLAN | <b>.</b> 79 |
| 8.1 | STAT | TISTICAL ANALYSIS PLAN SUMMARY | <b>.</b> 79 |
| 8.2 | Respo | onsibility for Analyses/In-House Blinding | . 82 |
| 8.3 | Нуро | theses/Estimation | . 83 |
| 8.4 | Analy | vsis Endpoints | . 84 |
| 8.4.1 | Eff | icacy /Pharmacokinetics Endpoints | . 84 |
| 8.4 | 4.1.1 | Efficacy Endpoints | . 84 |
| 8.4.2 | Saf | ety Endpoints | . 84 |
| 8.5 | Analy | sis Populations | . 86 |
| 8.5.1 | Eff | icacy Analysis Populations | . 86 |
| 8.5.2 | Saf | ety Analysis Populations | . 86 |

| 8.6 | Statistical Methods | 86 |
|---|---|---|
| 8.6 | 5.1 Statistical Methods for Efficacy Analyses | 87 |
| 8.6 | 5.2 Statistical Methods for Safety Analyses | 91 |
| 8.6 | 5.3 Summaries of Baseline Characteristics, Demographics, and Other Analyses | 94 |
| : | 8.6.3.1 Demographic and Baseline Characteristics | 94 |
| 8.7 | Interim Analyses | 94 |
| 8.8 | Multiplicity | 94 |
| 8.9 | SAMPLE SIZE AND POWER CALCULATIONS | 95 |
| 8.9 | 2.1 Sample Size and Power for Efficacy Analyses | 95 |
| 8.9 | 2.2 Sample Size and Power for Safety Analyses | 96 |
| 8.9 | 0.3 Overall Power | 98 |
| 8.10 | Subgroup Analyses and Effect of Baseline Factors (Base Study) | 99 |
| 8.11 | Compliance (Medication Adherence) | 99 |
| 8.12 | Extent of Exposure | 100 |
| | LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL | |
| | SUPPLIES | |
| 9.1 | Investigational Product | |
| 9.2 | Packaging and Labeling Information Clinical Supplies Disclosure | |
| 9.3<br>9.4 | Storage and Handling Requirements | |
| 9.4<br>9.5 | Returns and Reconciliation | |
| 9.6 | Standard Policies | |
| | ADMINISTRATIVE AND REGULATORY DETAILS | |
| 10.1 | Confidentiality | |
| | 1.1 Confidentiality of Data | |
| | 1.2 Confidentiality of Subject Records | |
| | 1.3 Confidentiality of Investigator Information | |
| | 1.4 Confidentiality of IRB/IEC Information | |
| 10.2 | Compliance with Financial Disclosure Requirements | |
| 10.2 | Compliance with Law, Audit and Debarment | |
| 10.3 | Compliance with Trial Registration and Results Posting Requirements | |
| 10.4 | Quality Management System | |
| | ~, | / |

| 10.6 | Data Management107 |
|---|---|
| 10.7 | Publications |
| 11.0 L | IST OF REFERENCES |
| 12.0 A | PPENDICES110 |
| 12.1 | Code of Conduct for Clinical Trials |
| 12.2 | Collection and Management of Specimens for Future Biomedical Research |
| 12.3 | Understanding the Intent, Scope and Public Health Benefits of Exploratory Biomarker Research: A Guide for IRBs/IECs and Investigational Site Staff |
| 12.4 | Approximate Blood Volumes Drawn/Collected by Trial Visit and by Sample Types |
| 12.4 | 1.1 Base Study |
| 12.4 | 4.2 Week 100 Through Week 192 Including Post-Study 14-Day Follow-up (Study Extension 1) |
| 12.5 | Plasma Assay—Sample Collection, Handling, Labeling, Storage, and Shipment |
| 12.6 | List of Preferred Neuropsychiatric Adverse Events |
| 12.7 | List of Abbreviations and Acronyms |
| 12.8 | DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS VERSION 1.0, DECEMBER, 2004; CLARIFICATION AUGUST 2009 |
| 13.0 S | IGNATURES |
| 13.1 | Sponsor's Representative |
| 13.2 | Investigator |

**Protocol/Amendment No.:** 021-09

### LIST OF TABLES

| Table 1 | Trial Treatment During the Base Study | 38 |
|---|---|---|
| Table 2 | Trial Treatment During the Study Extensions | |
| Table 3 | Stratification | |
| Table 4 | Laboratory Tests | 61 |
| Table 5 | Pharmacokinetic Sampling Timepoints | 64 |
| Table 6 | Study Drug Bottle (A and B) Components | 68 |
| Table 7 | Evaluating Adverse Events | 76 |
| Table 8 | Definition of Study Timepoint | 87 |
| Table 9 | Summary of the Two Approaches to Handle Missing Values | 89 |
| Table 10 | Analysis Strategy for Key Efficacy Variables | <mark>9</mark> 1 |
| Table 11 | Analysis Strategy for Safety Parameters | 93 |
| Table 12 | Power (%) Under Various Assumptions (With 340 Subjects Randomized | |
| | in Each Treatment Group) | 95 |
| Table 13 | Observed Percentage in MK-1439A Necessary to Demonstrate Superiority | |
| | versus ATRIPLA <sup>TM</sup> | 96 |
| Table 14 | Estimate of Incidence of AEs and 95% Upper Confidence Bound Based | |
| | on Hypothetical Numbers of Subjects with AEs Among 340 Subjects | |
| | Randomized in Each Treatment Group. | 97 |
| Table 15 | Differences in Incidences of AEs (MK-1439A q.d. minus ATRIPLA <sup>TM</sup> | |
| | q.d.) That Can Be Ruled Out With 340 Subjects in Each Treatment Group | 98 |
| Table 16 | Product Descriptions: Base Study and Study Extensions | . 101 |

**Protocol/Amendment No.:** 021-09

## LIST OF FIGURES

| Figure 1 | Trial Diagram Base Study | . 20 |
|----------|--------------------------------------------|------|
| Figure 2 | Trial Diagram Study Extensions 1, 2, and 3 | . 21 |

**Protocol/Amendment No.:** 021-09

### **DOCUMENT HISTORY**

| Document | Date of Issue | Overall Rationale |
|---|---|---|
| Amendment 09 | 02-NOV-2022 | This is a country-specific amendment for Colombia, Guatemala, Honduras, Mexico, Peru, Australia, New Zealand, Russia, South Africa, Thailand, Portugal, and Spain to inform regarding the Sponsor's name and address change and updates that were made to the Code of Conduct in the previous amendment. Note: Amendment 09 supersedes Amendment 08. |
| Amendment 08 | 23-AUG-2022 | Merck Sharp & Dohme Corp. underwent an entity name and address change to Merck Sharp & Dohme LLC, Rahway, NJ, USA. This conversion resulted only in an entity name change and update to the address. Note: Amendment 08 was not released to sites. |
| Amendment 07<br>(country-specific to Australia, Russia,<br>South Africa, New Zealand, Israel,<br>Columbia, Thailand, Peru, Honduras,<br>Guatemala) | 02-APR-2020 | • Study extension 3 was added to (1) provide continued access to MK-1439A for participants who are deriving benefit from MK-1439A until the drug is available locally in countries participating in the trial or for an additional 2 years (whichever comes first), and (2) collect key safety information from participants who continue on MK-1439A in this study extension. |

| Document | Date of Issue | Overall Rationale |
|---|---|---|
| Amendment 06<br>(country-specific to United States and<br>Puerto Rico) | 20-NOV-2018 | <ul> <li>Added 32 weeks past the Week 192 visit so that a subject may<br/>continue to receive MK-1439A during this time or until commercial<br/>MK-1439A is locally available (whichever occurs first).</li> </ul> |
| | | • Added 2 treatment visits in the Study Extension and updated blood volumes. |
| | | • Replaced the term HAART with cART. |
| | | • Added oxcarbazepine and rifapentine as prohibited medications/therapy due to interaction with MK-1439. |
| | | <ul> <li>Deleted herbal remedies from the list of prohibited medications.</li> </ul> |
| | | • Clarified that evaluation of IRIS causality applies only during the base study. |
| | | <ul> <li>Clarified emergency unblinding procedures.</li> </ul> |
| | | • Changed visit windows to correctly capture data pertinent to the specific milestones rather than specific study days. |

| Document | Date of Issue | Overall Rationale |
|---|---|---|
| Amendment 05 (applicable globally except for United States including Puerto Rico) | 26-NOV-2018 | • Added open-label study extension 2 to provide continued access to MK-1439A until the drug is available locally in countries participating in the trial or for an additional 2 years (whichever comes first). |
| | | Replaced the term HAART with cART. |
| | | • Added oxcarbazepine and rifapentine as prohibited medications/therapy due to interaction with MK-1439. |
| | | Deleted herbal remedies from the list of prohibited medications. |
| | | • Clarified that evaluation of IRIS causality applies only during the base study. |
| Amendment 04 (global) | 08-NOV-2016 | Added open-label study extension 1 for 2 years to collect long-term efficacy and safety data. |
| | | • Specified that concomitant medications prohibited due to interactions with EFV/FTC/TDF in the base study were allowed in the study extension. |
| | | • Clarified visits during which plasma samples were tested for resistance. |
| | | • Removed rosuvastatin as prohibited medication due to an interaction with DOR. |

| Document | Date of Issue | Overall Rationale |
|---|---|---|
| Amendment 03 (global) | 21-JUL-2015 | Added text to explain the rationale for the selected doses of the lamivudine and TDF components of MK-1439A. |
| | | • Added text to disallow concomitant use of interferon given that the occurrence of neuropsychiatric AEs associated with interferon use could confound the results of the trial. |
| | | • Added text to ensure consistency with the EFV/FTC/TDF, 3TC, and TDF prescribing information. |
| | | • Clarified that sites would receive the calculated creatinine clearance in the laboratory reports from the central laboratory. |
| Amendment 02 (global) | 21-MAY-2015 | Changed the pharmacokinetics/pharmacodynamics evaluation from an exploratory objective to a secondary objective. |
| | | • Added a baseline hemoglobin threshold (≥9.0 g/dL if female; ≥10.0 g/dL if male) to the Inclusion Criteria (#5). |
| | | • Added Exclusion Criterion #10 to exclude subjects with severe hepatic impairment. |
| | | • Updated list of medications prohibited during the use of ATRIPLA (EFV/FTC/TDF). |
| | | • Specified additional visits for the collection of plasma for potential viral resistance testing. |

| Document | Date of Issue | Overall Rationale |
|---|---|---|
| Amendment 01 (global) | 18-MAR-2015 | <ul> <li>Added instructions to the Inclusion Criteria directing investigators to provide appropriate guidance to subjects about the use of contraceptives after study completion.</li> <li>Modified Exclusion Criterion #4 to include the mutations D67N and K70R to those mutations indicative of resistance to emtricitabine, lamivudine, and tenofovir</li> </ul> |
| Original protocol | 14-JAN-2015 | Not applicable. |

**Protocol/Amendment No.:** 021-09

### **SUMMARY OF CHANGES**

# PRIMARY REASON(S) FOR THIS AMENDMENT:

| Section<br>Number (s) | Section Title(s) | Description of Change (s) | Rationale |
|---|---|---|---|
| | Title Page | Colombia, Guatemala, Honduras, Mexico, Peru, Australia, New Zealand, Russia, South Africa, Thailand, Portugal, and Spain were added to the Title Page. | This is a country-specific amendment for Colombia, Guatemala, Honduras, Mexico, Peru, Australia, New Zealand, Russia, South Africa, Thailand, Portugal, and Spain to inform regarding the Sponsor's name and address change and updates that were made to the Code of Conduct in the previous amendment. Note: Amendment 09 supersedes Amendment 08. |
| _ | _ | nent 08; however, Amendment 08 was not ron in the current country-specific amendment | <del>_</del> |
| 12.1<br>Throughout | Title Page Code of Conduct for Clinical Trials | Sponsor entity name and address change. | Merck Sharp & Dohme Corp. underwent an entity name and address change to Merck Sharp & Dohme LLC, Rahway, NJ, USA. This conversion resulted only in an entity name change and update to the address. |
| 12.1 | Code of Conduct for<br>Clinical Trials | The code of conduct was updated in Amendment 08. | To align with the current standard text for the code of conduct. |

# ADDITIONAL CHANGE(S) FOR THIS AMENDMENT:

No additional changes.

**Protocol/Amendment No.:** 021-09

## 1.0 TRIAL SUMMARY

| Abbreviated Title | MK-1439A versus ATRIPLA™ in treatment-naïve HIV-infected subjects. |
|---|---|
| Trial Phase | Phase 3 |
| Clinical Indication | Treatment of HIV-1 infection |
| Trial Type | Interventional |
| Type of control | Active control |
| Route of administration | Oral |
| Trial Blinding | Double-blind for the base study then open-label for the study extensions. |
| Treatment Groups | Base Study (double-blind) |
| | Group 1: MK-1439A q.d. MK-1439A is a single-tablet, fixed-dose regimen (FDR) containing MK-1439A 100 mg + lamivudine 300 mg + tenofovir disoproxil fumarate 300 mg. |
| | Group 2: ATRIPLA <sup>TM</sup> q.d. ATRIPLA <sup>TM</sup> is a single-tablet FDR containing efavirenz 600 mg + emtricitabine 200 mg + tenofovir disoproxil fumarate 300 mg (which is equivalent to 245 mg of tenofovir disoproxil). |
| | Study Extensions (open-label) |
| | All subjects participating in the extensions: MK-1439A q.d. |
| Number of trial subjects | Approximately 680 subjects will be enrolled. |
| Estimated duration of trial | The Sponsor estimates that the trial will require approximately 9 years from the time the first subject signs the informed consent until the last subject's last study-related phone call or visit. |
| Duration of Participation | The study consists of a screening phase of up to 45 days (~6.5 weeks) followed by a 96-week double-blind base study, 3 open-label study extensions (study extensions 1, 2, and 3), and a 14-day follow-up period. The treatment duration of study extension 1 is 96 weeks; and the treatment duration of study extensions 2 and 3 is up to 96 weeks for each, depending on when MK-1439A becomes commercially available once approved in the local country (whichever comes first). |
| | The approximate cumulative durations of participation in the trial (from informed consent through follow-up) are 104 weeks for subjects who complete the base study; 200 weeks for subjects who complete the base study and study extension 1; up to 296 weeks for subjects who complete the base study and study extensions 1 and 2; and up to 392 weeks for subjects who complete the base study and study extensions 1, 2, and 3. |
| Randomization Ratio | 1:1 with ~340 on MK-1439A and ~340 on ATRIPLA <sup>TM</sup> |

A list of abbreviations used in this document can be found in Section 12.7.

**Protocol/Amendment No.:** 021-09

#### 2.0 TRIAL DESIGN

#### 2.1 Trial Design

This is a multicenter, double-blind (with in-house blinding), randomized, active-controlled trial to evaluate the safety and efficacy of MK-1439A once-daily (q.d.) compared with ATRIPLA<sup>TM</sup> q.d. in antiretroviral treatment-naïve subjects with human immunodeficiency virus type 1 (HIV-1) infection.

MK-1439A is a single tablet FDR that combines MK-1439, an NNRTI, with 3TC and TDF, 2 approved and commercially available N(t)RTIs. As of the date of issuance of this protocol amendment, MK-1439A has been approved in multiple markets including the US, EU, Canada, Switzerland and Australia for the treatment of HIV-1 infection in adult patients.

A single tablet of MK-1439A contains a full daily HIV treatment regimen of MK-1439 100 mg + lamivudine 300 mg + TDF 300 mg. ATRIPLA<sup>TM</sup> is a single-tablet FDR that combines an approved and commercially available NNRTI, efavirenz, and 2 approved and commercially available NRTIs, FTC and TDF. A single tablet of ATRIPLA<sup>TM</sup> contains a full daily HIV treatment regimen of efavirenz 600 mg + FTC 200 mg + TDF 300 mg (which is equivalent to 245 mg of tenofovir disoproxil).

The study consists of a screening period of approximately 6.5 weeks, a 96-week blinded base study of MK-1439A compared with ATRIPLA<sup>TM</sup> followed by 3 consecutive open-label study extensions (study extensions 1, 2, and 3), and a 14-day post-study follow-up visit after the last treatment visit. The treatment duration of study extension 1 is 96 weeks; and the treatment duration of study extension 2 and study extension 3 is each up to 96 weeks, depending on when MK-1439A becomes commercially available once approved in the local country (whichever comes first).

The study is to be conducted in conformance with Good Clinical Practice.

Prior to enrolling in the base study and each of the study extensions, the subject must meet eligibility criteria (see Section 5.1.2) and provide consent.

Further detail for the base study and the 3 study extensions is provided below.

#### Base Study

Approximately 680 subjects will be stratified by screening HIV-1 ribonucleic acid (≤ or >100,000 copies/mL) and Hepatitis B and/or C co-infection status (yes/no) and randomized within strata in a 1:1 ratio to receive either MK-1439A or ATRIPLA™. The duration of treatment for a given subject is 96 weeks in the base study. The primary efficacy endpoint is the proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48. The primary safety endpoint is the proportion of subjects with certain neuropsychiatric adverse events by Week 48.

**Protocol/Amendment No.:** 021-09

The safety of the subjects in this trial will be monitored during the base study by an eDMC which will provide ongoing review of the safety data with suggested periodic reviews to occur approximately every 6 months. The eDMC will recommend steps to ensure the safety of study participants and the integrity of the trial. To guarantee the unrestricted performance of its task, the eDMC will receive study data from the unblinded statistician. Details regarding the eDMC will be described in a charter document.

Blood samples will be collected to support the evaluation of MK-1439 population PK from all subjects at Day 1 and Weeks 4, 8, 24 and 48.

Subjects will complete a WPAI at Day 1, and Weeks 4, 8, and 48 (or the early discontinuation visit). This patient-reported outcome questionnaire is designed to assess the quantitative impact of health conditions on loss of time and impaired productivity for functional activities such as work-for-pay, school work, and work around the house.

All subjects entering the study extensions will receive open-label treatment with MK-1439A (100 mg q.d.).

Treatment group assigned during the base study will not be unblinded when a subject enters study extension 1; unblinding will occur after all subjects have completed the base study and database lock has been achieved for the base study.

#### Study Extension 1

At Study Week 96, eligibility for enrollment into study extension 1 will be determined, thus continuing study treatment for approximately 96 weeks beyond the base study for subjects who meet eligibility criteria. The total duration of treatment for subjects who continue into study extension 1 is 192 weeks (approximately 4 years).

During study extension 1, subjects will continue to be monitored for safety and maintenance of virologic suppression. Long-term safety and efficacy data will be collected during study extension 1 and summarized descriptively.

#### Study Extension 2

At Study Week 192, eligibility for enrollment into study extension 2 will be determined. Subjects who meet eligibility criteria and continue into study extension 2 may continue to receive treatment with MK-1439A until it is commercially available once approved in the local country OR for an additional 96 weeks beyond study extension 1 (whichever comes first). The total duration of treatment for subjects who continue into study extension 2 is up to 288 weeks (up to approximately 2 years beyond extension 1, depending on when MK-1439A is commercially available once approved in the local country) (a total of approximately 5.5 years).

During study extension 2, pregnancy for female subjects and SAEs for all subjects will be monitored and collected. Efficacy data will not be collected for study extension 2.

Protocol/Amendment No.: 021-09

#### **Study Extension 3**

At Study Week 288, eligibility for enrollment into study extension 3 will be determined. Subjects who meet eligibility criteria and continue into study extension 3 may continue to receive treatment with MK-1439A until it is commercially available once approved in the local country OR for an additional 96 weeks beyond study extension 2 (whichever comes first). The total duration of treatment for subjects who continue into study extension 3 is 384 weeks (up to approximately 4 years beyond extension 1, depending on when MK-1439A is commercially available once approved in the local country) (a total of approximately 7.5 years).

During study extension 3, pregnancy for female subjects and SAEs for all subjects will be monitored and collected. Efficacy data will not be collected for study extension 3.

### Viral Resistance Testing

Subjects who meet virologic failure criteria during the base study and study extension 1 (see Section 4.2.3.1) will return to the site for repeat viral RNA testing between one week and 4 weeks (≥1 and ≤4 weeks) later (at a virologic failure confirmation visit). If virologic failure is confirmed and the viral load meets the criteria for resistance testing (>400 copies/mL), viral resistance testing will be performed. For subjects in the base study with confirmed virologic failures, the plasma sample collected for resistance testing from the virologic failure visit and the confirmation visit, will be sent for resistance testing provided the viral load meets the criteria for resistance testing.

For subjects in study extension 1 with confirmed virologic failure, the plasma sample from the virologic failure confirmation visit only will be sent for resistance testing provided the viral load meets the criteria for resistance testing.

Plasma samples for resistance testing collected at the early discontinuation visit from subjects who discontinue, from either the base study or study extension 1, for reasons other than virologic failure will be sent for testing (if viral load >400 copies/mL). Note that if a sample from the early discontinuation visit is not available, a sample from the most recent previous visit, if available, will be sent for testing in the base study (if viral load >400 copies/mL).

In addition, phenotypic testing will be conducted on screening samples for all subjects who discontinue for any reason or with confirmed virologic failure. See Section 7.1.3.5.

Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the Trial Flow Chart - Section 6.0. Details of each procedure are provided in Section 7.0 – Trial Procedures.

### 2.2 Trial Diagram

The trial design is depicted in Figure 1 (base study) and Figure 2 (study extensions 1, 2, and 3). Note that subjects who continue into the study extension(s) will have a single 14-day follow-up visit at the end of their last study extension only, and not in the base study.



<sup>&</sup>lt;sup>1</sup> Virologic failure or relapse is confirmed with 2 consecutive measurements of HIV-1 RNA at least one week apart.

Figure 1 Trial Diagram Base Study

Protocol/Amendment No.: 021-09



- Virologic failure or relapse is confirmed with 2 consecutive measurements of HIV-1-RNA at least 1 week apart.
- <sup>2</sup> Subjects enrolled in study extension 2 were discontinued from study therapy at the next scheduled study visit after MK1439A became available locally, ie, prior to Week 288.
- <sup>3</sup> Subjects enrolled in study extension 3 are discontinued from study therapy at the next scheduled study visit after MK-1439A becomes available locally, ie, prior to Week 384.

Figure 2 Trial Diagram Study Extensions 1, 2, and 3

#### 3.0 OBJECTIVE(S) & HYPOTHESIS(ES)

#### 3.1 Primary Objective(s) & Hypothesis(es)

#### 3.1.1 Base Study

In HIV-1 positive, treatment-naive subjects with pre-treatment HIV RNA ≥1,000 copies/mL:

1) **Objective:** To evaluate the non-inferior antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48.

**Hypothesis:** MK-1439A q.d. is non-inferior to ATRIPLA<sup>TM</sup> q.d. as assessed by the proportion of subjects with HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48. A margin of 10 percentage points is used to define non-inferiority.

- 2) **Objective:** To evaluate the safety and tolerability of MK-1439A q.d. compared with ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects with neuropsychiatric adverse events in the following categories:
  - Dizziness
  - Sleep disorders and disturbances
  - Altered Sensorium

Protocol/Amendment No.: 021-09

**Hypothesis**: MK-1439A q.d. is superior to ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects with neuropsychiatric adverse events in the following categories by Week 48 (superiority will be tested within category, sequentially, in the order indicated below):

- Dizziness
- Sleep disorders and disturbances
- Altered Sensorium

#### 3.2 Secondary Objective(s) & Hypothesis(es)

### 3.2.1 Base Study

In HIV-1 positive, treatment-naive subjects with pre-treatment HIV RNA  $\geq 1,000$  copies/mL:

- 1) **Objective**: To evaluate the safety and tolerability of MK-1439A q.d. compared to ATRIPLA™ q.d. as assessed by review of the accumulated safety data by Week 48 and Week 96.
- 2) **Objective**: To evaluate the effect of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. on fasting LDL-C as measured by the mean change from baseline at Week 48.
  - **Hypotheses**: MK-1439A q.d. is superior to ATRIPLA<sup>TM</sup> q.d. as assessed by the mean change from baseline in LDL-C at Week 48.
- 3) **Objective**: To evaluate the effect of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. on fasting non-HDL-C as measured by the mean change from baseline at Week 48.
  - **Hypotheses**: MK-1439A q.d. is superior to ATRIPLA<sup>TM</sup> q.d. as assessed by the mean change from baseline in non-HDL-C at Week 48.
- 4) **Objective:** To evaluate the safety and tolerability of MK-1439A q.d. compared with ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects with neuropsychiatric adverse events in the following categories:
  - Depression and suicide/self-injury
  - Psychosis and psychotic disorders
- 5) **Objective:** To evaluate the safety and tolerability of MK-1439A q.d. compared with ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects with at least one neuropsychiatric adverse event across the 5 categories of: dizziness, sleep disorders and disturbances, altered sensorium, depression and suicide/self-injury, and psychosis and psychotic disorders.

Protocol/Amendment No.: 021-09

6) **Objective:** To evaluate the safety and tolerability of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. as measured by the time to discontinuation from study due to an adverse experience.

- 7) **Objective**: To evaluate the immunologic effect of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d., as measured by the change from baseline in CD4 cell count at Week 48 and Week 96.
- 8) **Objective:** To evaluate the superior antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48.

**Hypothesis:** MK-1439A q.d. is superior to ATRIPLA<sup>TM</sup> q.d. as assessed by the proportion of subjects with HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48.

9) **Objective**: To evaluate the non-inferior antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d., as measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 96.

**Hypothesis**: MK-1439A q.d. is non-inferior to ATRIPLA<sup>TM</sup> q.d. as assessed by the proportion of subjects with HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 96. A margin of 10 percentage points is used to define non-inferiority.

10) **Objective**: To evaluate the superior antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d., as measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 96.

**Hypothesis**: MK-1439A q.d. is superior to ATRIPLA<sup>TM</sup> q.d. as assessed by the proportion of subjects with HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 96.

- 11) **Objective:** To evaluate the antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects achieving HIV-1 RNA below the limit of quantification of the Abbott RealTime HIV-1 Assay (<40 copies/mL) at Week 48 and Week 96.
- 12) **Objective:** To evaluate the pharmacokinetics of MK-1439, when administered as a component of MK-1439A, and the pharmacokinetic-pharmacodynamic association, if supported by the data

**Protocol/Amendment No.:** 021-09

### 3.3 Exploratory Objectives

#### 3.3.1 Base Study

In HIV-1 positive, treatment-naive subjects with pre-treatment HIV RNA  $\geq$ 1,000 copies/mL:

- 1) Objective: To evaluate the antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d. as measured by the proportion of subjects achieving HIV-1 RNA <200 copies/mL at Week 48 and Week 96.
- 2) **Objective:** To evaluate the antiretroviral activity of MK-1439A q.d. compared to ATRIPLA<sup>TM</sup> q.d., as measured by the TLOVR.
- 3) Objective: To assess the development of resistance to MK-1439A in subjects who have virologic failure.
- 4) Objective: To describe the outcomes for productivity and activity impairment related to general health during the study in MK-1439A relative to ATRIPLA<sup>TM</sup> q.d.
- 5) Objective: To explore the relationship between genetic variation and response to the treatment(s) administered. Variation across the human genome will be analyzed for association with clinical data collected in this study.

#### 3.3.2 Study Extension 1

- 1) **Objective:** To assess long-term efficacy and safety of MK-1439A administered for up to 192 weeks in subjects initially randomized to MK-1439A and enrolled in study extension 1.
- 2) **Objective:** To assess efficacy and safety of switching to MK-1439A for up to 96 weeks in subjects initially randomized to ATRIPLA<sup>TM</sup> q.d. and enrolled in study extension 1.

#### 4.0 BACKGROUND & RATIONALE

### 4.1 Background

Refer to the IB for detailed background information on MK-1439A.

### 4.1.1 Pharmaceutical and Therapeutic Background

HIV infection, which causes AIDS and for many years was associated with substantial morbidity and mortality, has now become a chronic disease that can be controlled through lifelong cART or HAART. Currently, there are more than 30 individual drugs and fixed-dose combinations available for the treatment of HIV-1 infection. These agents belong to 5 distinct mechanistic classes known as N(t)RTIs and NNRTIs, PIs, fusion inhibitors, entry inhibitors (CCR5 co–receptor antagonists), and InSTIs. Successful combinations of

**Protocol/Amendment No.:** 021-09

antiretroviral medications generally utilize 3 agents from at least 2 different mechanistic classes. The goal of cART is to suppress HIV to undetectable levels so that immune function is preserved or restored. Yet, while cART can delay disease progression and death, as well as reduce the risk of HIV transmission, it does not cure the infection. As a result, lifelong treatment must be maintained, which may lead to therapy fatigue and to non-compliance if the treatment regimen is difficult to adhere to (e.g., pill burden, frequency of treatment) and associated with intolerable side-effects. This can potentially lead to treatment failures with the possible development of resistant virus. Additionally, there is currently still significant concern regarding toxicities of some widely-used antiretroviral agents, including neuropsychiatric toxicities associated with efavirenz (EFV, an NNRTI), gastrointestinal toxicities such as diarrhea associated with multiple protease inhibitors (PIs), and serum lipid abnormalities associated with multiple mechanistic classes. Thus, potent treatment regimens that have an excellent safety and tolerability profile and are convenient to take are highly desirable.

For initiation of combination antiretroviral therapy for HIV infection, currently available NNRTIs constitute an important option for use as anchor agents, along with 2 NRTIs. Efavirenz and rilpivirine are both among the recommended therapies for treatment initiation according to multiple guidelines [1] [2]; however, each has limitations. For example, while efavirenz has shown excellent efficacy over many years of use, it is associated with substantial neuropsychiatric intolerance and skin rash, as well as lipid abnormalities. In addition it can be a perpetrator of drug-drug interactions as a mixed inducer or inhibitor of CYP3A and CYP2B6 enzymes. Rilpivirine has shown suboptimal efficacy in patients with high viral load or low baseline CD4 cells, and thus is not indicated in patients with baseline viral load above 100,000 copies/mL or CD4 count below 200 u/L. In addition, rilpivirine requires dosing with food, and while it is not a metabolic inducer or inhibitor, it is subject to metabolic induction/inhibition of CYP3A isoenzymes and should not be co-administered with proton pump inhibitors and several anticonvulsants. Importantly, high level resistance may occur in response to a single mutation for all currently available NNRTIs except etravirine, which must be dosed twice daily. Therefore, new agents of the NNRTI class that offer high potency, a distinct resistance profile, dosing convenience and a favorable safety and tolerability profile are needed.

As of the date of issuance of this protocol amendment, both MK-1439 and MK-1439A have been approved in multiple markets including the US, EU, Canada, Switzerland, and Australia for the treatment of HIV-1 infection in adult patients. MK-1439 is a potent inhibitor of HIV-1 replication in vitro and is active against both wild type virus and the most common NNRTI resistant variants at concentrations achieved with once-daily dosing. MK-1439 displays excellent potency against wild type virus with an IC<sub>50</sub> of 12 nM in the presence of 100% normal human serum. Preclinical studies also indicate a favorable in vitro resistance profile that is distinct from other NNRTIs, with IC<sub>50</sub>'s of 21, 31, and 55 nM against mutants containing the most frequently transmitted NNRTI mutations, K103N, Y181C and G190A, respectively, under the same conditions. The preclinical toxicity profile of MK-1439 is favorable in rats following dosing for up to 6 months at 3, 30, and 450 mg/kg/day, and in dogs following dosing for up to 9 months at 1, 10, and 1000 mg/kg/day. Clinical pharmacology studies indicate that MK-1439 can be dosed once-daily, without regard to

Protocol/Amendment No.: 021-09

food, and MK-1439 is not a metabolic inducer or inhibitor, reducing the likelihood of significant drug-drug interactions. Furthermore, the available long-term (beyond Week 48) data from a Phase 2 study in treatment-naive HIV-infected patients demonstrate that MK-1439 in combination with TDF/emtricitabine has a favorable safety and tolerability profile and potent efficacy, with ~76% of patients receiving MK-1439 achieving undetectable viral load (see Section 4.2.2.). These data provide key support for the initiation of the Phase 3 program, which includes evaluations of both MK-1439 as a single agent and MK-1439A as a fixed-dose regimen.

#### 4.2 Rationale

#### 4.2.1 Rationale for the Trial and Selected Subject Population

Factors that impact HIV treatment success include efficacy, safety and tolerability, barrier to resistance, simplicity/convenience of administration and drug-drug interactions. There is a clear medical need for new regimens that are highly effective, have a high barrier to resistance development, are very well tolerated, and are simple to administer (and thus facilitate increased adherence and prevent treatment fatigue). Therapies and regimens with these characteristics are particularly important for treatment-naïve patients for whom initial success is predictive of long-term outcomes and in the setting of lifelong treatment of HIV infection as many HIV patients become increasingly older with co-morbid diseases/conditions.

Currently, efavirenz is the preferred NNRTI for first-line therapy of treatment-naïve HIVinfected subjects. ATRIPLA<sup>TM</sup>, an FDR consisting of efavirenz 600 mg + emtricitabine 200 mg + TDF 300 mg, is the leading agent in HIV treatment. Efavirenz has demonstrated potent viral suppression but is associated with an increased risk of neuropsychiatric adverse experiences (AEs) (especially dizziness and sleep disorders) and lipid abnormalities relative to other therapies [1]. Efavirenz is also a perpetrator of numerous drug-drug interactions and, thus, may have limitations for use in aging patients who have an increased likelihood of using concomitant mediations. MK-1439 has been observed to have a more favorable neuropsychiatric AE and lipid profile relative to efavirenz in a Phase 2b study comparing the 2 agents, and, therefore, may result in improved patient tolerability and adherence [3] [4]. Additionally, based on in vitro data and drug-drug interactions studies conducted to date, MK-1439 is not expected to have many of the drug-drug interaction concerns currently hampering the use of efavirenz. Therefore, both MK-1439 and MK-1439A will provide valuable new treatment options for patients.

#### 4.2.2 Rationale for Dose Selection/Regimen

The FDR of MK-1439A contains 100 mg of MK-1439, a potent NNRTI, and standard doses of 2 commercially available and commonly used NRTIs, TDF (300 mg) and lamivudine (300

A 100 mg dose of MK-1439 was selected for Phase 3 development based on Phase 1b and 2 data and several other factors.


08K3V5

Protocol/Amendment No.: 021-09

In a Phase 1b study (Protocol 005), q.d. oral administration of 25 mg and 200 mg of MK-1439 as monotherapy for 7 days to treatment-naïve HIV-infected patients reduced plasma viral RNA burden as compared to placebo-treated controls. The mean change from baseline in log<sub>10</sub> HIV RNA copies/mL on Day 7 (24 hours postdose) was -1.52 for the MK-1439 25 mg group and was -1.41 for the MK-1439 200 mg group, while that for the placebo group was -0.15. The mean differences between MK-1439 25 mg and 200 mg versus placebo in change from baseline in log<sub>10</sub> HIV RNA copies/mL were -1.37 and -1.26, respectively.

Protocol 007 (Part 1) is a Phase 2 study designed to assess MK-1439 at doses of 25, 50, 100, and 200 mg q.d. versus efavirenz at 600 mg q.d., both in combination with the fixed-dose combination of TDF/FTC (TRUVADA<sup>TM</sup>) in treatment-naïve HIV-1 infected subjects. The MK-1439 dose range was selected based upon projections from in vitro data as well as the Phase 1b data in HIV-1 infected treatment-naïve individuals, which showed comparable virologic suppression at the 25 mg and 200 mg doses given once daily for 7 days.

In Protocol 007 (Part 1) 208 treatment-naïve HIV-1 infected subjects were treated with study drug (MK-1439 or efavirenz). At Week 24, all MK-1439 doses had rates of virologic suppression comparable to efavirenz for the key efficacy endpoints including the proportion of subjects with HIV-1 RNA levels <40 copies/mL (primary) or <200 copies/mL (secondary). All MK-1439 doses showed numerically higher response rates compared to efavirenz (80.0%, 76.2%, 71.4%, 78.0% versus 64.3% of patients with <40 copies/mL for the MK-1439 25 mg, 50 mg, 100 mg, 200 mg versus efavirenz arms, respectively) [3] [4]. The treatment differences (MK-1439 minus efavirenz) were not significant, and there was no dose response for efficacy observed. Overall 76.4% of patients receiving MK-1439 (at any dose) achieved <40 copies/mL compared with 64.3% for efavirenz. In addition. approximately 30% of subjects in the study had baseline HIV RNA above 100,000 copies/mL, and, in this subgroup, MK-1439 at all dosing levels showed virologic responses comparable to efavirenz. It should be acknowledged that this high viral load subgroup was relatively small, with approximately 12 subjects per dosing group. However, the totality of these efficacy data strongly support that the dose range studied (25-200 mg daily) was on the plateau of the dose response curve [4].

Similarly, the data from Protocol 007 showed an overall favorable safety and tolerability profile for MK-1439 compared with efavirenz, with no differentiation among MK-1439 doses (25 mg - 200 mg daily) with regard to safety. Based upon the 24-week results of Protocol 007, MK-1439 at doses ranging from 25-200 mg was generally well-tolerated, with no apparent dose related toxicity. Fewer drug-related AEs were observed for MK-1439 than for efavirenz (34.9% for MK-1439 overall vs. 57.1% for EFV), and fewer neuropsychiatric AEs were reported both at Week 8 and Week 24 (20.5% for MK-1439 overall vs. 33.3% for EFV at Week 8 and 23.4% for MK-1439 overall vs. 33.3% for EFV at Week 24) [3].

Because the safety and efficacy data from Protocol 007 did not distinguish among the doses tested, the selection of the MK-1439 100-mg daily dose for study in Part 2 of Protocol 007 and in the Phase 3 studies has taken into consideration a number of additional factors. Firstly, MK-1439 is a substrate of CYP3A metabolism and is subject to induction and inhibition of CYP3A by other concomitant medications. Consequently, the 100 mg dose is

Protocol/Amendment No.: 021-09

more likely than the lower doses to provide adequate MK-1439 exposures even in the setting of moderate metabolic inducers, and it allows for a safety margin in the setting of moderate metabolic inhibitors (since acceptable safety and tolerability were seen at the 200 mg dose in the Phase 2 study as well as at multiple doses and single doses as high as 750 mg and 1200 mg, respectively, in Phase 1 studies). Secondly, the 100-mg dose may provide forgiveness in the setting of the occasional missed dose. Thirdly, based on modeling and simulation, the 100-mg dose is predicted to provide adequate exposures and C<sub>trough</sub> concentrations in the setting of certain common NNRTI resistance mutations against which MK-1439 is considered to be active in vitro, including the K103N, Y181C, and Y190A mutations, as well as the dual K103N/Y181C mutation.

Patients receiving MK-1439 at 25, 50 or 200 mg in Part 1 of Protocol 007 were switched to 100 mg after dose selection. An additional 132 patients were randomized in Part 2, 66 to receive MK-1439 100 mg and 66 to receive EFV 600 mg. Combining Part 1 and 2, a total of 108 patients received MK-1439 100 mg, and 108 patients received EFV. By Week 8, at least one neuropsychiatric AE was reported in 22.2% of the MK-1439 group and 43.5% of the EFV group (p<0.001). The most commonly-reported neuropsychiatric AEs were dizziness (in 9.3% of patients receiving MK-1439 and 27.8% of patients receiving EFV), insomnia (in 6.5% of patients receiving MK-1439 and 2.8% of patients receiving EFV), abnormal dreams (in 5.6% of patients receiving MK-1439 and 16.7% of patients receiving EFV), and nightmares (in 5.6% of patients receiving MK-1439 and 8.3% of patients receiving EFV).

Standard marketed doses of lamivudine and TDF were selected for inclusion in MK-1439A because these dose levels have demonstrated efficacy and safety in treatment-naive subjects, and no antagonism was observed between MK-1439 and either of these drugs in in vitro studies.

ATRIPLA™, the active comparator in the base study will be administered at the standard approved dose of one tablet once daily. Each tablet contains 600 mg of efavirenz, 300 mg of tenofovir disoproxil fumarate (which is equivalent to 245 mg of tenofovir disoproxil) and 200 mg of emtricitabine.

#### 4.2.3 Rationale for Endpoints

#### 4.2.3.1 Efficacy Endpoints

The primary efficacy parameter in the study is viral load as measured by HIV-1 RNA, which is consistent with other clinical trials in HIV-infected patients and the current regulatory guidance. Suppressing HIV RNA to low levels preserves the immune system and prevents the development of opportunistic infections and progression of the disease. Clinical trials of antiretroviral agents in multiple classes have demonstrated that suppression of HIV RNA to levels below 50 copies/mL is a clinically meaningful endpoint. Therefore, the primary efficacy endpoint of this study is the proportion of subjects achieving HIV-1 RNA <50 copies/mL by the Abbott RealTime HIV-1 Assay. Week 48 was chosen as the primary efficacy time point and Week 96 as the secondary efficacy time point, as recommended by regulatory agencies for HIV treatment-naïve studies.

Protocol/Amendment No.: 021-09

Secondary and exploratory measurements for efficacy include HIV RNA <40 copies/mL (the lower limit of quantification of the Abbott RealTime HIV-1 Assay), HIV RNA <200 copies/mL, change from baseline in CD4 cell counts, time to loss of virologic response (TLOVR), and viral resistance for subjects who meet protocol-defined virologic failure criteria and whose virus can be amplified.

PDVF for this study is defined as one of the following:

1) Confirmed (2 consecutive measures at least one week apart) HIV-1 RNA ≥50 copies/mL after initial response of HIV-1 RNA <50 copies/mL at any time during the study

OR

2) Confirmed (2 consecutive measures at least one week apart) HIV-1 RNA ≥200 copies/mL at Week 24 or Week 36

OR

3) Confirmed (2 consecutive measures at least one week apart) HIV-1 RNA ≥50 copies/mL at Week 48.

Subjects should be discontinued, regardless of compliance with study therapy, if they meet the protocol-defined virologic failure criteria.

#### 4.2.3.2 Safety Endpoints

The primary safety endpoint in this study is assessed in the base study. The primary safety endpoint is the proportion of subjects with neuropsychiatric AEs by Week 48 in three categories; dizziness, sleep disorders, and altered sensorium (for example, depressed level of consciousness, lethargy, somnolence, syncope). The proportion of subjects with neuropsychiatric AEs by Week 48 in two additional categories, depression/suicide/self-injury and psychosis/psychotic disorders, will be secondary endpoints. All MedDRA preferred terms that fall under these categories will be grouped for the statistical tests on the difference in incidence rates between treatment groups within the categories. The full list of preferred terms defining these 5 categories is provided in Section 12.6.

Safety evaluations will include physical examinations (including vital signs) and laboratory tests (blood) performed at the visits indicated in the Trial Flow Chart (see Section 6.0). For subjects who continue into study extension 1, safety evaluations will include physical examinations (including vital signs) and laboratory test (blood) performed at each of the study visits, and if applicable, at the early discontinuation visit and/or a virologic failure confirmation visit and at a 14-day follow-up visit as shown in Trial Flow Chart B. AEs will be evaluated at each visit and graded according to the guidelines provided in Section 7.2. Subjects may be asked to return for unscheduled visits in order to perform additional safety monitoring.

Protocol/Amendment No.: 021-09

Note that after the administration of open-label study medication at Week 96, the first visit in study extension 1 is at Week 100, such that there is a 4-week interval following the last study treatment visit in the base study (Week 96). This interval was made shorter than the 12- to 16-week intervals beginning with Week 24 in the base study (and between subsequent visits in study extension 1) in order to more closely monitor all subjects, including those who are switched from ATRIPLA<sup>TM</sup> to MK-1439A, since treatment in the base study remains blinded at the beginning of study extension 1. Treatment group assigned during the base study will not be unblinded when a subject enters study extension 1; unblinding will occur after all subjects have completed the base study and database lock has been achieved for the base study (96-week treatment).

During study extension 2 and study extension 3, SAEs and pregnancy test results will be collected at each study visit (study extension 2: Week 208, Week 224, Week 240, Week 256, Week 272, and Week 288; study extension 3: Week 304, Week 320, Week 336, Week 352, Week 368, and Week 384, as applicable, depending on when MK-1439A is commercially available once approved in the local country, and, if applicable, at the early discontinuation and 14-day follow-up visits).

Secondary and exploratory measurements for safety include clinical and laboratory adverse experiences, change from baseline in fasting serum lipids, time to discontinuation due to an adverse experience and pre-defined limits of change in laboratory parameters.

### 4.2.3.3 Pharmacokinetic Endpoints

PK samples to be assayed for MK-1439 plasma concentrations will be collected at the Day 1 randomization visit as a predose sample. Population PK samples will also be taken at Weeks 4, 8, 24 and 48. At Week 4, the sample is to be collected predose. At Weeks 24 and 48, the samples are to be collected predose and within 0.5 to 2 hours postdose; at Week 8, the sample may be collected irrespective of time of dose (time of last dose and time of PK sample collection must be documented).

#### 4.2.3.4 Patient-Reported Outcome Endpoints

Subjects will complete a WPAI at Day 1, Week 4, Week 8, Week 16, and Week 48 (or the discontinuation visit). This patient-reported outcome questionnaire is designed to assess the quantitative impact of health conditions on loss of time and impaired productivity for functional activities such as work-for-pay, school work, and work around the house.

#### 4.2.3.5 Planned Exploratory Biomarker

08K3V5

Understanding genetic determinants of drug response is an important endeavor during medical research. This research will evaluate whether genetic variation within a clinical trial population correlates with response to the treatment(s) under evaluation. If genetic variation is found to predict efficacy or adverse events, the data might inform optimal use of therapies in the patient population. This research contributes to understanding genetic determinants of efficacy and safety associated with the treatments in this study.

02-Nov-2022

**Protocol/Amendment No.:** 021-09

#### 4.2.3.6 Future Biomedical Research

The Sponsor will conduct future biomedical research on specimens for which consent was provided during this study. This research may include genetic analyses (DNA), gene expression profiling (RNA), proteomics, metabolomics (serum, plasma), and/or the measurement of other analytes, depending on which specimens are consented for future biomedical research.

Such research is for biomarker testing to address emergent questions not described elsewhere in the protocol (as part of the main study) and will only be conducted on specimens from appropriately consented participants. The objective of collecting/retaining specimens for future biomedical research is to explore and identify biomarkers that inform the scientific understanding of diseases and/or their therapeutic treatments. The overarching goal is to use such information to develop safer, more effective drugs/vaccines, and/or to ensure that participants receive the correct dose of the correct drug/vaccine at the correct time. The details of future biomedical research are presented in Appendix 12.2. Additional informational material for institutional review boards/ethics committees (IRBs/ECs) and investigational site staff is provided in Appendix 12.3.

### 4.2.4 Rationale for Study Extensions

Because HIV infection is chronic, with treatment generally lifelong, collection of long-term safety and efficacy data will provide useful information on MK-1439A. Thus, after the 96-week double-blind period to evaluate the key primary and secondary objectives and hypotheses, there will be an open-label study extension ("study extension 1") for an additional 96-week period where all eligible subjects can continue to receive an open-label MK-1439A regimen.

Study extensions 2 and 3 were added to avoid interruption of treatment with MK-1439A for eligible subjects who are deriving benefit from treatment until MK-1439A is commercially available once approved in the local countries participating in the trial. This will also reduce the well-recognized, but small, risk of treatment failure associated with a change from a successfully suppressive and tolerated cART regimen.

#### 4.3 Benefit/Risk

08K3V5

Subjects in clinical trials generally cannot expect to receive direct benefit from treatment during participation, as clinical trials are designed to provide information about the safety and effectiveness of an investigational medicine.

MK-1439 is a promising new NNRTI for the treatment of HIV-1 infection. It is a potent inhibitor of HIV-1 replication in vitro and is active against both wild type virus and most common NNRTI resistant variants at concentrations achieved with once-daily dosing. In early studies, MK-1439 has been shown to be efficacious in combination with other ARTs in treatment-naïve patients. MK-1439 is not expected to have many of the safety concerns associated with EFV (especially neuropsychiatric AEs and dyslipidemia). In addition, MK-

02-Nov-2022

Protocol/Amendment No.: 021-09

1439 is not expected to have major drug-drug interactions that would limit its utility in clinical practice. Therefore, MK-1439 could represent a valuable addition to the HIV armamentarium for treatment-naïve patients. Additionally, the FDR, MK-1439A, which is used in this protocol, is a simplified regimen that could result in increased adherence, thereby potentially decreasing the risk of virologic failure.

Additional details regarding specific benefits and risks for subjects participating in this clinical trial may be found in the accompanying Investigator Brochure (IB) and Informed Consent documents.

#### 5.0 METHODOLOGY

#### 5.1 Entry Criteria

### 5.1.1 Diagnosis/Condition for Entry into the Trial

Male and female subjects 18 years of age or older who are HIV-1 positive and naïve to ART will be enrolled in this trial.

#### 5.1.2 Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

- 1. be at least 18 years of age on the day of signing the informed consent
- 2. understand the study procedures and voluntarily agree to participate by giving written informed consent (or have a legal representative provide written informed consent, if considered acceptable by local regulatory agencies and/or ERCs/IRBs) for the trial. The subject or his/her legal representative (if considered acceptable by local regulatory agencies and/or ERCs/IRBs) may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
- 3. be HIV-1 positive as determined by a positive result on an enzyme immunoassay, have screening plasma HIV-1 RNA (determined by the central laboratory) ≥1000 copies/mL within 45 days prior to the treatment phase of this study, and have HIV treatment indicated based on physician assessment. Local treatment guidelines should be considered in the decision to initiate therapy.
- 4. be naïve to ART including investigational antiretroviral agents.

<u>Note</u>: Naïve is defined as having received no (0 days of) ART therapy for the treatment of HIV infection.

**Protocol/Amendment No.:** 021-09

5. have the following laboratory values at screening within 45 days prior to the treatment phase of this study:

- a. Alkaline phosphatase  $\leq 3.0$  x upper limit of normal
- b. AST (SGOT) and ALT (SGPT) ≤5.0 x upper limit of normal
- c. Hemoglobin  $\geq 9.0 \text{ g/dL}$  (if female) or  $\geq 10.0 \text{ g/dL}$  (if male).

<u>Note</u>: A single repeat of a laboratory screening test will be allowed for test results that are unexpected based on documented prior laboratory results.

6. have a calculated creatinine clearance at the time of screening ≥50 mL/min, based on the Cockcroft-Gault equation which is as follows:

For males: 
$$Cl_{cr}(mL/min) = (140\text{-age}) \times weight (in kg)$$
  
72 x serum creatinine (mg/dL)

For females: 
$$Cl_{cr}$$
 (mL/min) =  $\underline{(140\text{-age})}$  x weight (in kg) x 0.85  
72 x serum creatinine (mg/dL)

- 7. in the opinion of the investigator, be considered clinically stable with no signs or symptoms of active infection at the time of entry into the study (i.e., clinical status and all chronic medications should be unchanged for at least 2 weeks prior to the start of treatment in this study).
- 8. be highly unlikely to become pregnant or to impregnate a partner since the subject falls into at least one of the following categories:
  - a. The subject is a male who is not of reproductive potential, defined as a male who has azoospermia (whether due to having had a vasectomy or due to an underlying medical condition).
  - b. The subject is a female who is not of reproductive potential, defined as a female who either: (1) is postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age); (2) has had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR (3) has a congenital or acquired condition that prevents childbearing.
  - c. The subject is a female or a male who is of reproductive potential and agrees to avoid becoming pregnant or impregnating a partner while receiving study drug and for 12 weeks after the last dose of study drug in the base study and 14 days after the last dose of study drug in the study extensions by complying with one of the following: (1) practice abstinence† from heterosexual activity OR (2) use (or have their partner use) acceptable contraception during heterosexual activity. Acceptable methods of contraception are‡:

**Protocol/Amendment No.:** 021-09

Single method (one of the following is acceptable):

- intrauterine device (IUD)
- vasectomy of a female subject's male partner

Combination method (requires use of 2 of the following):

- diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide)
- cervical cap with spermicide (nulliparous women only)
- contraceptive sponge (nulliparous women only)
- male condom or female condom (cannot be used together)
- hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, contraceptive rod implanted into the skin or subcutaneous contraceptive injection

Use of barrier methods of contraception is strongly encouraged to reduce the risk of HIV-1 transmission during sexual contact.

†Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.

‡If a contraceptive method listed above is restricted by local regulations/guidelines, then it does not qualify as an acceptable method of contraception for subjects participating at sites in this country/region.

Investigators should provide appropriate guidance to the subjects regarding use of contraceptives after completion of the study treatment. It is recommended that all subjects should continue to use contraception for 12 weeks following their last dose of study treatment in the base study (continued contraceptive use for 12 weeks following the last dose of ATRIPLA<sup>TM</sup> is required as per ATRIPLA<sup>TM</sup> prescribing information, and patients' study drug assignments will likely still be blinded following study completion). However, continued contraceptive use for 14 days following the last dose of study treatment is recommended in the study extensions since all subjects will be on MK-1439A.

**Protocol/Amendment No.:** 021-09

In order to be eligible for participation in **study extension 1** at the Week 96 visit, the subject must:

9. have completed the Week 96 visit.

- 10. be considered, in the opinion of the investigator, to have derived benefit from study participation through Week 96.
- 11. be considered, in the opinion of the investigator, a clinically appropriate candidate for an additional 96 weeks of treatment with MK-1439A following the end of the base study.
- 12. understand the procedures in study extension 1 and provide written informed consent to enter the study extension, thus continuing for approximately 2 years beyond the base study.

In order to be eligible to continue receiving study treatment in **study extension 2** at the Week 192 visit, the subject must:

- 13. have completed the Week 192 visit.
- 14. be considered, in the opinion of the investigator, to have derived benefit from MK-1439A by Week 192 of the study.
- 15. be considered, in the opinion of the investigator, a clinically appropriate candidate for an additional 2 years (additional 96 weeks) of treatment with MK-1439A.
- 16. understand the procedures in study extension 2 and have provided written informed consent to enter study extension 2, thus continuing until MK-1439A is commercially available once approved in the local country, or for up to approximately 2 years (whichever comes first) beyond study extension 1.

In order to be eligible to continue receiving study treatment in **study extension 3** at the Week 288 visit, the subject must:

- 17. have completed the Week 288 visit.
- 18. be considered, in the opinion of the investigator, to have derived benefit from MK-1439A by Week 288 of the study.
- 19. be considered, in the opinion of the investigator, a clinically appropriate candidate for an additional 2 years (additional 96 weeks) of treatment with MK-1439A.
- 20. understand the procedures in study extension 3 and have provided written informed consent to enter study extension 3, thus continuing until MK-1439A is commercially available once approved in the local country, or for up to approximately 2 years (whichever comes first) beyond study extension 2.
**Protocol/Amendment No.:** 021-09

# 5.1.3 Subject Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

1. has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

- 2. is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence. The nature and potential clinical context of the subject's illicit drug use, in relation to their exclusion from this trial, will be at the discretion of the Investigator.
- 3. has been treated for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1, including, but not limited to, adefovir, tenofovir, entecavir, emtricitabine, or lamivudine.

**Note**: Subjects may be enrolled if treatment occurred prior to the diagnosis of HIV.

- 4. has documented or known resistance to study drugs including MK-1439, efavirenz, emtricitabine, lamivudine, and/or tenofovir, as defined below:
  - a. Resistance to MK-1439 or efavirenz for the purpose of this study includes the following NNRTI mutations: L100I, K101E, K101P, K103N, K103S, V106A, V106I, V106M, V108I, E138A, E138G, E138K, E138Q, E138R, V179L, Y181C, Y181I, Y181V, Y188C, Y188H, Y188L, G190A, G190S, H221Y, L234I, P225H, F227C, F227L, F227V, M230L, M230I
  - b. Resistance to emtricitabine, lamivudine and tenofovir includes the following mutations: K65R, M41L, T69S (insertion complex), Q151M, M184I, M184V, L210W, T215F, T215Y, K219E, K219O, D67N, K70R and K70E.
- 5. has participated in a study with an investigational compound/device within 30 days prior to signing informed consent or anticipates participating in such a study involving an investigational compound/device during the course of this study.
- 6. has used systemic immunosuppressive therapy or immune modulators within 30 days prior to treatment in this study or is anticipated to need them during the course of the study.

<u>Note</u>: Short courses of corticosteroids (e.g., as for asthma exacerbation) will be allowed.

7. requires or is anticipated to require any of the prohibited medications noted in the protocol (refer to Section 5.5).

**Protocol/Amendment No.:** 021-09

8. has significant hypersensitivity or other contraindication to any of the components of the study drugs as determined by the investigator.

9. has a current (active) diagnosis of acute hepatitis due to any cause.

<u>Note</u>: Subjects with chronic hepatitis B and C may enter the study as long as they fulfill all entry criteria, have stable liver function tests, and have no significant impairment of hepatic synthetic function (significant impairment of hepatic synthetic function is defined as a serum albumin <2.8 mg/dL or an INR >1.7 in the absence of another explanation for the abnormal laboratory value).

10. has evidence of decompensated liver disease manifested by the presence of or a history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver diseases

or

has liver cirrhosis and a CPT score >9.

**Note:** To calculate the CPT score and associated Child-Pugh Class, refer to the following website: http://www.mdcalc.com/child-pugh-score-for-cirrhosis-mortality.

- 11. is pregnant, breastfeeding, or expecting to conceive.
- 12. is female and is expecting to donate eggs (at any time during the study) or is male and is expecting to donate sperm (at any time during the study).

<u>Note</u>: Investigators should provide appropriate guidance to the subjects regarding egg and sperm donation after completion of the study treatment. Consistent with the recommendations for contraceptive use, it is recommended that all subjects refrain from egg or sperm donation for 12 weeks following their last dose of study treatment in the base study and 14 days after the last dose of study treatment in the study extensions.

13. is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial.

#### 5.2 Trial Treatment(s)

Following completion of the Day 1 procedures and confirmation of eligibility, the site will contact the IVRS/IWRS for assignment of the study drug to be administered (MK-1439A or ATRIPLA). To maintain blinding, both drugs will be administered with a placebo matched to the other active drug in the study. Sites should not call IVRS/IWRS for drug administration until the subject has met all criteria for the study and is ready to receive the first dose of study medication on Day 1. The treatment groups to be used in this trial are outlined below in Table 1 for the base study and Table 2 for the extensions.

**Protocol/Amendment No.:** 021-09

Table 1 Trial Treatment During the Base Study

| Group 1 | n = 340 | MK-1439A one tablet PO q.d. <sup>†</sup> + placebo to match ATRIPLA <sup>TM</sup> one tablet PO q.d. <sup>#</sup> |
|---|---|---|
| Group 2 | n = 340 | ATRIPLA <sup>TM</sup> one tablet PO q.d. <sup>‡</sup> + placebo to match MK-1439A one tablet PO q.d. <sup>#</sup> |

<sup>&</sup>lt;sup>†</sup> MK-1439A is a single tablet FDR containing MK-1439 100 mg, lamivudine 300 mg, and tenofovir disoproxil fumarate (TDF) 300 mg.

Table 2 Trial Treatment During the Study Extensions

| Group 1 | Open-Label MK-1439A q.d. <sup>†</sup> |
|---|---|
| Group 2 | Open-Laber MK-1439A q.d. |
| † All subjects will receive MK-1439A (single-tablet, fixed-dose regimen (FDR) containing MK-1439 100 mg + lamivudine 300 mg + tenofovir disoproxil fumarate 300 mg) in the study extensions. | |

Subjects will receive study medication at the Day 1 visit and should take the first dose of medication on the same day.

MK-1439A (during the base study and study extensions) and the placebo to match MK-1439A are to be taken once daily without regard to food at approximately the same time each day.

ATRIPLA<sup>TM</sup> and the placebo to match ATRIPLA<sup>TM</sup> are to be taken once daily at bedtime on an empty stomach.

Study medications for the base study (MK-1439A/placebo or ALTRIPA<sup>TM</sup>/placebo) and for the study extensions (MK-1439A) will be provided centrally by the Sponsor.

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of trial treatments in accordance with the protocol and any applicable laws and regulations.

#### **5.2.1** Dose Selection

# **5.2.1.1** Dose Selection (Preparation)

The rationale for selection of doses to be used in this trial is provided in Section 4.0 – Background & Rationale. There are no specific calculations or evaluations required to be performed in order to administer the proper dose to each subject.

<sup>&</sup>lt;sup>‡</sup> ATRIPLA™ is a single tablet FDR containing efavirenz 600 mg, emtricitabine 200 mg, and TDF 300 mg (which is equivalent to 245 mg of tenofovir disoproxil).

<sup>&</sup>lt;sup>#</sup> Placebos are used to maintain blinding.

Protocol/Amendment No.: 021-09

# **5.2.1.2** Dose Modification/Interruption (Base Study or the Study Extensions)

#### Dose Modification:

No dose modification of study therapy is allowed during the study.

#### Dose Interruption:

Consideration should be given to interrupting study therapy for toxicity management (see Section 7.1.2.6).

Interruptions from the protocol specified treatment plan that are expected to be 7 days or greater require consultation between the investigator and the Sponsor and written documentation of the collaborative decision on subject management.

#### **5.2.2** Timing of Dose Administration

#### **5.2.2.1** Base Study

#### Bottle A (MK-1439A or placebo):

Subjects will be instructed to take one tablet from Bottle A once a day (q.d.) orally, with or without food at the approximately the same time each day.

If a subject misses a dose of drug from Bottle A and it is less than 12 hours before the next dose, the missed dose should be skipped and the normal dosing schedule resumed. The subject should not double the next dose in order to compensate for what has been missed. If a subject misses a dose and it is greater than 12 hours before the next dose, the missed dose should be taken and the normal dosing schedule resumed.

# Bottle B (ATRIPLA<sup>TM</sup> or placebo):

Subjects will be instructed to take one tablet from Bottle B once a day orally, on an empty stomach at bedtime.

If a subject misses a dose of drug from Bottle B and it is less than 12 hours before the next dose, the missed dose should be skipped and the normal dosing schedule resumed. The subject should not double the next dose in order to compensate for what has been missed. If a subject misses a dose and it is greater than 12 hours before the next dose, the missed dose should be taken and the normal dosing schedule resumed.

#### 5.2.2.2 Study Extensions

# Bottle C (MK-1439A), open-label:

Subjects will be instructed to take one tablet from Bottle C once a day (q.d.) orally, with or without food at the approximately the same time each day.

Protocol/Amendment No.: 021-09

If a subject misses a dose of drug from Bottle C and it is less than 12 hours before the next dose, the missed dose should be skipped and the normal dosing schedule resumed. The subject should not double the next dose in order to compensate for what has been missed. If a subject misses a dose and it is greater than 12 hours before the next dose, the missed dose should be taken and the normal dosing schedule resumed.

# 5.2.3 Trial Blinding/Masking

A double-blind/masking technique will be used. MK-1439A, ATRIPLA™, and their respective placebos will be packaged so that blind/masking is maintained in the base trial. The subject, the investigator and Sponsor personnel or delegate(s) who are involved in the treatment or clinical evaluation of the subjects are unaware of the group assignments. During the trial extensions, MK-1439A will be provided open-label.

See Section 7.1.4.2, Blinding/Unblinding, for a description of the method of unblinding a subject during the trial, should such action be warranted.

#### 5.3 Randomization or Treatment Allocation

Randomization will occur centrally using an interactive voice response system / integrated web response system (IVRS/IWRS). There are 2 treatment arms. Subjects will be assigned randomly in a 1:1 ratio to MK-1439A q.d. or ATRIPLA<sup>TM</sup> q.d. in the base study.

#### 5.4 Stratification

Randomization in the base study will be stratified according to the following factors:

- 1. Screening HIV-1 RNA (≤100,000 or >100,000 copies/mL), based on central laboratory result
- 2. Chronic Hepatitis B and/or C infection status (yes or no). Hepatitis status is defined by serologic evidence of chronic hepatitis B surface antigen and/or evidence of HCV RNA by a PCR quantitative test for hepatitis C virus.

Thus, IVRS/IWRS will randomize subjects within 4 strata as outlined in Table 3.

Table 3 Stratification

| Stratum | Screen HIV-1 RNA levels (copies/mL) | Chronic Hepatitis B and/or<br>Chronic Hepatitis C |
|---|---|---|
| I | ≤100,000 | No |
| II | ≤100,000 | Yes |
| III | >100,000 | No |
| IV | >100,000 | Yes |

**Protocol/Amendment No.:** 021-09

# 5.5 Concomitant Medications/Vaccinations (Allowed & Prohibited)

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for any medication or vaccination specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Sponsor Clinical Director. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician. However, the decision to continue the subject on trial therapy or vaccination schedule requires the mutual agreement of the investigator, the Sponsor and the subject.

No medications are to be taken within 30 days of the start of the study without the knowledge of the investigator.

Listed below are specific restrictions for concomitant therapy or vaccination during the course of the trial:

# Permitted Concomitant Medications/Therapies

The concomitant use of other medications/therapies is allowed unless specifically prohibited in the Prohibited Concomitant Medications/Therapies section below. Before placing a subject on a specific medication/therapy, it is the responsibility of the investigator to check on potential drug-drug interactions between that medication/therapy and ATRIPLA<sup>TM</sup>.

- 1. Use of oral or other hormonal contraception is permitted.
- 2. Newly approved regimens for the treatment of HCV infection are permitted, as long as there are no known potential drug-drug interactions between those treatments and any of the study medications. The MSD Clinical Director or designee should be contacted if there are any questions about whether there is a potential drug-drug interaction with a specific treatment that the Investigator is planning to give the subject.

# **Prohibited Concomitant Medications/Therapies**

In general, concomitant use of immune therapy agents or other immunosuppressive therapy, including interferon-based treatment for hepatitis, is not allowed during the course of the study. Important **exceptions** to this rule include:

- Short courses of corticosteroids (e.g., as for asthma exacerbation) are allowed.
- Intralesional or localized electron beam therapy for cutaneous Kaposi's sarcoma is permitted.
- If a subject develops a malignancy (for example lymphoma) after randomization, the subject **may receive** chemotherapy (including cancer immunotherapy) and remain in the study if, in the opinion of the investigator, the benefits outweigh the risks.

MK-1439A-021-09 Final Protocol 02-Nov-2022 Confidential

Protocol/Amendment No.: 021-09

Depending on the type of chemotherapy, study medication may need to be interrupted until completion of the chemotherapy.

Antiretroviral therapies other than those used in the study (MK-1439A, and ATRIPLA<sup>TM</sup>) are also not permitted during the course of the study.

Investigational agents must be discontinued 30 days prior to treatment in this study and are not permitted during the course of the study.

# Prohibited Concomitant Therapy Due to Potential Interactions with MK-1439A

MK-1439 is expected to be eliminated mainly via CYP-mediated oxidation.

The medications and/or substances below are prohibited in this study because they are moderate or potent inducers of CYP3A4 and their co-administration with MK-1439A could possibly result in reduced drug levels of MK-1439 or has the potential for additional drugdrug interactions.

Since this list is not comprehensive, the investigator should use his/her medical judgment when a subject presents with a medication not on the list or call the Sponsor Clinical Director or Designee for clarification.

# **Prohibited Medication/Therapy Due to MK-1439 Interactions During the Base Study and Study Extensions** Carbamazepine Enzalutamide Mitotane Oxcarbazepine Rifapentine Phenobarbital Phenytoin Rifabutin Rifampin St. John's Wort Modafinil Bosentan Nafcillin

# Prohibited Concomitant Therapy Due to Potential Interactions with ATRIPLA<sup>TM</sup>

Specific medications are prohibited during the base study due to potential interactions with ATRIPLA<sup>TM</sup>. Efavirenz induces CYP3A4 metabolism and may significantly reduce the exposure of CYP3A4 substrates. In addition, there are some medications that may significantly alter the metabolism of efavirenz. In some cases, co-administration of certain

Protocol/Amendment No.: 021-09

drugs with ATRIPLA<sup>TM</sup> may lead to significant safety risks. The following medications are prohibited in this study because they: (1) are contraindicated for concomitant use with ATRIPLA<sup>TM</sup> (according to one or more available ATRIPLA<sup>TM</sup> package circulars), (2) may alter the plasma concentration of one or more of the ATRIPLA<sup>TM</sup> components and/or (3) may have significant changes in their plasma concentrations when co-dosed with ATRIPLA<sup>TM</sup> that would require additional monitoring or dose adjustment, which is not feasible in the setting of a double-blind trial.

# Prohibited Medication/Therapy Due to ATRIPLA<sup>TM</sup> Interactions During the Base Study

Artermether Astemiazole Bepridil **Boceprevir** Carbamazepine<sup>†</sup> Cisapride Clarithromycin Cyclosporine Dihydroatenisinin Ergot derivatives Itraconazole Ketoconazole Lumefantrine Midazolam Phenobarbital<sup>†</sup> Phenytoin<sup>†</sup> Pimozide Rifabutin<sup>†</sup> Rifampin<sup>†</sup> Simeprevir Sirolimus St. John's Wort<sup>†</sup> **Tacrolimus Telaprevir** Terfenadine Triazolam Voriconazole

<sup>†</sup> Several of these medications are also prohibited during the study extensions because of interaction with MK-1439A: specifically, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin and St. John's Wort are prohibited throughout the base study and the study extensions.

**Protocol/Amendment No.:** 021-09

The investigator should discuss any questions regarding this with the Sponsor Clinical Director.

# **Concomitant Therapy to be Used With Caution**

For complete information, please refer to the ATRIPLA<sup>TM</sup> package circular available locally for drugs that are permitted in the protocol but that should be used with caution, since they have established drug interactions with ATRIPLA<sup>TM</sup>.

# **5.6** Rescue Medications & Supportive Care

No rescue or supportive medications are specified to be used in this trial.

# 5.7 Diet/Activity/Other Considerations

#### Diet

MK-1439A (or placebo) can be taken without regard to food and should generally be taken at approximately the same time each day.

ATRIPLA<sup>TM</sup> (or placebo) should be taken at bedtime on an empty stomach.

#### Alcohol/Substance Abuse

Subjects should be questioned about their estimated daily intake of alcohol and about substance abuse during the screening evaluation of eligibility. Any subject who in the opinion of the investigator has an excessive intake of any of these substances must be excluded from the study.

# 5.8 Subject Withdrawal/Discontinuation Criteria

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the discretion of the investigator should any untoward effect occur. In addition, a subject may be withdrawn by the investigator or the Sponsor if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons. Specific details regarding discontinuation or withdrawal procedures; including specific details regarding withdrawal from Future Biomedical Research, are provided in Section 7.1.4 — Other Procedures.

Discontinuation from treatment is "permanent". Once a subject is discontinued, he/she shall not be allowed to restart treatment.

A subject must be discontinued from the trial for any of the following reasons:

• The subject or legal representative (such as a parent or legal guardian) withdraws consent.

Protocol/Amendment No.: 021-09

Note: Please provide additional detail for the reason the subject withdrew consent on the Subject Disposition eCRF.

- The subject has a medical condition or personal circumstance which, in the opinion of the investigator and/or Sponsor, places the subject at unnecessary risk through continued participation in the trial or does not allow the subject to adhere to the requirements of the protocol; these may include, but are not limited to:
  - clinical or laboratory findings suggestive of lactic acidosis or pronounced hepatotoxicity (which may include symptomatic hyperlactatemia, metabolic/lactic acidosis, progressive hepatomegaly, rapidly elevating aminotransferase levels, and hepatomegaly and steatosis even in the absence of marked transaminase elevations).
  - o severe rash associated with blistering, desquamation, mucosal involvement or fever (base study)
  - o severe depression, psychosis or suicidal ideation (base study).
- The subject has a confirmed positive serum/urine pregnancy test.

<u>Note</u>: Subjects who become pregnant during the study will be asked to join a pregnancy registry which collects information about the outcome of the pregnancy.

- The subject fails to comply with the dosing, evaluations, or other requirements of the trial.
- A physician investigator feels it is in the best interest of the subject to discontinue.
- The subject has an adverse experience or tolerability issue related to study medication which requires discontinuation of the medication.
- Subject has a creatinine clearance of <50 mL/min (confirmed by repeat measurement) based on the Cockcroft-Gault equation:

#### Male:

 $Cl_{cr}(mL/min) = (140-age) \times weight (in kg)$ 72 x serum creatinine (mg/dL)

#### Female:

08K3V5

 $Cl_{cr}$  (mL/min) =  $\underline{(140\text{-age}) \text{ x weight (in kg)}}$  X 0.85 72 x serum creatinine (mg/dL)

or subject has serum phosphorous <0.32 mmol/l.

**Note**: Subjects with serum phosphorous <0.48 mmol/l should be closely monitored.

**Protocol/Amendment No.:** 021-09

• Subject requires interferon-based treatment for hepatitis.

- Subjects should be discontinued, regardless of compliance with study therapy, if they meet the protocol-defined virologic failure criteria in Section 4.2.3.1.
- Subjects who participate in study extension 2 or study extension 3 should be discontinued at the next scheduled visit after MK-1439A is commercially available once approved in the local country.

Subjects who require discontinuation of study therapy must be discontinued from the trial.

Subjects who discontinue study therapy prior to the last scheduled treatment visit should have an Early Discontinuation visit and a 14-day follow-up visit conducted.

Due to the potential for severe acute exacerbations of hepatitis B following discontinuation of ATRIPLA<sup>TM</sup>, lamivudine and tenofovir, subjects who are co-infected with hepatitis B who stop their assigned study therapy at or prior to the end of the study must be closely monitored for such exacerbations for at least 6 months. This requirement applies to subjects in both treatment arms.

If approved by the Sponsor, a subject can remain on study if they cannot make it to regularly scheduled study visits due to unforeseen circumstances but are able to remain on study therapy and the Investigator believes it is in the best interest of the subject to do so.

Once discontinued from the base study, a subject is not eligible to enter study extension 1. A subject who completes the base study and does not elect to participate in study extension 1 is considered to have completed the study. Once discontinued from study extension 1, a subject is not eligible to enter study extension 2. Once discontinued from study extension 2, a subject is not eligible to enter study extension 3.

#### 5.9 Subject Replacement Strategy

A subject who discontinues from the trial will not be replaced.

#### 5.10 Beginning and End of the Trial

The overall trial begins when the first subject signs the informed consent form. The overall trial ends when the last subject completes the last study-related phone call or visit, discontinues from the trial or is lost to follow-up (i.e. the subject is unable to be contacted by the investigator).

**Protocol/Amendment No.:** 021-09

#### 5.11 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

1. The eDMC recommends the trial be terminated and the EOC agrees.

Further recruitment in the trial or at a particular trial site(s) may be stopped due to insufficient compliance with the protocol, GCP, and/or other applicable regulatory requirements, procedure-related problems, or the number of discontinuations for administrative reasons is too high.

**Protocol/Amendment No.:** 021-09

#### **6.0 TRIAL FLOW CHART**

Flow Chart A applies to all subjects in the base study from screening through follow-up after the Week 96 visit. Flow Chart B applies to those subjects continuing into study extension 1 from Week 96 through follow-up after the Week 192 visit. Flow Chart C applies to those subjects continuing into study extension 2 from Week 208 through follow-up after the Week 288 visit. Flow Chart D applies to those subjects continuing into study extension 3 from Week 304 through follow-up after the Week 384 visit.

Flow Chart A (Base Study): Screening Through Week 96 Plus 14 Days Follow-up<sup>b</sup>

| Visit Number/Title: | 1 | 2<br>Random-<br>ization | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | U (Virologic<br>Failure<br>Confirmation) | U (Early<br>Discontinuation) | 99 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period | Screen-<br>ing | | | | | Tre | atment | ı | | | | | | | Post-<br>treatment <sup>b</sup> |
| | | Fasting | WK | WK | WK | Fast-<br>ing <sup>c</sup><br>WK | WK | Fast-<br>ing <sup>c</sup><br>WK | WK | WK | WK | Fast-<br>ing <sup>c</sup><br>WK | ≥1 to ≤4 wks<br>after initial<br>virologic | At time of | Post-study<br>14-day |
| Trial Procedures | Screen | Day 1 <sup>d</sup> | 4 | 8 | 16 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | failure | Discon | follow-up <sup>b</sup> |
| Administrative Procedures | T | 1 | | 1 | | | | | | | | | | • | |
| Informed Consent | X | | | | | | | | | | | Xe | | | |
| Informed Consent for Future<br>Biomedical Research <sup>f</sup> | X | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | Xe | | | |
| Provide Subject Identification Card | X | | | | | | | | | | | | | | |
| Medical History <sup>g</sup> | X | | | | | | | | | | | | | | |
| Concomitant Medication Review | X | X | X | X | X | X | X | X | X | X | X | X | | X | X |
| Treatment Allocation/Randomization | | X | | | | | | | | | | | | | |
| Register Study Visit via Interactive<br>Voice (Web) Response System<br>(IVRS/IWRS) | X | X | X | X | X | X | X | X | X | X | X | X | | X | |
| Dispense Study Therapy via IVRS/IWRS | | X | X | X | X | X | X | X | X | X | X | X <sup>h</sup> | | | |
| Provide/Review Study Medication<br>Diary | | X | X | X | X | X | X | X | X | X | X | X | | X | |
| Patient-Reported Outcomes <sup>i</sup> | | X | X | X | X | • | | X | | | | | | $\mathbf{X}^{\mathrm{j}}$ | |
| Assess Subject Eligibility for Study<br>Extension 1e | | | | | | | | | | | | X | | | |

**Protocol/Amendment No.:** 021-09

| Visit Number/Title: | 1 | 2<br>Random-<br>ization | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | U (Virologic<br>Failure<br>Confirmation) | U (Early<br>Discon-<br>tinuation) | 99 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period | Screen-<br>ing | | | | | Tre | atment | ı | | | | | , | Í | Post-<br>treatment <sup>b</sup> |
| | | Fasting <sup>c</sup> | WK | WK | WK | Fast-<br>ing <sup>c</sup><br>WK | WK | Fast-<br>ing <sup>c</sup><br>WK | WK | WK | WK | Fast-<br>ing <sup>c</sup><br>WK | ≥1 to ≤4 wks<br>after initial<br>virologic | At time of | Post-study<br>14-day |
| Trial Procedures | Screen | Day 1 <sup>d</sup> | 4 | 8 | 16 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | failure | Discon | follow-up <sup>b</sup> |
| Clinical Procedures/Assessments | • | | | | | | | | | | | | | | |
| Full Physical Examination | X | | | | | | | | | | | | | | |
| Directed Physical Examination | | X | X | X | X | X | X | X | X | X | X | X | | X | X |
| Height | X | | | | | | | | | | | | | | |
| Vital Signs (including pulse rate,<br>blood pressure, respiratory rate, and<br>body temperature) and Weight | X | X | X | X | X | X | X | X | X | X | X | X | | X | X |
| 12-Lead Electrocardiogram (ECG) (Local) <sup>k</sup> | | $X^{k,l}$ | | | | | | | | | | | | | |
| Adverse Events Monitoring | X | X | X | X | X | X | X | X | X | X | X | X | | X | X |
| Birth Control Confirmation | X | X | X | X | X | X | X | X | X | X | X | X | | X | X |
| <b>Laboratory Procedures/Assessments</b> | | | | | | | | | | | | | | | |
| Serum Pregnancy Test <sup>m</sup> | X | | | | | | | | | | | | | | |
| Urine Pregnancy Test <sup>m</sup> | | $X^{l}$ | X | X | X | X | X | X | X | X | X | X | | X | X |
| Collect Blood for Safety Laboratory<br>Tests (Hematology/Chemistry) <sup>n</sup> | $X^l$ | X | X | X | X | X | X | X | X | X | X | X | Xº | X | X |
| Hemostatic Function Test <sup>p</sup> | $X^{l}$ | | | | | | | | | | | | | | |
| HIV/Hepatitis Screen <sup>q</sup> | $X^{l}$ | | | | | | | | | | | | | | |
| Virology Test Plasma HIV viral RNA<br>quantification test (Abbott Real Time<br>HIV-1) | X <sup>l</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Collect Blood for CD4 Cell Count | X | X | | X | | X | | X | | X | | X | | | |
| Collect Blood for MK-1439 PK <sup>r</sup> | | X | X | X | | X | | X | | | | | | | |
| Collect Plasma for Viral Resistance<br>Test | X | | X | X | X | X | X | X | X | X | X | X | X | Xs | |
| Collect Blood (DNA) for Genetic<br>Analysis <sup>f</sup> | | X | | | | | | | | | | | | | |
| Collect Plasma for Future Biomedical Research <sup>f</sup> | | X | | | | | | X | | | | X | | | |

Protocol/Amendment No.: 021-09

| Visit Number/Title: | 1 | 2<br>Random-<br>ization | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | U (Virologic<br>Failure<br>Confirmation) | U (Early<br>Discon-<br>tinuation) | 99 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period | Screen-<br>ing | | | | | Tre | atment | ı | | | | | | | Post-<br>treatment <sup>b</sup> |
| Trial Procedures | Screen | Fasting <sup>c</sup><br>Day 1 <sup>d</sup> | WK | WK<br>8 | WK<br>16 | Fast-<br>ing <sup>c</sup><br>WK<br>24 | WK<br>36 | Fast-<br>ing <sup>c</sup><br>WK<br>48 | WK<br>60 | WK<br>72 | WK<br>84 | Fast-<br>ing <sup>c</sup><br>WK<br>96 | ≥1 to ≤4 wks<br>after initial<br>virologic<br>failure | At time of Discon | Post-study<br>14-day<br>follow-up <sup>b</sup> |

- a. Visit window periods are approximately ±3 days for the Week 4 to Week 24 visits and approximately ±7 days for the Week 36 to Week 96 visits. The timing of each visit is relative to the randomization (Day 1) visit. Every attempt must be made to keep subjects on schedule.
- b. The follow-up visit 14 days after the Week 96 visit in the base study applies only to subjects who do not enter study extension 1. The visit window period for the Post-study 14-day follow-up visit is approximately -2 to 0 days.
- c. Fasting for at least 8 hours. Fasting is required at these visits for lipids measurement.
- d. Within 45 days of screening visit and prior to the first dose on Day 1.
- e. If the subject is eligible and elects to enter study extension 1, he/she will be considered to have completed the base study and will, after providing informed consent for study extension 1, immediately enter study extension 1.
- f. This sample should be drawn for planned genetic analysis of DNA and drug response unless there is either a documented law or regulation prohibiting collection, or unless the IRB/IEC does not approve of the collection of the sample for these purposes. If the sample is collected, any leftover extracted DNA will be stored for future biomedical research if the subject signs the Future Biomedical Research consent. Plasma samples for Future Biomedical Research should be collected at Day 1, and Weeks 48 and 96.
- g. Includes smoking history.
- h. For Week 96, drug will be dispensed only to subjects who enter study extension 1, after providing informed consent.
- i. Includes 1 questionnaire: Work Productivity and Activity Impairment Questionnaire (WPAI).
- Not applicable for subjects who discontinue after Week 48.
- k. A local ECG should be performed prior to the subject's first dose of study medication (within 7 days prior to the Study Day 1 visit).
- 1. Results of test must be available prior to randomization.
- m. For women of childbearing potential.
- n. Refer to Table 4 for listing of specific blood safety tests.
- o. For creatinine clearance only.
- p. Hemostatic Function Test includes: Prothrombin time (PT), Activated Partial Thromboplastin Time (APTT), and International Normalized Ratio (INR).
- q. HIV/Hepatitis Screen tests includes: Enzyme immunoassay HIV antibody screen, Serum Hepatitis B surface antigen, Serum Hepatitis B surface antibody, Serum Hepatitis B e-antigen and Serum Hepatitis C antibody. A plasma hepatitis C virus PCR quantitative test will be performed if the Hepatitis C antibody test is positive.
- r. One sample for assay of MK-1439 plasma concentrations will be collected at Day 1 (Pre-dose), Week 4 (pre-dose), and Week 8 (random). At Weeks 24 and 48, 2 samples will be collected, pre-dose and 30 mins to 2 hours postdose (the subject should be fasting for both samples).
- s. If virologic failure is confirmed (with a confirmatory HIV-1 RNA at least one week later), and the decision is made to discontinue the subject, plasma for resistance need not be collected again at the early discontinuation visit. All other early discontinuation tests should be performed at the early discontinuation visit.

**Protocol/Amendment No.:** 021-09

# Flow Chart B (Study Extension 1): Week 100 Through Week 192 Plus 14 Days Follow-up

| Visit Number/Title: | 13ª | 14 | 15 | 16 | 17 | 18 | 19 | U (Virologic Failure<br>Confirmation) | U (Early<br>Discontinuation) | 99 |
|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period | | | | Treatmen | t <sup>b</sup> | | | | | |
| TRIAL PROCEDURES | WK<br>100 | WK<br>116 | WK<br>132 | Fasting<br>WK<br>148 | WK<br>164 | WK<br>180 | Fasting<br>WK<br>192 | ≥1 to ≤4 wks<br>after the time virologic<br>failure is first identified | At time of Discontinuation | Post-study<br>14-day<br>follow-up |
| Administrative Procedures | | | | | | | | | | |
| Concomitant Medication Review | X | X | X | X | X | X | X | | X | X |
| Register Study Visit via Interactive Voice Response System (IVRS/IWRS) <sup>c</sup> | X | X | X | X | X | X | X | | X | |
| Dispense Study Therapy (Open-Label MK-1439A) | X | X | X | X | X | X | X <sup>d</sup> | | | |
| Provide/Review Study Medication Diary | X | X | X | X | X | X | X | | X | |
| Assess Subject Eligibility for Study Extension 2 <sup>e</sup> | | | | | | | X | | | |
| Informed Consent for Study Extension 2 <sup>e</sup> | | | | | | | X | | | |
| Clinical Procedures/Assessments | | | | | | | | | | |
| Directed Physical Examination | X | X | X | X | X | X | X | | X | X |
| Vital Signs (including pulse rate, blood pressure, respiratory rate, & body temperature) and Weight | X | X | X | X | X | X | X | | X | X |
| Adverse Events Monitoring | X | X | X | X | X | X | X | | X | X |
| <b>Laboratory Procedures/Assessments</b> | | | | | | | | | | |
| Urine Pregnancy test <sup>f</sup> | X | X | X | X | X | X | X | | X | X |
| Collect Blood for Safety Laboratory Tests<br>Hematology/Chemistry <sup>g</sup> | X | X | X | X <sup>h</sup> | X | X | X <sup>h</sup> | X <sup>i</sup> | X | X |
| Virology Test Plasma HIV viral RNA quantification test (Abbott RealTime HIV-1) | X | X | X | X | X | X | X | X | X | X |
| Collect Blood for CD4 Cell Count | X | | | X | | | X | | | |
| Collect Plasma for Viral Resistance Test | | | | | | | | X | $X^{j}$ | |

**Protocol/Amendment No.:** 021-09

| Visit Number/Title: | 13 <sup>a</sup> | 14 | 15 | 16 | 17 | 18 | 19 | U (Virologic Failure<br>Confirmation) | U (Early<br>Discontinuation) | 99 |
|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period | | | | Treatmen | t <sup>b</sup> | | | | | |
| TRIAL PROCEDURES | WK<br>100 | WK<br>116 | WK<br>132 | Fasting<br>WK<br>148 | WK<br>164 | WK<br>180 | Fasting<br>WK<br>192 | ≥1 to ≤4 wks<br>after the time virologic<br>failure is first identified | At time of Discontinuation | Post-study<br>14-day<br>follow-up |

- a. Subjects who enter study extension 1 are considered enrolled in study extension 1 upon providing written informed consent for study extension 1 at the Week 96 study visit of the base study.
- b. The visit window for Week 100 is approximately ±7 days, for all visits from Week 116 through Week 192 the windows are approximately ±14 days and, for the post-study 14-day follow-up visit, the window is approximately -2 to 0 days. The timing of each visit is relative to the randomization (Day 1) visit. Every attempt must be made to keep subjects on schedule.
- c. IVRS/IWRS will be used to allocate drug and to manage distribution of clinical supplies.
- d. Study drug for extension 2 will be dispensed at Week 192, if subject is continuing into extension 2.
- e. If the subject is eligible and elects to enter study extension 2, he/she will be considered to have completed study extension 1 and will, after providing informed consent, immediately enter study extension 2 and be dispensed MK-1439A.
- f. For women of childbearing potential.
- g. Refer to Table 4 for listing of specific blood safety and chemistry tests.
- h. Fasting at least 8 hours prior to study visit is required for lipids measurement at Week 148 and Week 192.
- i. For creatinine clearance only.
- j. If virologic failure is confirmed (with a confirmatory HIV-1 RNA at least one week later), and the decision is made to discontinue the subject, plasma for resistance need not be collected again at the early discontinuation visit. All other early discontinuation tests should be performed at the early discontinuation visit.

**Protocol/Amendment No.:** 021-09

# Flow Chart C (Study Extension 2): Week 208 Through Up to Week 288 Plus 14 Days Follow-up

| Visit Number/Title | 20ª | 21 | 22 | 23 | 24 | 25 | U (Early<br>Discontinuation) | 99 |
|---|---|---|---|---|---|---|---|---|
| Trial Period | | | 7 | Γreatn | nent <sup>b,c</sup> | | | |
| TRIAL PROCEDURES | WK<br>208 | | | | WK<br>272 | WK<br>288 | At time of Discontinuation | Post-study<br>14-day follow-up <sup>d</sup> |
| Administrative Procedures | | | | | | | | |
| Register Study Visit via Interactive Voice Response System (IVRS/IWRS) | X | X | X | X | X | X | X | |
| Dispense Study Therapy (Open-Label MK-1439A) <sup>e</sup> | X | X | X | X | X | $X^{f}$ | | |
| Assess Subject Eligibility for Study Extension 3 | | | | | | X <sup>g</sup> | | |
| Informed Consent for Study Extension 3 | | | | | | X <sup>g</sup> | | |
| Clinical Procedures/Assessments | | | | | | | | |
| Serious Adverse Events Monitoring | X | X | X | X | X | X | X | X |
| Birth Control Confirmation | X | X | X | X | X | X | X | X |
| Laboratory Procedures/Assessments | | | | | | | | |
| Urine Pregnancy test <sup>h</sup> | X | X | X | X | X | X | X | X |

- a. Subjects who enter study extension 2 are considered enrolled in study extension 2 upon providing written informed consent for study extension 2 at the Week 192 study visit of study extension 1.
- b. The total duration is dependent on when MK-1439A becomes locally available, with a maximum total duration of treatment of 288 weeks. Subjects should discontinue at the next scheduled visit after MK-1439A becomes locally available in the market.
- c. The visit windows are approximately ±14 days for all visits from Week 208 through Week 288. The timing of each visit is relative to the randomization (Day 1) visit. Every attempt must be made to keep subjects on schedule.
- d. The visit window for the post-study 14-day follow-up visit is approximately -2 to 0 days.
- e. IVRS/IWRS will be used to allocate drug and to manage distribution of clinical supplies.
- f. Study drug for extension 3 will be dispensed at Week 288, if subject is continuing into extension 3.
- g. If the subject is eligible and elects to enter study extension 3, he/she will be considered to have completed study extension 2 and will, after providing informed consent, immediately enter study extension 3 and be dispensed MK-1439A.
- h. For women of childbearing potential.

**Protocol/Amendment No.:** 021-09

# Flow Chart D (Study Extension 3): Week 304 Through Up to Week 384 Plus 14 Days Follow-up

| Visit Number/Title | 26ª | 27 | 28 | 29 | 30 | 31 | U (Early<br>Discontinuation) | 99 |
|---|---|---|---|---|---|---|---|---|
| Trial Period | | | - | Γreatn | nent <sup>b,c</sup> | | | |
| TRIAL PROCEDURES | WK<br>304 | | | | WK<br>368 | | At time of Discontinuation | Post-study<br>14-day follow-up <sup>d</sup> |
| Administrative Procedures | | | | | | | | |
| Register Study Visit via Interactive Voice Response System (IVRS/IWRS) | X | X | X | X | X | X | X | |
| Dispense Study Therapy (Open-Label MK-1439A) <sup>e</sup> | X | X | X | X | X | | | |
| Clinical Procedures/Assessments | | | | | | | | |
| Serious Adverse Events Monitoring | X | X | X | X | X | X | X | X |
| Birth Control Confirmation | X | X | X | X | X | X | X | X |
| Laboratory Procedures/Assessments | | | | | | | | |
| Urine Pregnancy test <sup>f</sup> | X | X | X | X | X | X | X | X |

a. Subjects who enter study extension 3 are considered enrolled in study extension 3 upon providing written informed consent for study extension 3 at the Week 288 study visit of study extension 2.

b. The total duration is dependent on when MK-1439A becomes locally available, with a maximum total duration of treatment of 384 weeks. Subjects should discontinue at the next scheduled visit after MK-1439A becomes locally available in the market.

c. The visit windows are approximately  $\pm 14$  days for all visits from Week 304 through Week 384. The timing of each visit is relative to the randomization (Day 1) visit. Every attempt must be made to keep subjects on schedule.

d. The visit window for the post-study 14-day follow-up visit is approximately –2 to 0 days.

e. IVRS/IWRS will be used to allocate drug and to manage distribution of clinical supplies.

f. For women of childbearing potential.

Protocol/Amendment No.: 021-09

#### 7.0 TRIAL PROCEDURES

#### 7.1 Trial Procedures

The Trial Flow Chart - Section 6.0 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below. It may be necessary to perform these procedures at unscheduled time points if deemed clinically necessary by the investigator.

Furthermore, additional evaluations/testing may be deemed necessary by the investigator and or the Sponsor for reasons related to subject safety. In some cases, such evaluation/testing may be potentially sensitive in nature (e.g., HIV, Hepatitis C, etc.), and thus local regulations may require that additional informed consent be obtained from the subject. In these cases, such evaluations/testing will be performed in accordance with those regulations.

#### 7.1.1 Administrative Procedures

#### 7.1.1.1 Informed Consent

The investigator or qualified designee must obtain documented consent from each potential subject or each subject's legally acceptable representative prior to participating in a clinical trial or Future Biomedical Research.

#### 7.1.1.1.1 General Informed Consent

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the subject before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB/ERC requirements, applicable laws and regulations and Sponsor requirements.

Protocol/Amendment No.: 021-09

# 7.1.1.1.2 Consent and Collection of Specimens for Future Biomedical Research

The investigator or qualified designee will explain the Future Biomedical Research consent to the subject, answer all of his/her questions, and obtain written informed consent before performing any procedure related to Future Biomedical Research. A copy of the informed consent will be given to the subject.

#### 7.1.1.2 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the trial. A review of these criteria should occur at the Screening visit and on the Day 1 visit (prior to randomization). For subjects who wish to continue into study extension 1, the additional inclusion criteria (9 to 12, Section 5.1.2) are to be reviewed at the Week 96 study visit. For subjects who wish to continue into study extension 2, the additional inclusion criteria (13 to 16, Section 5.1.2) are to be reviewed at the Week 192 study visit. For subjects who wish to continue into study extension 3, the additional inclusion criteria (17 to 20, Section 5.1.2) are to be reviewed at the Week 288 study visit.

# 7.1.1.3 Subject Identification Card

All subjects will be given a Subject Identification Card identifying them as participants in a research trial. The card will contain trial site contact information (including direct telephone numbers) to be utilized in the event of an emergency. The investigator or qualified designee will provide the subject with a Subject Identification Card immediately after the subject provides written informed consent.

The subject identification card also contains contact information for the emergency unblinding call center so that a health care provider can obtain information about trial medication/vaccination in emergency situations where the investigator is not available.

# 7.1.1.4 Medical History

A medical history will be obtained by the investigator or qualified designee at the Screening visit. The medical history should include information pertaining to the diagnosis of HIV infection and the year diagnosed. If a subject has previously been diagnosed with any AIDS defining condition, or CD4 <200, the condition as well as a corresponding medical history of Acquired Immune Deficiency Syndrome must be reported. In addition, the subject's history of smoking should be obtained and recorded on the appropriate eCRF.

#### 7.1.1.5 Prior and Concomitant Medications Review

#### 7.1.1.5.1 Prior Medications

08K3V5

The investigator or qualified designee will review prior medication use and record all medication taken by the subject within 30 days before starting the study.

Protocol/Amendment No.: 021-09

Investigational agents must be discontinued 30 days prior to receiving study therapy.

#### 7.1.1.5.2 Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the subject during the trial.

#### 7.1.1.6 Assignment of Screening Number

All consented subjects will be given a unique screening number that will be used to identify the subject for all procedures that occur prior to randomization or allocation. Each subject will be assigned only one screening number. Screening numbers must not be re-used for different subjects.

The site must access the IVRS/IWRS system to register each screening subject.

Specific details on the screening visit requirements are provided in Section 7.1.5.1.

# 7.1.1.7 Assignment of Randomization Number

All eligible subjects will be randomly allocated and will receive a randomization number. The randomization number identifies the subject for all procedures occurring after randomization. Once a randomization number is assigned to a subject, it can never be reassigned to another subject.

A single subject cannot be assigned more than 1 randomization number.

#### 7.1.1.8 Trial Compliance (Medication/Diet/Activity/Other)

Subject Diary Cards will be used to ensure and document drug compliance for the base study and study extension 1.

On Day 1, the investigator/study coordinator will give the subject a diary card to be completed during the study period. The study coordinator will be responsible for entering the subject's identification (randomization number) before giving the diary card to the subject. The subject should follow the instructions on the diary card for recording all study drugs. Aside from the initial information entered by the study coordinator, only the subject should enter information on the diary card. The subject is to return the completed diary card at each scheduled visit. The study coordinator will be responsible for reviewing the diary card for completeness and accuracy with the subject. Only the subject shall make any changes to the entries on the card. The subject will initial the card to confirm that the information is accurate. The study coordinator will be responsible for transferring the appropriate information from the diary card onto the appropriate case report form.

Rigorous monitoring is especially important during the early part of the study, specifically between the Day 1 and Week 4 visits to ascertain if there are problems with non-compliance

Protocol/Amendment No.: 021-09

as early as possible, to access whether the subject is taking study medication as directed and to ensure that subjects experiencing difficulties are re-educated, as appropriate.

Subject Medication Diary will not be used during study extension 2 or study extension 3. Sites are responsible for source documentation of drug accountability.

Interruptions from the protocol specified treatment plan that are expected to be 7 days or greater due to non-compliance require consultation between the investigator and the Sponsor and written documentation of the collaborative decision on subject management.

# 7.1.1.9 Patient-Reported Outcomes

Subjects will complete the WPAI at Day 1, Weeks 4, 8, 16, and 48 or at the Early Discontinuation visit if the subject discontinues from the study early.

# Work Productivity and Activity Impairment Questionnaire

This WPAI is a validated 6-item questionnaire that was created as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to general health or a specific health problem. The questionnaire utilizes a one-week recall period. The measure assesses the quantitative impact of health conditions on loss of time and impaired productivity for functional activities such as workfor-pay, school work, and work around the house. The WPAI has been used in studies of HIV-infected patients.

#### Administration

Subjects are to complete the questionnaire on their own at the site using an electronic data capture tool at the beginning of the appropriate study visit (see trial flow chart). Every attempt should be made for the subjects to complete the questionnaire prior to receiving study treatment, discussing any medical conditions with the study personnel, or receiving any medical results. Subjects will be eligible to complete the questionnaire only if language translations are available in the subject's native language.

#### 7.1.2 Clinical Procedures/Assessments

#### 7.1.2.1 Physical Examination

All physical examinations should be performed as indicated in the Trial Flow Charts (Section 6.0). All physical examinations must be performed by the principal investigator or subinvestigator (physician, physician assistant or nurse practitioner).

A complete (full) physical examination (including vital signs [weight, pulse, respiratory rate, blood pressure, and body temperature]) must be obtained at the Screening visit. A complete physical examination generally includes the following assessments: general appearance, head, eyes, ears/nose/ throat, neck, lymph nodes, skin, lungs, heart, abdomen,

Protocol/Amendment No.: 021-09

musculoskeletal, and neurologic evaluations. Breast, rectal, and genitourinary/pelvic exams should be performed when clinically indicated.

Physical examinations after the Screening visit will be directed exams and will include vital signs. Any significant changes between the Screening and Day 1 visits should be noted in the Medical History eCRF at Day 1. Any significant changes in the physical examination after receiving study therapy at Day 1 must be reported as adverse events and entered on the adverse event eCRF. If the subject is discontinued for any reason during the treatment phase, every attempt should be made to perform a final physical examination.

# 7.1.2.2 Height Assessment

The subject's height should be assessed as indicated in the Trial Flow Chart (Section 6.0). If height is measured after the Screening visit, the site should indicate whether or not the result is clinically significant and the result should be documented in the subject's chart. If the result is clinically significant, it should be captured as an adverse event on the eCRF.

# 7.1.2.3 Vital Signs and Weight

Vital signs, including pulse rate, respiratory rate, blood pressure and body temperature, and weight should be assessed as indicated in the Trial Flow Charts (Section 6.0). Subjects should be resting in a semi-recumbent position for at least 10 minutes prior to having vital sign measurements obtained.

<u>Note</u>: Oral temperatures should be taken. If an oral temperature measurement is not possible, a tympanic, rectal, or axillary temperature measurement may be taken and should be recorded appropriately.

After the Screening visit, the site should indicate whether or not the result is clinically significant and document in the subject's chart. If any result is clinically significant, it should be captured as an adverse event on the eCRF.

#### 7.1.2.4 12-Lead ECG (performed locally)

A local 12-Lead ECG should also be performed prior to the subject's first dose of study medication (within 7 days prior to the Study Day 1 visit), as indicated in the Trial Flow Chart A (Section 6.0), and any abnormalities documented. Results <u>must be</u> available prior to subject randomization. Subjects should be resting in a semi-recumbent position for at least 10 minutes prior to having ECG readings obtained. Clinically significant findings from the pre-Day 1/Day 1 ECG must be documented in the subject's chart and captured in the medical history eCRF.

If an ECG is performed for any medical reason while patient is on the study treatment, or during the follow-up period, any clinically significant changes compared with the Day 1 ECG must be captured as AEs on the eCRF and documented in the subject's chart.

Protocol/Amendment No.: 021-09

#### 7.1.2.5 Adverse Events

When evaluating an adverse event, the investigator should document in the eCRF if there is a likely causality relationship to IRIS during the base study.

If a subject has been diagnosed with an AIDS defining condition following randomization, the condition must be reported as an AE.

Due to the use of lamivudine and ATRIPLA<sup>TM</sup> in this trial, subjects should be monitored for symptoms of hyperlactatemia in the base study and in the study extensions.

Details on assessing and recording adverse events can be found in Section 7.2.

# 7.1.2.6 Toxicity Management

Guidelines for grading the severity of laboratory adverse events are based on criteria for grading severity of adverse events (Section 12.8). Decisions to temporarily withhold study therapy because of an adverse experience will be reviewed on a case-by-case basis by the investigator.

The investigator should consider temporarily withholding study therapy if the severity of the adverse experience is Grade 3 or above and/or if clinically indicated. The decision to interrupt study therapy should take into account the subject's baseline laboratory values and any concomitant medication that could be contributory. At the discretion of the investigator, therapy may generally be reinitiated when laboratory abnormalities or clinical adverse events return to near normal or baseline values.

If the adverse experience is considered serious and may have been caused by study medication (as defined in Section 7.2.4) or if re-exposure to the test drug poses additional potential significant risk to the subject, then the rechallenge must be approved in advance by the MSD Clinical Director or Designee and, if required, by the Independent Ethics Committee/Institutional Review Board and a rechallenge consent is needed prior to reinitiation of study therapy. If advance approval of rechallenge is not required by local regulations, the IEC/IRB will receive notification for information only.

If, after re-initiation of study therapy, there is a recurrence of the laboratory abnormality or clinical adverse event, consideration should be given to permanently discontinuing all study therapy. Whenever study drugs are interrupted, the MSD Clinical Director or Designee should be notified.

#### 7.1.2.7 Birth Control Confirmation

Care must be taken to avoid pregnancy in female subjects of childbearing potential and in the female partners of childbearing potential of male subjects.

Site personnel must confirm that subjects and their partner(s) are using acceptable methods of contraception. This confirmation must be documented in the subject's chart.

Protocol/Amendment No.: 021-09

# 7.1.3 Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below. The total amount of blood/tissue to be drawn/collected over the course of the trial (from pre-trial to post-trial visits), including approximate blood/tissue volumes drawn/collected by visit and by sample type per subject can be found in Section 12.4.

# 7.1.3.1 Serum /Urine Pregnancy Test

For women of childbearing potential, serum pregnancy is to be done at the Screening visit, and urine pregnancy is to be done at the Day 1 visit prior to randomization. Urine pregnancy tests must also be subsequently done at each study visit (except at Virologic Failure Confirmation) including the Early Discontinuation Visit (if applicable) and 14-day Follow-up visits in both the base study and the study extensions. Results must be documented in the subject's chart. A subject found to be pregnant must be discontinued from the study.

# 7.1.3.2 Laboratory Safety Evaluations (Hematology, Chemistry and Others)

Laboratory tests (hematology, chemistry and other) which are to be performed during the base study and study extension 1 are specified in Table 4.

Table 4 Laboratory Tests

| Hematology | Chemistry <sup>9</sup> | Other |
|---|---|---|
| Hematocrit | Aspartate aminotransferase (AST, SGOT) | Prothrombin time (PT) <sup>3</sup> |
| Hemoglobin | Alanine aminotransferase (ALT, SGPT) | Activated partial thromboplastin time (APTT) <sup>3</sup> |
| Platelet count | Alkaline phosphatase | International Normalized Ratio (INR) <sup>3</sup> |
| Red Blood Cell Count | Creatine Kinase | Hepatitis B Virus surface antigen <sup>3</sup> |
| Erythrocyte Mean corpuscular volume | Total Bilirubin | Hepatitis B Virus surface antibody <sup>3</sup> |
| White Blood Cell Count (Total and Differential) | Direct Bilirubin | Hepatitis B e-Antigen <sup>3</sup> |
| CD4% and Absolute CD4/<br>Lymphocytes | Indirect Bilirubin | Hepatitis C Antibody <sup>3</sup> |
| CD8% and Absolute<br>CD8/Lymphocytes | Amylase | Plasma hepatitis C virus PCR quantitative <sup>4</sup> |
| CD4/CD8 ratio | Lipase | Enzyme immunoassay HIV antibody (with confirmation WB) <sup>3</sup> |
| | Glucose, fasting <sup>1</sup> | HIV viral RNA Quantification |
| | Glucose, non-fasting <sup>2</sup> | Serum β-human chorionic gonadotropin (hCG) test <sup>5</sup> |
| | Blood Urea Nitrogen | Urine β-human chorionic gonadotropin (hCG) test <sup>6</sup> |
| | Creatinine <sup>8</sup> | HIV Viral resistance <sup>7</sup> |
| | Calcium | |

**Protocol/Amendment No.:** 021-09

| Hematology | Chemistry <sup>9</sup> | Other |
|------------|-------------------------------------------|-------|
| | Phosphorus | |
| | Magnesium | |
| | Protein | |
| | Albumin | |
| | Sodium | |
| | Potassium | |
| | Chloride | |
| | Bicarbonate | |
| | High density lipoprotein cholesterol | |
| | (HDL-C) (Fasting <sup>1</sup> ) | |
| | Low-density lipoprotein cholesterol | |
| | (LDL-C) (fasting <sup>1</sup> ) | |
| | Triglycerides (fasting <sup>1</sup> ) | |
| | Total Cholesterol (fasting <sup>1</sup> ) | |

<sup>1.</sup> Perform at Randomization (Day 1), and the Weeks 24, 48, and 96 visits in base study; and at the Week 148 and 192 visits in study extension 1. Subjects should be fasting for 8 hours.

- 3. Perform at the screening visit only.
- 4. If the result of the Hepatitis C Antibody testing is positive, then a plasma hepatitis C virus PCR quantitative test will also be performed.
- 5. Serum  $\beta$  hCG test at the Screening visit to be performed by central laboratory.
- 6. Urine  $\beta$  hCG test to be performed at the investigator site at Day 1 and every study visit thereafter.
- 7. Collect plasma samples at the Screening visit, all scheduled study visits in the base study (except the Day 1 and Post-Study 14-day follow-up visit), the Virologic Failure confirmation visit, and the Early Discontinuation visit (if not collected at Virologic Failure confirmation visit). In study extension 1, sample will be collected at the Virologic Failure Confirmation visit and at the Early Discontinuation Visit (if not already obtained at Virologic Failure Confirmation visit). The samples will be tested as specified in Section 7.1.3.5 Viral Resistance Testing.
- 8. Creatinine clearance will be computed at every visit by the central laboratory and provided to the site in the report that the site receives from the central laboratory
- 9. Sample taken at virologic failure confirmation visits for creatinine clearance only.

# 7.1.3.3 HIV/ Hepatitis Screening

At the Screening visit, serum HIV/Hepatitis screening tests will be performed including: Enzyme immunoassay HIV antibody (with confirmation WB), serum Hepatitis B surface antigen, serum Hepatitis B surface antibody, serum Hepatitis B e-antigen and serum Hepatitis C antibody. A plasma hepatitis C virus PCR quantitative test will be performed if the Hepatitis C antibody test is positive.

#### 7.1.3.4 Virology Test

Plasma HIV-1 RNA quantification will be performed at all visits in the base study and study extension 1. The testing will be performed at the central laboratory using the Abbott RealTime HIV-1 assay.

#### 7.1.3.5 Viral Resistance Testing

Blood samples will be collected for genotypic HIV viral resistance testing at the Screening visit to determine MK-1439, efavirenz, emtricitabine, tenofovir, and lamivudine resistance. Additional resistance testing on screening samples may be performed. In the base study, blood samples will also be collected for potential HIV viral resistance testing at all scheduled

<sup>2.</sup> Perform at the Screening and Randomization visits, the Week 4, 8, 16, 36, 60, 72 and 84 visits in base study; in study extension 1 at the Week 100, 116, 132, 164 and 180 visits; and the 14-day follow-up visit.

Protocol/Amendment No.: 021-09

study visits (except the Day 1 and Post-Study 14-day follow-up visit), the Virologic Failure Confirmation visit and at the Early Discontinuation Visit (if not already obtained at Virologic Failure Confirmation visit). In study extension 1, resistance sample will be collected at the Virologic Failure Confirmation Visit and at the Early Discontinuation Visit (if not already obtained at Virologic Failure Confirmation Visit). All resistance testing in the base study and in study extension 1 will be performed by the central laboratory.

#### **7.1.3.6 CD4 Cell Counts**

CD4 cell count (absolute and percentage) will be determined at Screening, Day 1, and at the Week 8, 24, 48, 72, and 96 visits in the base study; for subjects who continue into study extension 1, CD4 cell count will also be determined at the Week 100, 148, and 192 visits. The testing (in the base study and study extension 1) will be performed at the central laboratory using a commercially available assay.

#### 7.1.3.7 Pharmacokinetic/Pharmacodynamic Evaluations

MK-1439 population PK samples will be collected from all subjects as outlined in Table 5. The exact time the dose of study medication (Bottle A) was taken prior to the sample collection will be recorded on the appropriate eCRF. The type of meal (full, medium, light or no meal) consumed with the last dose of study medication (Bottle A) prior to the collection of the PK sample will also be recorded on the appropriate eCRF. The type of meal is defined as the following:

- No Meal the subject did not have a meal
- Light Meal the subject consumed a snack (less than 250 calories)
- Medium Meal the subject consumed a small meal (from 250 to 750 calories)
- Full Meal the subject consumed a large meal (greater than 750 calories)

Note: At Week 24 (Visit 6) and Week 48 (Visit 8), 2 PK samples will be collected, one predose and one 0.5-2.0 hours post-dose. Subjects should be fasting for the collection of both samples. Subjects will be given their dose of Bottle A in the office following the collection of the pre-dose sample and may stay in the office or return to the office for the collection of the post-dose sample.

Protocol/Amendment No.: 021-09

Table 5 Pharmacokinetic Sampling Timepoints

| Visit<br>Number | Study<br>Day/Week | Time Relative to Bottle A Dose<br>(MK-1439 or placebo) |
|---|---|---|
| 2 | Day 1 | Sample to be collected predose |
| 3 | Week 4 | Sample to be collected predose |
| 4 | Week 8 | Sample to be collected pre or postdose |
| 6 | Week 24 | Sample to be collected predose <u>and</u> within 0.5 to 2 hours postdose (Subject should remain fasting until the postdose PK sample is collected). |
| 8 | Week 48 | Sample to be collected predose <u>and</u> within 0.5 to 2 hours postdose (Subject should remain fasting until the postdose PK sample is collected). |

Sample collection, storage and shipment instructions for the PK samples will be provided in the operations/laboratory manual.

#### 7.1.3.8 Future Biomedical Research

The following specimens are to be obtained as part of Future Biomedical Research:

- Leftover DNA for future use
- Plasma for future biomedical research

#### 7.1.4 Other Procedures

#### 7.1.4.1 Withdrawal/Discontinuation

When a subject discontinues/withdraws from participation in the trial, all applicable activities scheduled for the Early Discontinuation Visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 - Assessing and Recording Adverse Events. In addition, all investigative products must be retrieved from the subject.

#### 7.1.4.1.1 Withdrawal From Future Biomedical Research

Subjects may withdraw their consent for Future Biomedical Research and have their specimens and all derivatives destroyed. Subjects may withdraw consent at any time by

**Protocol/Amendment No.:** 021-09

contacting the principal investigator for the main trial. If medical records for the main trial are still available, the investigator will contact the Sponsor using the designated mailbox (clinical.specimen.management@MSD.com), and a form will be provided by the Sponsor to obtain appropriate information to complete specimen withdrawal. Subsequently, the subject's specimens will be removed from the biorepository and be destroyed. A letter will be sent from the Sponsor to the investigator confirming the destruction. It is the responsibility of the investigator to inform the subject of completion of destruction. Any analyses in progress at the time of request for destruction or already performed prior to the request being received by the Sponsor will continue to be used as part of the overall research trial data and results. No new analyses would be generated after the request is received.

In the event that the medical records for the main trial are no longer available (e.g., if the investigator is no longer required by regulatory authorities to retain the main trial records) or the specimens have been completely anonymized, there will no longer be a link between the subject's personal information and their specimens. In this situation, the request for specimen destruction cannot be processed.

# 7.1.4.2 Blinding/Unblinding

Procedures for blinding and unblinding apply only to the base study; treatment during the study extensions is open-label.

STUDY TREATMENT IDENTIFICATION INFORMATION IS TO BE UNMASKED ONLY IF NECESSARY FOR THE WELFARE OF THE SUBJECT. EVERY EFFORT SHOULD BE MADE NOT TO UNBLIND THE SUBJECT UNLESS NECESSARY.

For emergency situations where the investigator or subinvestigator needs to identify the drug used by a subject and/or the dosage administered in case of emergency, he/she will contact the emergency unblinding call center by telephone and make a request for emergency unblinding. As requested by the investigator or subinvestigator the emergency unblinding call center will provide the information to him/her promptly and report unblinding to the sponsor. The emergency unblinding call center will make a record promptly however, the investigator or subinvestigator must enter the intensity of the adverse experiences observed, their relation to study drug, the reason thereof, etc., in the medical chart etc., before unblinding is performed.

Additionally, the investigator must go into the IVRS system and perform the unblind in the IVRS system to update drug disposition. In the event that the emergency unblinding call center is not available for a given site in this trial, IVRS/IWRS should be used for emergency unblinding in the event that this is required for subject safety.

Study treatment identification information is to be unmasked ONLY if necessary for the welfare of the subject. Every effort should be made not to unblind the subject unless necessary.

Protocol/Amendment No.: 021-09

In the event that unblinding has occurred, the circumstances around the unblinding (eg, date, reason and person performing the unblinding) must be documented promptly, and the Sponsor Clinical Director notified as soon as possible. Once an emergency unblinding has taken place, the principal investigator, site personnel, and Sponsor personnel may be unblinded so that the appropriate follow-up medical care can be provided to the subject.

# 7.1.4.3 Calibration of Equipment

The investigator or qualified designee has the responsibility to ensure that any device or instrument used for a clinical evaluation/test during a clinical study that provides information about inclusion/exclusion criteria and/or safety or efficacy parameters shall be suitably calibrated and/or maintained to ensure that the data obtained is reliable and/or reproducible. Documentation of equipment calibration must be retained as source documentation at the study site.

Please refer to the central laboratory manuals for equipment requirements and necessary maintenance or calibration.

# 7.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

# **7.1.5.1** Screening

Written informed consent/assent must be obtained from the subject prior to performing any study-specific procedures. Potential subjects will be evaluated to determine if they fulfill the Inclusion/Exclusion entry requirements as set forth in Section 5.1. The investigator will discuss with each potential subject the study, its requirements, and its restrictions. The study screening period is 45 days.

- All procedures listed for the Screening visit (Visit 1) in the Trial Flow Chart (Section 6.0) must be completed and the subjects eligibility confirmed by the investigator prior to the subject's randomization and drug administration on Day 1.
- Blood will be collected for safety laboratory evaluations, hemostatic function tests, HIV/Hepatitis Screen, HIV-1 RNA quantification, CD4 cell counts, and viral resistance testing. These samples will be sent to the appropriate central laboratory(ies) following the procedure(s) set forth in the manual(s).
- Female subjects of childbearing potential will have a serum pregnancy test (hCG) collected at the screening visit. Women who are found to be pregnant will be excluded from the study.
- Subjects will be instructed about the restrictions for concomitant medications, as noted in Section 5.5.

**Protocol/Amendment No.:** 021-09

• Subjects will be given a study participation identification card. The card will contain contact information (including direct telephone numbers) to be utilized in the event of an emergency.

# 7.1.5.2 Treatment Visits in Base Study (Visit 2 to 12)

#### Randomization Day 1 (Visit 2)

- Procedures listed for Day 1 (Visit 2) on the Trial Flow Chart A (Section 6.0) should be performed prior to the subject's randomization and drug administration on Day 1, unless otherwise specified.
- For a female subject who is of childbearing potential, a urine pregnancy test will be performed at the site prior to study drug initiation. If the urine pregnancy test result is negative and the subject meets the other criteria, the subject will be eligible for randomization and the remainder of the pre-treatment (Day 1) testing/procedures will be performed. If the urine pregnancy test result is positive, the subject must not be randomized.
- Fasting blood will be collected for safety laboratory evaluations, HIV-1 RNA quantification, CD4 cell counts, and PK measurements. These samples will be sent to the appropriate central laboratory(ies) following the procedure(s) set forth in the manual(s).
- Following completion of the Day 1 pre-treatment procedures and confirmation of eligibility, the site pharmacist or study coordinator will contact the IVRS/IWRS for assignment of the drug to be administered. Sites should not call IVRS/IWRS for drug administration until the subject has met all criteria for the study and are ready to receive the first dose of study medication on Day 1.
- Randomized subjects will receive a 4-week supply of study medication (1 bottle each labeled A and B) on Day 1 (Visit 2). Subjects will be instructed to take their first dose of all study medication on the same day as the Day 1 study visit.
- The investigator/study coordinator will give the subject a study medication diary to be completed starting on Day 1 and continuing through the treatment period. The site must ensure that the subject is properly trained and comfortable with completing the medication diary prior to leaving the clinic.

# **Drug Administration**

Subjects will be dispensed study drug as outlined in Table 6 for the base study.

Protocol/Amendment No.: 021-09

Table 6 Study Drug Bottle (A and B) Components

| Bottle Label | Component |
|--------------|---------------------|
| Bottle A | MK-1439A or placebo |
| Bottle B | ATRIPLA™ or placebo |

# Subjects will be instructed to take the study medication as follows:

All Subjects will take one tablet once-daily from each of the bottles as follows:

#### Bottle A (MK-1439A or placebo):

Subjects will be instructed to take one tablet from Bottle A once a day (q.d.) orally, with or without food at approximately the same time each day. Tablets from Bottle A <u>must</u> be kept in the bottle prior to taking study medication since the formulation being used in this study is moisture sensitive.

# Bottle B (ATRIPLA<sup>TM</sup> or placebo):

Subjects will be instructed to take one tablet from Bottle B once a day (q.d.) orally, at bedtime, on an empty stomach.

Note: Study medication should be taken directly from the study bottle.

#### Week 4 (Visit 3) to Week 96 (Visit 12)

- All procedures for treatment Week 4 (Visit 3) to Week 96 (Visit 12) listed on the Trial Flow Chart A (Section 6.0) should be performed.
- Blood will be collected for safety laboratory evaluations, HIV-1 RNA quantification, CD4 cell counts, HIV viral resistance and PK measurements at the time points specified on the Trial Flow Chart. These samples will be sent to the appropriate central laboratory(ies) following the procedure(s) set forth in the manual(s).
- For a female subject who is of childbearing potential, a urine pregnancy test will be performed at all study visits. If the urine pregnancy test result is positive, the subject must be discontinued.
- Subjects will be required to fast for at least 8 hours prior to study visits at Weeks 24, 48, and 96.
- All bottles of study drug will be returned to the study coordinator at each visit, at which time the drug supplies for the following time period will be dispensed. The number of

Protocol/Amendment No.: 021-09

tablets remaining in the bottle will be counted and recorded in the source documentation. The primary source of adherence data, however, will be the subjects study medication diary.

- Subjects will receive a 4-week supply of study drug (1 bottle each labeled A and B) at Week 4 (Visit 3); an 8-week supply (2 bottles each labeled A and B) at Week 8 (Visit 4) and Week 16 (Visit 5); and a 12-week supply (3 bottles each labeled A and B) at each visit from Week 24 (Visit 6) through Week 84 (Visit 11).
- At Week 96 (Visit 12), subjects who continue into study extension 1 will receive a 4-week supply of unblinded study drug: this will consist, for all subjects, of MK-1439A, packaged in a single bottle labeled 'Bottle C'.
- At each treatment visit, the study coordinator and subject will review the study medication diary information.

# 7.1.5.3 Treatment Visits in Study Extension 1 (Visit 13 to Visit 19)

- All procedures listed in the Trial Flow Chart B (Section 6.0) should be performed, as applicable to each study visit, including collection of blood and urine (urine only for female subjects of childbearing potential) for laboratory evaluations.
- Subjects will be required to fast for at least 8 hours prior to the Week 148 (Visit 16) and Week 192 (Visit 19) visits.
- In study extension 1, subjects will receive a 16-week supply of MK-1439A at each study visit through Week 164 (Visit 17) and a 12-week supply of MK-1439A at Week 180 (Visit 18). Subjects continuing into study extension 2, if applicable, will receive a 16-week supply of study drug for study extension 2 at Week 192 (Visit 19).
- All bottles of study drug will be returned to the study coordinator at each visit, at which time the drug supplies for the following time period will be dispensed (except for Week 192 for subjects not continuing into extension 2). The number of tablets remaining in the bottle will be counted and recorded in the source documentation. The primary source of adherence data, however, will be the subject's study medication diary.
- At each visit, the study coordinator and subject will review the study medication diary information.

# 7.1.5.4 Treatment Visits in Study Extension 2 (Visit 20 to Visit 25)

• All procedures for Study Week 208 (Visit 20), Week 224 (Visit 21), Week 240 (Visit 22), Week 256 (Visit 23), Week 272 (Visit 24), and Week 288 (Visit 25) listed on Study Flow Chart C (Section 6.0) should be performed.

Protocol/Amendment No.: 021-09

• For a female subject who is of childbearing potential, a urine pregnancy test will be performed at all study visits. If the urine pregnancy test result is positive, the subject must be discontinued.

- All bottles of study drug will be returned to the study coordinator at each visit, at which time the drug supplies for the following time period will be dispensed. The number of tablets remaining in the bottle will be counted and recorded in the source documentation. Only first dose, last dose, overdose (if applicable) and study drug interruption (if applicable) due to any toxicity, ECI or (S)AE will be collected in the database.
- Site staff will access the IVRS/IWRS for registration of visits.
- In study extension 2, starting at Week 192 (Visit 19), subjects will receive a 16-week supply of MK-1439A at each study visit through Week 272 (Visit 24), as applicable. Subjects continuing into study extension 3, if applicable, will receive a 16-week supply of study drug for study extension 3 at Week 288 (Visit 25).

# 7.1.5.5 Treatment Visits in Study Extension 3 (Visit 26 to Visit 31)

- All procedures for Study Week 304 (Visit 26), Week 320 (Visit 27), Week 336 (Visit 28), Week 352 (Visit 29), Week 368 (Visit 30), and Week 384 (Visit 31) listed on Study Flow Chart D (Section 6.0) should be performed.
- For a female subject who is of childbearing potential, a urine pregnancy test will be performed at all study visits. If the urine pregnancy test result is positive, the subject must be discontinued.
- All bottles of study drug will be returned to the study coordinator at each visit, at which time the drug supplies for the following time period will be dispensed. The number of tablets remaining in the bottle will be counted and recorded in the source documentation. Only first dose, last dose, overdose (if applicable) and study drug interruption (if applicable) due to any toxicity, ECI or (S)AE will be collected in the database.
- Site staff will access the IVRS/IWRS for registration of visits.
- In study extension 3, starting at Week 288 (Visit 25), subjects will receive a 16-week supply of MK-1439A at each study visit through Week 368 (Visit 30), as applicable.

# 7.1.5.6 Virologic Failure Confirmation Visit - Base Study and Study Extension 1

• When a subject has a virologic failure confirmation visit performed, all procedures for the virologic failure confirmation visit listed on the Trial Flow Charts should be performed.

Protocol/Amendment No.: 021-09

PDVF for this study is defined as one of the following:

1) Confirmed (2 consecutive measures at least one week apart) HIV-1 RNA ≥50 copies/mL after initial response of HIV-1 RNA <50 copies/mL at any time during the study

OR

2) Confirmed (2 consecutive measures at least one week apart) HIV-1 RNA ≥200 copies/mL at Week 24 or Week 36

OR

3) Confirmed (2 consecutive measures at least one week apart) HIV-1 RNA ≥50 copies/mL at Week 48.

The virologic failure confirmation visit should be done between 1 and 4 weeks after the first measurement of HIV-1 RNA  $\geq$ 50 copies/ml.

Subjects should be discontinued, regardless of compliance with study therapy, if they meet the protocol-defined virologic failure criteria.

# 7.1.5.7 Early Discontinuation Visit - Base Study, Study Extension 1, Study Extension 2, and Study Extension 3

• When a subject discontinues/withdraws from participation in the trial, all procedures for the Early Discontinuation visit listed on the Trial Flow Charts should be performed.

At a minimum, the following information should be collected when a subject discontinues:

- o The reason the subject discontinued
- o The date of the last dose of study medications from the trial
- The date of the last assessment and/or contact
- o All adverse events (including serious adverse events) in the base study and study extension 1
- Only serious adverse events in study extension 2 and study extension 3. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 Assessing and Recording Adverse Events.
- Subjects who discontinue early from the study are expected to return for a 14-day post therapy follow-up visit.
**Protocol/Amendment No.:** 021-09

## 7.1.5.8 Post-Trial (Base Study and Study Extensions)

• Following the completion of study therapy in the base study (at 96 weeks) or in the study extensions (at 192, 288, or 384 weeks) or in the event of early discontinuation, subjects will be required to return to the clinic approximately 14 days after the last dose of study drug for the post-study visit as outlined in the Trial Flow Charts (Section 6.0).

• If the post-study visit occurs less than 14 days after the last dose of study drug, a subsequent follow-up phone call should be made at 14 days post the last dose of study drug to determine if any adverse events have occurred since the post-study clinic visit.

### 7.2 Assessing and Recording Adverse Events

An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.

Changes resulting from normal growth and development that do not vary significantly in frequency or severity from expected levels are not to be considered adverse events. Examples of this may include, but are not limited to, teething, typical crying in infants and children and onset of menses or menopause occurring at a physiologically appropriate time.

Sponsor's product includes any pharmaceutical product, biological product, device, diagnostic agent or protocol-specified procedure, whether investigational (including placebo or active comparator medication) or marketed, manufactured by, licensed by, provided by or distributed by the Sponsor for human use.

Adverse events may occur during clinical trials, or as prescribed in clinical practice, from overdose (whether accidental or intentional), from abuse and from withdrawal.

All adverse events that occur after the consent form is signed but before treatment allocation/randomization must be reported by the investigator if they cause the subject to be excluded from the trial, or are the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure. From the time of treatment allocation/randomization through 14 days following cessation of treatment, all adverse events must be reported by the investigator during the base study and study extension 1 as specified in Section 2. During study extension 2 and study extension 3, serious adverse events must be reported by the investigator as specified in Section 2; and if an investigator chooses to report a non-serious adverse event (NSAE), it should be submitted using the same process used to submit NSAEs in the base study and

Protocol/Amendment No.: 021-09

study extension 1. Such events will be recorded at each examination on the Adverse Event case report forms/worksheets. The reporting timeframe for adverse events meeting any serious criteria is described in section 7.2.3.1. The investigator will make every attempt to follow all subjects with non-serious adverse events for outcome.

Electronic reporting procedures can be found in the EDC data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent).

# 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor

In this trial, an overdose is any dose higher than twice the recommended daily dose in a calendar day.

If an adverse event(s) is associated with ("results from") the overdose of Sponsor's product or vaccine, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.

If a dose of Sponsor's product or vaccine meeting the protocol definition of overdose is taken without any associated clinical symptoms or abnormal laboratory results, the overdose is reported as a non-serious Event of Clinical Interest (ECI), using the terminology "accidental or intentional overdose without adverse effect."

All reports of overdose with and without an adverse event must be reported within 24 hours to the Sponsor either by electronic media or paper. Sponsor Contact information can be found in the Investigator Trial File Binder (or equivalent).

## 7.2.2 Reporting of Pregnancy and Lactation to the Sponsor

Although pregnancy and lactation are not considered adverse events, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject (spontaneously reported to them) that occurs during the trial.

Pregnancies and lactations that occur after the consent form is signed but before treatment allocation/randomization must be reported by the investigator if they cause the subject to be excluded from the trial, or are the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure. Pregnancies and lactations that occur from the time of treatment allocation/randomization through 14 days following cessation of Sponsor's product must be reported by the investigator. All reported pregnancies must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

**Protocol/Amendment No.:** 021-09

Such events must be reported within 24 hours to the Sponsor either by electronic media or paper. Electronic reporting procedures can be found in the EDC data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent).

#### 7.2.3 Immediate Reporting of Adverse Events to the Sponsor

#### 7.2.3.1 Serious Adverse Events

A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that:

- Results in death;
- Is life threatening;
- Results in persistent or significant disability/incapacity;
- Results in or prolongs an existing inpatient hospitalization;
- Is a congenital anomaly/birth defect;
- Is an other important medical event

**Note:** In addition to the above criteria, adverse events meeting either of the below criteria, although not serious per ICH definition, are reportable to the Sponsor in the same timeframe as SAEs to meet certain local requirements. Therefore, these events are considered serious by the Sponsor for collection purposes.

- Is a cancer;
- Is associated with an overdose.

Refer to Table 7 for additional details regarding each of the above criteria.

For the time period beginning when the consent form is signed until treatment allocation/randomization, any serious adverse event, or follow up to a serious adverse event, including death due to any cause, that occurs to any subject must be reported within 24 hours to the Sponsor if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment allocation/randomization through 14 days following cessation of treatment, any serious adverse event, or follow up to a serious adverse event, including death due to any cause, whether or not related to the Sponsor's product, must be reported within 24 hours to the Sponsor either by electronic media or paper. Electronic reporting procedures can be found in the EDC data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent).

Additionally, any serious adverse event, considered by an investigator who is a qualified physician to be related to the Sponsor's product that is brought to the attention of the investigator at any time outside of the time period specified in the previous paragraph also must be reported immediately to the Sponsor.

Protocol/Amendment No.: 021-09

All subjects with serious adverse events must be followed up for outcome.

#### 7.2.3.2 Events of Clinical Interest

Selected non-serious and serious adverse events are also known as Events of Clinical Interest (ECI) and must be reported to the Sponsor.

For the time period beginning when the consent form is signed until treatment allocation/randomization, any ECI, or follow up to an ECI, that occurs to any subject must be reported within 24 hours to the Sponsor if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment allocation/randomization through 14 days following cessation of treatment, any ECI, or follow up to an ECI, whether or not related to the Sponsor's product, must be reported within 24 hours to the Sponsor, either by electronic media or paper. Electronic reporting procedures can be found in the EDC data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent).

Events of clinical interest for this trial include:

- 1. an overdose of Sponsor's product, as defined in Section 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor, that is not associated with clinical symptoms or abnormal laboratory results.
- 2. an elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing.\*

\*Note: These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology. The trial site guidance for assessment and follow up of these criteria can be found in the Investigator Trial File Binder (or equivalent).

### 7.2.4 Evaluating Adverse Events

An investigator who is a qualified physician will evaluate all adverse events with respect to the elements outlined in Table 7. The investigator's assessment of causality is required for each adverse event. Refer to Table 7 and Appendix 12.8 for additional instructions for evaluating adverse events.

**Protocol/Amendment No.:** 021-09

Table 7 **Evaluating Adverse Events** 

| Maximum | Mild | awareness of sign or symptom, but easily tolerated (for pediatric trials, awareness of symptom, but easily tolerated) |
|---|---|---|
| Intensity | Moderate | discomfort enough to cause interference with usual activity (for pediatric trials, definitely acting like something is wrong) |
| | Severe | incapacitating with inability to work or do usual activity (for pediatric trials, extremely distressed or unable to do usual activities) |
| Seriousness | A serious adverse | event (AE) is any adverse event occurring at any dose or during any use of Sponsor's product that: |
| | †Results in death; or<br>†Is life threatening; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred [Note: This does not include | |
| | adverse event that | , had it occurred in a more severe form, might have caused death.]; or |
| | †Results in a pers | istent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or |
| | | rolongs an existing inpatient hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay, even if the |
| | | a precautionary measure for continued observation. (Note: Hospitalization for an elective procedure to treat a pre-existing condition that has not |
| | | serious adverse event. A pre-existing condition is a clinical condition that is diagnosed prior to the use of an MSD product and is documented in the |
| | patient's medical h | • // |
| | | nomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis); or |
| | | igh not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements); or |
| | | an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection |
| | | lose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. |
| | | medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, |
| | | riate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed |
| D | previously (designated | • 1/ |
| Duration | | d stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units |
| Action taken | Did the adverse ev | ent cause the Sponsor's product to be discontinued? |
| Relationship to | | product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an |
| Sponsor's<br>Product | | a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below |
| rroduct | | Ference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the |
| | available informati | |
| | | on apponents are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and |
| | | ments (in number and/or intensity), the more likely the Sponsor's product caused the adverse event: |
| | Exposure | Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill |
| | Laposure | count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? |
| | Time Course | Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? |
| | | Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? |
| | Likely Cause | Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental factors |

**Protocol/Amendment No.:** 021-09

| Relationship | The following components are to be used to assess the relationship between the Sponsor's product and the AE: (continued) | |
|---|---|---|
| to Sponsor's | Dechallenge | Was the Sponsor's product discontinued or dose/exposure/frequency reduced? |
| Product | | If yes, did the AE resolve or improve? |
| (continued) | | If yes, this is a positive dechallenge. If no, this is a negative dechallenge. |
| | | (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE resolved/improved despite continuation |
| | | of the Sponsor's product; (3) the trial is a single-dose drug trial); or (4) Sponsor's product(s) is/are only used one time.) |
| | Rechallenge | Was the subject re-exposed to the Sponsor's product in this trial? |
| | | If yes, did the AE recur or worsen? |
| | | If yes, this is a positive rechallenge. If no, this is a negative rechallenge. |
| | | (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) the trial is a single-dose drug trial); or |
| | | (3) Sponsor's product(s) is/are used only one time.) |
| | | NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS AND WHICH MAY HAVE BEEN |
| | | CAUSED BY THE SPONSOR'S PRODUCT, OR IF RE-EXPOSURE TO THE SPONSOR'S PRODUCT POSES ADDITIONAL POTENTIAL |
| | | SIGNIFICANT RISK TO THE SUBJECT THEN THE RECHALLENGE MUST BE APPROVED IN ADVANCE BY THE SPONSOR |
| | | CLINICAL DIRECTOR AND IF REQUIRED, BY THE INSTITUTIONAL REVIEW BOARD/INDEPENDENT ETHICS COMMITTEE. IF |
| | | ADVANCED APPROVAL OF RECHALLENGE IS NOT REQUIRED BY LOCAL REGULATIONS, THE IRB/IEC WILL RECEIVE |
| | ~ | NOTIFICATION OF INFORMATION ONLY. |
| | Consistency with | Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Sponsor's product or drug class pharmacology |
| | Trial Treatment | or toxicology? |
| | Profile | |
| | | reported on the case report forms /worksheets by an investigator who is a qualified physician according to his/her best clinical judgment, including |
| consideration of the | | |
| Record one of the | following: | Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Sponsor's product relationship). |
| Yes, there is a reasonable possibility of Sponsor's product relationship. | | There is evidence of exposure to the Sponsor's product. The temporal sequence of the AE onset relative to the administration of the Sponsor's product is reasonable. The AE is more likely explained by the Sponsor's product than by another cause. |
| No, there is not a reasonable | | Subject did not receive the Sponsor's product OR temporal sequence of the AE onset relative to administration of the Sponsor's product is not |
| possibility of Sponsor's product relationship | | reasonable OR the AE is more likely explained by another cause than the Sponsor's product. (Also entered for a subject with overdose without an associated AE.) |

Protocol/Amendment No.: 021-09

### 7.2.5 Sponsor Responsibility for Reporting Adverse Events

All Adverse Events will be reported to regulatory authorities, IRB/IECs and investigators in accordance with all applicable global laws and regulations, i.e., per ICH Topic E6 (R1) Guidelines for Good Clinical Practice.

#### 7.3 TRIAL GOVERNANCE AND OVERSIGHT

## 7.3.1 Scientific Advisory Committee

This trial was developed in collaboration with a Scientific Advisory Committee (SAC). The SAC comprises both Sponsor and non-Sponsor scientific experts who provide input with respect to trial design, interpretation of trial results and subsequent peer-reviewed scientific publications.

#### 7.3.2 Executive Oversight Committee

The Executive Oversight Committee (EOC) comprises members of Sponsor Senior Management. The EOC will receive and decide upon any recommendations made by the eDMC regarding the trial.

## 7.3.3 Data Monitoring Committee

To supplement the routine trial monitoring outlined in this protocol, an external Data Monitoring Committee (DMC) will monitor the interim data from this trial. The voting members of the committee are external to the Sponsor. The members of the DMC must not be involved with the trial in any other way (e.g., they cannot be trial investigators) and must have no competing interests that could affect their roles with respect to the trial. The DMC will include at least 3 clinicians experienced in Infectious Disease and 1 external statistician; this is in addition to the unblinded trial statistician who will be a non-voting member of the committee. The eDMC will monitor the trial at an appropriate frequency, with suggested periodic reviews to occur approximately every 6 months during the base trial; there will be no involvement of the eDMC in the trial extensions. Details regarding the eDMC will be described in a charter document.

The DMC will make recommendations to the EOC regarding steps to ensure both subject safety and the continued ethical integrity of the trial. Also, the DMC will review interim trial results, consider the overall risk and benefit to trial participants (see Section 8.7 - Interim Analyses) and recommend to the EOC if the trial should continue in accordance with the protocol.

Specific details regarding composition, responsibilities, and governance, including the roles and responsibilities of the various members and the Sponsor protocol team; meeting facilitation; the trial governance structure; and requirements for and proper documentation of DMC reports, minutes, and recommendations will be described in a separate charter that is reviewed and approved by the DMC. The DMC will monitor the trial at an appropriate

Protocol/Amendment No.: 021-09

frequency, as described in the detailed DMC charter. The DMC will also make recommendations to the Sponsor protocol team regarding steps to ensure both subject safety and the continued ethical integrity of the trial.

#### 8.0 STATISTICAL ANALYSIS PLAN

This section outlines the statistical analysis strategy and procedures for the study. If, after the study has begun, but prior to any unblinding, changes are made to primary and/or key secondary hypotheses, or the statistical methods related to those hypotheses, then the protocol will be amended (consistent with ICH Guideline E-9). Changes to exploratory or other non-confirmatory analyses made after the protocol has been finalized, but prior to unblinding, will be documented in a supplemental statistical analysis plan (sSAP) and referenced in the CSR for the study. Separate analysis plans (i.e., separate documents from the sSAP) will be developed to detail other planned analyses (analysis of PK data, patientreported outcomes, and future biomedical research). Post hoc exploratory analyses will be clearly identified in the CSR.

The key objectives and hypotheses are to be addressed by the base study (double-blind with active comparator for 96 weeks). Thus, between treatment comparisons that address key efficacy and safety objectives will be limited to data from the base study. Demography, efficacy and safety data from study extension 1 for those subjects who continue into the extension 1 will be summarized separately using descriptive statistics only. Serious adverse event data from study extension 2 and study extension 3 will be summarized separately from data for the base and study extension 1 portions of the study.

#### 8.1 STATISTICAL ANALYSIS PLAN SUMMARY

Key elements of the SAP are summarized below; the comprehensive plan is provided in Sections 8.2 through 8.12.

| Study Design Overview | A Phase III Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-1439A Once-Daily Versus ATRIPLA™ Once-Daily in Treatment-Naïve HIV-1 Infected Subjects |
|---|---|
| Treatment Assignment | Approximately 680 subjects will be randomized in a 1:1 ratio with $\sim$ 340 on MK-1439A and $\sim$ 340 on ATRIPLA <sup>TM</sup> in a double-blind fashion with stratification for screening viral load (HIV RNA $\leq$ 100,000 vs. $>$ 100,000 copies /mL) and chronic hepatitis B and/or C status (yes, no). |
| Analysis Populations | Efficacy: Treatment Full Analysis Set (FAS) |
| | Safety: All Subjects as Treated (ASaT) |
| Primary Endpoints | 1. Proportion of subjects with HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48 |
| | 2. Proportion of subjects with neuropsychiatric AEs in the following categories by Week 48: |
| | o Dizziness |
| | <ul> <li>Sleep disorders and disturbances</li> </ul> |
| | Altered Sensorium |


08K3V5

## **Key Secondary Endpoints**

- 1. Safety and tolerability by Week 48 and Week 96
- 2. Fasting LDL-C as measured by the mean change from baseline at Week 48
- 3. Fasting non-HDL-C as measured by the mean change from baseline at Week 48
- 4. Proportion of subjects with neuropsychiatric AEs in the following categories by Week 48:
  - Depression and suicide/self-injury
  - Psychosis and psychotic disorders
- 5. Proportion of subjects with at least one neuropsychiatric AE in any of the 5 categories of: dizziness, sleep disorders and disturbances, altered sensorium, depression and suicide/self-injury, and psychosis and psychotic disorders.
- 6. Time to discontinuation from study due to an adverse experience
- 7. Change from baseline in CD4 cell count at Week 48 and Week 96
- 8. The proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 96
- 9. The proportion of subjects achieving HIV-1 RNA <40 copies/mL (BLoQ) (by the Abbott RealTime HIV-1 Assay) at Week 48 and Week 96
- 10. PK of MK-1439 and the PK/PD association

## Statistical Methods for Key Efficacy Analyses

The primary hypothesis will be assessed based upon the proportion of subjects maintaining HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48 post-randomization. The Non-Completer=Failure approach (NC=F) as defined by the FDA "snapshot" approach will be used as the primary approach for handling missing data. All missing data will be treated as failures regardless of the reason.

The difference in proportions of subjects with HIV-1 RNA <50 copies/mL between treatment groups and the associated 95% confidence interval will be calculated using the stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of the sample size per arm for each stratum (screening HIV RNA  $\leq$ 100,000 or  $\geq$ 100,000 copies/mL). Chronic hepatitis B or C co-infection is not considered to be associated with virologic response; therefore, stratification by hepatitis B or C status will not be included in the analyses of virologic response.

For the primary hypothesis, MK-1439A will be considered non-inferior to ATRIPLA<sup>TM</sup> if the lower bound of the two-sided 95% confidence interval (CI) for the between treatment difference in proportion of subjects with HIV-1 RNA <50 copies/mL at Week 48 (MK-1439A minus ATRIPLA<sup>TM</sup>) is greater than -10 percentage points (non-inferiority margin). It can be further concluded that MK-1439A is superior to ATRIPLA<sup>TM</sup> if the lower bound of the two-sided 95% CI for the difference in the response rates (MK-1439A minus ATRIPLA<sup>TM</sup>) is greater than zero contingent upon satisfying the multiplicity criteria. A similar approach will be used for the supportive secondary efficacy hypotheses for non-inferiority and superiority at Week 96.

#### Statistical Methods for Key Safety Analyses

Neither stratification factor is considered to be associated with the Tier I safety endpoints; therefore, stratification will not be included in the analyses of Tier I events.

#### Tier I

Neuropsychiatric AEs (primary safety hypothesis):

The treatment differences and the associated 95% confidence intervals will be calculated using the Miettinen and Nurminen method [5]. The treatment differences (95% confidence intervals) will be provided for the proportion of subjects with at least one neuropsychiatric AE in any category as well as at least one AE in each category, and p-values will be provided for dizziness, sleep disorders and disturbances, and altered sensorium. MK-1439A will be considered superior to ATRIPLA<sup>TM</sup> if the upper bound of the two-sided 95% CI for the difference in proportion of subjects with neuropsychiatric AEs (each category separately) by Week 48 (MK-1439A minus ATRIPLA<sup>TM</sup>) is less than zero.

Lipids (secondary safety hypothesis):

The change from baseline in fasting lipids (total cholesterol, LDL-C, non-HDL-C, and triglycerides) will be analyzed using Analysis of Covariance models adjusted by baseline lipid level and treatment group. The treatment differences (95% confidence intervals) will be provided for all lipid parameters, and p-values for between treatment comparisons will be provided for LDL-C and non-HDL-C.

#### Tier I

The treatment differences and the associated 95% confidence intervals will be provided for the percentage of subjects with the following events based on specific AE categories (i.e., Tier-2 events): (1) at least one adverse experience; (2) at least one drug-related adverse experience; (3) at least one serious adverse experience; (4) at least one serious and drug-related adverse experience; (5) discontinued study therapy due to an adverse experience. Other Tier-2 events require a minimum of 4 subjects in at least one treatment group. These analyses will be performed using the Miettinen and Nurminen [5] method, an unconditional, asymptotic method.

#### **Interim Analyses**

No interim analyses for efficacy are planned. However, an external data monitoring committee will convene to review safety data approximately every 6 months during the study.

| Multiplicity | The following hypotheses will be tested sequentially at the one-sided Type 1 error rate of 2.5% (unadjusted for the efficacy hypotheses [#1,7] and after adjusting for interim DMC safety reviews for the safety hypotheses [#2-6]) in the following order: |
|---|---|
| | <ol> <li>Primary efficacy hypothesis testing non-inferiority at Week 48</li> <li>Primary safety hypothesis for dizziness</li> <li>Primary safety hypothesis for sleep disorders and disturbances</li> <li>Primary safety hypothesis for altered sensorium</li> <li>Secondary safety hypothesis for LDL-C</li> <li>Secondary safety hypothesis for non-HDL-C</li> <li>Secondary efficacy hypothesis testing superiority at Week 48</li> </ol> |
| | Testing will stop with the first of these tests failing to reach statistical significance and all subsequent tests would not be considered for statistical significance. In this way, the overall one-sided Type 1 error rate in testing these hypotheses is strongly controlled at a 2.5% level. |
| | Note the secondary efficacy hypotheses testing non-inferiority and superiority at Week 96 are supportive only to the primary and secondary efficacy hypotheses at Week 48 and are not considered in the strong control for the Type 1 error for this study. |
| | There are no other hypotheses that will be tested and analyses associated with objectives without hypotheses will be considered supportive and/or explanatory. |
| Sample Size and Power | The planned sample size is 340 subjects in each treatment group (680 total) to achieve 90% power to demonstrate the primary hypothesis that MK-1439A is non-inferior to ATRIPLA <sup>TM</sup> at an overall one-sided 2.5% alpha level, as measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL at Week 48 (by the Abbott RealTime HIV-1 Assay). The power calculation assumes a true response rate of 80% at Week 48 for both MK-1439A and ATRIPLA <sup>TM</sup> using the NC=F approach as defined by the FDA "snapshot" approach. |

### 8.2 Responsibility for Analyses/In-House Blinding

The statistical analysis of the data obtained from this study will be the responsibility of the Clinical Biostatistics department of the Sponsor.

The base study will be conducted as a double-blind study under in-house blinding procedures; the study extensions, for eligible subjects who elect to continue into the extensions, will be conducted as an open-label study. At Week 48 of the base study, when the primary efficacy hypothesis will be evaluated, a copy of the database will be frozen after medical/scientific review has been completed and data have been declared final and complete. This version of the database will be used for initial regulatory submissions. The study (after Week 48, when longer-term safety and efficacy data will be evaluated) will be unblinded to the Sponsor with the exception of a limited group of Sponsor personnel who will remain blinded at the subject level and continue to be responsible for the integrity of the database for ongoing study management. All Sponsor personnel who are unblinded at the subject level for the base period will be excluded from any future data review at the

Protocol/Amendment No.: 021-09

individual subject level. The Week 96 analysis for the base study will follow the same approach as the Week 48 analysis. For the purpose of the final analysis (after all subjects complete their final visit in the base study), the official clinical database will not be unblinded until medical/scientific review has been completed, and data have been declared final and complete. Results from the Week 96 (base study) and from the study extensions will be presented in separate CSRs (separate from the CSR for the Week 48 analysis of the base study).

The designee/Clinical Biostatistics department will generate the randomized allocation schedule(s) for study treatment assignment. Randomization will be implemented in an IVRS/IWRS.

Treatment-level results of the periodic safety reviews will be provided by the unblinded statistician (external to the Sponsor) to the DMC. Limited additional Sponsor personnel may be unblinded to the treatment-level results of the safety analyses, if required, in order to act on the recommendations of the DMC. The extent to which individuals are unblinded with respect to results of safety reviews will be documented by the unblinded statistician.

The DMC will serve as the primary reviewer of the safety results from this study with respect to the periodic safety reviews and will make recommendations for discontinuation of or modifications to the study to an executive committee of the Sponsor. If the DMC recommends modifications to the design of the protocol or discontinuation of the study, this executive oversight committee (internal to the Sponsor) may be unblinded to results at the treatment level in order to act on these recommendations. Additional logistical details will be provided in the DMC Charter. Key aspects of the periodic safety reviews are described in Section 8.7.

Prior to final study unblinding, the unblinded statistician will not be involved in any discussions regarding modifications to the protocol, statistical methods, identification of protocol violators, or data validation efforts after the initial safety review.

PK data may be unblinded early for the purpose of preparing a population PK model. A separate Modeling and Simulation Plan authored by the department of Quantitative Pharmacology and Pharmacometrics will describe the modeling work to be performed. If early unblinding occurs, a Clinical Research Organization, external to the Sponsor, will perform the modeling. Efficacy and safety data will not be unblinded. Interim data or results will be not shared with the study team prior to study unblinding. No alpha adjustment will be made for this early unblinding for modeling and simulation analysis.

### 8.3 Hypotheses/Estimation

Objectives and hypotheses of the study are stated in Section 2.1.

## 8.4 Analysis Endpoints

Efficacy and safety endpoints for the base study and study extension 1 that will be evaluated for within- and/or between treatment differences are listed below, followed by the descriptions of the derivations of selected endpoints.

## 8.4.1 Efficacy / Pharmacokinetics Endpoints

#### **8.4.1.1** Efficacy Endpoints

An initial description of efficacy measures is provided in Section 4.2.3.

<u>Proportions of Subjects Achieving HIV-1 RNA <50 copies/mL, <40 copies/mL and <200 copies/mL (by the Abbott RealTime HIV-1 Assay)</u>

The proportions of subjects achieving HIV-1 RNA <50 copies/mL (and <40 and <200 copies/mL) will be estimated at each time point. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification of 40 copies/mL, will be used to measure the HIV-1 RNA level in blood samples obtained at each visit.

The primary hypothesis will be assessed based upon the proportion of subjects achieving HIV-1 RNA <50 copies/mL at Week 48.

#### Change from Baseline in CD4 Cell Count

Change from baseline in CD4 cell count will be estimated at each time point at which CD4 cell count is collected with a key interest at Week 48.

For the calculations of change from baseline, baseline measurements are defined as the Day 1 (Randomization) value for each subject. In the rare event when data for this visit are missing, the value obtained at the most recent screening visit will be used as baseline. This rule will also be applied to define the baseline measurements for other laboratory tests.

#### Protocol-Defined Virologic Failure

Subjects with PDVF as defined in Section 4.2.3.1 will be identified and summarized for each treatment group.

## 8.4.2 Safety Endpoints

An initial description of safety measures is provided in Section 4.2.3.

Protocol/Amendment No.: 021-09

## Neuropsychiatric Adverse Events

The following categories of specific neuropsychiatric adverse events will be used to address the primary and secondary safety objectives:

- Dizziness
- Sleep disorders and disturbances
- Altered Sensorium
- Depression and suicide/self-injury
- Psychosis and psychotic disorders

A complete list of the preferred terms (based on MedDRA version 17.0) that will be used to define the neuropsychiatric categories can be found in Section 12.6.

#### Change From Baseline in Fasting Lipids

The change from baseline in fasting lipids (LDL-C, non-HDL-C, total cholesterol, HDL-C, and triglycerides) will be analyzed with primary interest in LDL-C and non-HDL-C.

#### Adverse Experiences

The following clinical and laboratory adverse experiences will be summarized: 1) subjects with at least one adverse experience; 2) subjects with at least one drug-related adverse experience; 3) subjects with at least one serious adverse experience; 4) subjects with at least one serious and drug-related adverse experience; and 5) subjects who discontinued study therapy due to an adverse experience.

#### Time to Discontinuation From Study Due to Adverse Experience

In addition to the counts of subjects who discontinued study therapy due to an adverse experience, the time to discontinuation from study due to an adverse experience will also be estimated.

#### Predefined Limits of Change in Laboratory Parameters

For the summaries of laboratory tests, subjects must have both a baseline and post-randomization on-treatment measurement to be included. Subjects' laboratory values (based on their most abnormal laboratory test values, in the direction of interest, while on study therapy) will be classified as to whether or not they fall outside of the PDLC and are worse in grade (i.e., more abnormal in the direction of interest) than at baseline. The criteria are adapted from DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS, PUBLISH DATE: AUGUST 2009 Version 1 (Section 12.8). A listing of the subjects who meet the criteria will be provided.

Protocol/Amendment No.: 021-09

## 8.5 Analysis Populations

## **8.5.1** Efficacy Analysis Populations

The Full Analysis Set (FAS) population will serve as the primary population for the analysis of efficacy data in this study. The FAS population consists of all randomized subjects who:

- receive at least one dose of study treatment,
- have baseline data for those analyses that require baseline data

Subjects will be included in the treatment group to which they are randomized for the analysis of efficacy data using the FAS population. Details on the approach to handling missing data are provided in Section 8.6 Statistical Methods.

## 8.5.2 Safety Analysis Populations

The ASaT population will be used for the analysis of safety data in this study. The ASaT population consists of all randomized subjects who received at least one dose of study treatment. Subjects will be included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data using the ASaT population. For most subjects this will be the treatment group to which they are randomized. Subjects who take incorrect study treatment for the entire treatment period will be included in the treatment group corresponding to the study treatment actually received. Otherwise, subjects will be included in their randomized treatment group.

At least one laboratory or vital sign measurement obtained subsequent to at least one dose of study treatment is required for inclusion in the analysis of each specific parameter. To assess change from baseline, a baseline measurement is also required.

Details on the approach to handling missing data for safety analyses are provided in Section 8.6 Statistical Methods.

#### **8.6** Statistical Methods

Statistical testing and inference for safety analyses are described in Section 8.6.2. Efficacy results that will be deemed to be statistically significant after consideration of the Type I error control strategy are described in Section 8.8, Multiplicity. Nominal p-values may be computed for other efficacy analyses, but should be interpreted with caution due to potential issues of multiplicity, sample size, etc. Unless otherwise stated, all statistical tests will be conducted at the  $\alpha$ =0.025 (1-sided) level.

The key objectives and hypotheses are to be addressed by the base study (double-blind with active comparator for 96 weeks). Thus, between treatment comparisons that address key efficacy and safety objectives will be limited to data from the base study. Demography, efficacy and safety data from study extension 1, for those subjects who continue into the study extension 1, will be summarized separately using descriptive statistics only. Serious

02-Nov-2022

**Protocol/Amendment No.:** 021-09

adverse event data will be collected and summarized for study extension 2 and study extension 3 separately.

## **8.6.1** Statistical Methods for Efficacy Analyses

## Time Window

Table 8 lists the definition of time windows and the target relative day for the scheduled visits in the study which will be used for all analyses by timepoint. The measurement closest to the target date within a window will be used for analyses at a specific timepoint.

Table 8 Definition of Study Timepoint

| Treatment Phase | Treatment<br>Period | Protocol<br>Time | Day-Range Rules | Target<br>Day <sup>1</sup> | CSR Time <sup>2</sup> |
|---|---|---|---|---|---|
| Pre-treatment | Baseline | Day 1<br>(Baseline) | ≤1 | 1 | Day 1 |
| | | Week 4 | >1 and ≤42 | 29 | Week 4 |
| | | Week 8 | ≥43 and ≤84 | 57 | Week 8 |
| | | Week 16 | ≥85 and ≤140 | 113 | Week 16 |
| | | Week 24 | ≥141and ≤210 | 169 | Week 24 |
| | | Week 36 | ≥211 and ≤294 | 253 | Week 36 |
| Treatment | Double-Blind | Week 48 | ≥295 and ≤378 | 337 | Week 48 |
| | (Base Study) | Week 60 | ≥379 and ≤462 | 421 | Week 60 |
| | | Week 72 | ≥463 and ≤546 | 505 | Week 72 |
| | | Week 84 | ≥547 and ≤630 | 589 | Week 84 |
| | | Week 96 | ≥631 and ≤the last day of double-blind treatment period | 673 | Week 96 |
| | | Week 100 | ≥the first day of open-<br>label extension<br>treatment period and<br>≤756 | 701 | Week 100 |
| | | Week 116 | ≥757 and ≤868 | 813 | Week 116 |
| | Open-label | Week 132 | ≥869 and ≤980 | 925 | Week 132 |
| Treatment | (Study | Week 148 | ≥981 and ≤1092 | 1037 | Week 148 |
| | Extension 1) | Week 164 | ≥1093 and ≤1204 | 1149 | Week 164 |
| | | Week 180 | ≥1205 and ≤1302 | 1261 | Week 180 |
| | | Week 192 | ≥1303 and ≤the last day<br>of open-label<br>extension 1 treatment<br>period | 1345 | Week 192 |

<sup>1</sup> Relative days and target day are counted from the first day of study medication.

<sup>2</sup> The clinical study report (CSR) time is the time label to be used in the analysis tables.

Protocol/Amendment No.: 021-09

## Missing Values

There are 3 types of missing values:

• intermittent missing values due to a missed or skipped visit or due to an inadequate sample;

- non-intermittent missing values due to premature discontinuations because of treatment-related reasons such as, "clinical adverse experience" (regardless of relationship to study drug), "laboratory adverse experience" (regardless of relationship to study drug), and "withdrew based on HIV-1 RNA results";
- non-intermittent missing values due to premature discontinuations because of other reasons which are not related to treatment such as loss to follow-up, protocol violation, subject withdrew consent, etc.

Two approaches will be used to handle missing values (Table 9). The primary approach for the analysis of the proportion of subjects achieving HIV-1 RNA <50 copies/mL is the NC=F approach as defined by the FDA "snapshot" approach. Under this approach, only subjects meeting the following can be classified as virologic success at a given time point: 1) subject is on study-assigned double-blind-treatment, 2) subject has HIV-1 RNA measurement(s) within the time window specified in Table 8, and 3) subject has the measurement closest to the target date of the time point <50 copies/mL. The other subjects, either with an HIV-1 RNA measurement of ≥50 copies/mL or no virologic data within the time window due to intermittent missing or premature discontinuation regardless of reasons, will be considered as failures in the analyses of the proportion of subjects achieving HIV-1 RNA <50 copies/mL at that timepoint.

A second approach, the OF approach will be performed as a sensitivity analysis for the proportion of subjects achieving HIV-1 RNA<50 copies/mL at Week 48. Under this approach, non-intermittent missing data for subjects who prematurely discontinued assigned treatment due to lack of efficacy are considered as failures at timepoints thereafter. Subjects with other reasons for missing data will be excluded from the analyses.

The same approaches as described above will be used for the analysis of the proportion of subjects achieving HIV-1 RNA <40 and <200 copies/mL.

Protocol/Amendment No.: 021-09

Table 9 Summary of the Two Approaches to Handle Missing Values

| | | Non-intermittent Missing<br>Not Related to Treatment | | Non-intermittent Missing<br>Related to Treatment | |
|---|---|---|---|---|---|
| Approaches§ | Intermittent<br>Missing | Success at Study<br>Therapy<br>Discontinuation | Failure at Study<br>Therapy<br>Discontinuation | Study Therapy Discontinuation Due to Clinical/Lab Adverse Experience | Study Therapy<br>Discontinuation<br>Due to Lack of<br>Efficacy |
| OF | Excluded | Excluded | Failures | Excluded | Failures |
| NC=F | Failure | Failures Failures | | Failures Failures | |
| § OF (Observe | d Failure); NC=F | (Non-Completer=Fail | ure) is the primary app | proach. | |

#### Proportion of Subjects Achieving HIV-1 RNA <50 copies/mL

The proportion of subjects achieving HIV-1 RNA <50 copies/mL will be summarized by treatment group at each time point, with primary interest at Week 48. For each time point of interest, the difference in proportions between treatment groups and the associated 95% confidence interval will be calculated using the stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of the sample size per arm for each stratum (screening HIV-1 RNA ≤100,000 copies/mL or HIV-1 RNA >100,000 copies/mL). The study has 2 stratification factors: screening HIV-1 RNA level and chronic hepatitis B or C status. Chronic hepatitis B or C co-infection may be associated with serious liver function abnormalities but is not considered to be associated with virologic response; therefore, stratification by hepatitis B or C status will not be included in the analyses of virologic response.

The NC=F approach as defined by FDA "snapshot" approach will be used as the primary approach to analysis with respect to the proportion of subjects with virologic response (HIV-1 RNA <50 copies/mL). All missing data will be treated as failures regardless of the reason.

To provide a full picture of virologic outcome at a timepoint, subjects who are not classified as virologic success will be further categorized as virologic failure (HIV-1 RNA ≥50 copies/mL) or as having no virologic data at the time window with reasons of 1) discontinued study due to an AE, 2) discontinued study for other reasons (includes withdraw consent, loss to follow-up, moved, etc.), or 3) on study but missing data in window. The full categorization of virologic outcome at Week 48 and Week 96 will be summarized by treatment group.

A sensitivity analysis will be performed using the OF approach under which non-intermittent missing data for subjects who prematurely discontinued assigned treatment due to lack of efficacy are considered as failures at timepoints thereafter. This sensitivity analysis will be limited to the primary efficacy analysis only (i.e., the proportion of subjects achieving HIV-1 RNA <50 copies/mL at Week 48).

**Protocol/Amendment No.:** 021-09

A margin of 10 percentage points is used to define the non-inferiority of MK-1439A q.d. to ATRIPLA<sup>TM</sup> q.d.; this is consistent with regulatory recommendations. MK-1439A q.d. will be concluded non-inferior to ATRIPLA<sup>TM</sup> q.d. if the lower bound of the two-sided 95% CI for the difference in the proportion of subjects with HIV-1 RNA <50 copies/mL at Week 48 (MK-1439A minus ATRIPLA<sup>TM</sup> q.d) is greater than -10 percentage points. It can be further concluded that MK-1439A q.d. is superior to ATRIPLA<sup>TM</sup> q.d. if the lower bound of the two-sided 95% CI for the difference in response rates (MK-1439A minus ATRIPLA<sup>TM</sup> q.d) is greater than zero contingent upon satisfying the multiplicity criteria.

For the summary of virologic response over time, the difference in proportions between treatment groups at each time point will also be estimated and the associated two-sided 95% CI will be derived in a similar fashion to that described for the primary efficacy analysis.

#### Change from Baseline in CD4 cell counts

Change from baseline in CD4 cell counts will be summarized by treatment group at each time point at which CD4 cell count is collected, with a key interest at Week 48. The treatment difference in changes from baseline in CD4 cell count at each time point will be estimated between the 2 treatment groups. However, these estimates will not be subject to an absolute criterion for similarity. The clinical interpretation of the treatment difference is dependent upon the absolute value at baseline, and the magnitude and direction of the CD4 changes seen in each treatment arm.

The OF approach will be used for the calculations of change from baseline in CD4 cell count. Under this approach, baseline values will be carried forward for subjects who discontinue due to lack of efficacy.

#### Protocol-Defined Virologic Failure

The number of subjects with protocol-defined virologic failure will be summarized for each treatment group.

Table 10 summarizes the key efficacy analyses.

**Protocol/Amendment No.:** 021-09

Table 10 Analysis Strategy for Key Efficacy Variables

| Endpoint/Variable (Description, Time Point) | Primary vs.<br>Supportive<br>Approach <sup>†</sup> | Statistical Method | Analysis<br>Population | Missing Data<br>Approach |
|---|---|---|---|---|
| <b>Primary Hypothesis</b> | | | | |
| Proportion of subjects<br>achieving HIV-1 RNA<br><50 copies/mL at Week 48 | P | Stratum-adjusted<br>Mantel-Haenszel <sup>‡</sup> | FAS | NC=F approach |
| Proportion of subjects<br>achieving HIV-1 RNA<br><50 copies/mL at Week 48 | S | Stratum-adjusted<br>Mantel-Haenszel‡ | FAS | OF approach |
| Secondary Objectives | | | | |
| Proportion of subjects<br>achieving HIV-1 RNA<br><50 copies/mL at Week 96 | P | Stratum-adjusted<br>Mantel-Haenszel <sup>‡</sup> | FAS | NC=F approach |
| Change from baseline in CD4 cell counts at Week 48 and Week 96 | P | Two sample t-test | FAS | OF approach<br>assuming<br>baseline-carried-<br>forward |

P=Primary approach; S=Secondary approach.

The strategy to address multiplicity issues with regard to multiple treatment comparisons, multiple endpoints, multiple timepoints, and/or interim analyses is described in Section 8.7, Interim Analyses and in Section 8.8, Multiplicity.

## **8.6.2** Statistical Methods for Safety Analyses

Safety and tolerability will be assessed by clinical review of all relevant parameters including AEs, laboratory tests and vital signs.

The analysis of safety results will follow a tiered approach Table 11. The tiers differ with respect to the analyses that will be performed. Safety parameters or adverse experiences of special interest that are identified *a priori* constitute "Tier 1" safety endpoints that will be subject to inferential testing for statistical significance with p-values and 95% confidence intervals provided for between-group comparisons. Other safety parameters will be considered Tier 2 or Tier 3. Tier 2 parameters will be assessed via point estimates with 95% confidence intervals provided for between-group comparisons; only point estimates by treatment group are provided for Tier 3 safety parameters.

AEs (specific terms as well as system organ class terms) and predefined limits of change in laboratory parameters that are not pre-specified as Tier-1 endpoints will be classified as belonging to "Tier 2" or "Tier 3", based on the number of events observed. Membership in Tier 2 requires that at least 4 subjects in any treatment group exhibit the event; all other adverse experiences and predefined limits of change will belong to Tier 3.

<sup>&</sup>lt;sup>‡</sup> Stratum-adjusted (screening HIV RNA-1 ≤100,000 vs. >100,000 copies /mL) Mantel-Haenszel method with the difference weighted by the harmonic mean of the sample size per arm for each stratum.

Protocol/Amendment No.: 021-09

The threshold of at least 4 events was chosen because the 95% confidence interval for the between-group difference in percent incidence will always include zero when treatment groups of equal size each have less than 4 events and thus would add little to the interpretation of potentially meaningful differences. Because many 95% confidence intervals may be provided without adjustment for multiplicity, the confidence intervals should be regarded as a helpful descriptive measure to be used in review, not a formal method for assessing the statistical significance of the between-group differences in adverse experiences and predefined limits of change.

Continuous measures such as changes from baseline in laboratory and vital signs parameters that are not pre-specified as Tier-1 endpoints will be considered Tier 3 safety parameters. Summary statistics for baseline, on-treatment, and change from baseline values will be provided by treatment group in table format.

For this protocol, the proportion of subjects with neuropsychiatric AEs by Week 48 in 3 prespecified categories (dizziness, sleep disorders and disturbances, and altered sensorium with each tested separately) and the change from baseline in fasting LDL-C and non-HDL-C at Week 48 are considered Tier 1 events.

The proportion of subjects with neuropsychiatric AEs by Week 48 in the depression and suicide/self-injury and psychosis and psychotic disorders categories as well as the proportion of subjects experiencing one or more AE in any of the 5 pre-specified categories of neuropsychiatric adverse events will be considered Tier 2 events. For these as well as Tier 1 neuropsychiatric AEs, the treatment difference and the associated 95% confidence interval will be calculated using the Miettinen and Nurminen's method (1985) [5], an unconditional, asymptotic method, and p-values based on this method will be provided for the Tier 1 categories of dizziness, sleep disorders and disturbances, and altered sensorium.

Note that there is no adjustment for safety stratification (Hepatitis B/C status) in the calculation of the confidence intervals or p-values, since the purpose of this stratification factor is to help balance the treatment groups for better interpretation of any potential imbalance in serious liver function abnormalities. This stratification factor has no expected impact on the primary safety endpoint of neuropsychiatric AEs.

The change from baseline in fasting lipids will be analyzed using ANCOVA models adjusted by baseline lipid level and treatment group. The treatment differences and 95% confidence intervals will be provided for all lipid parameters, and the p-value for the between treatment comparison will be provided for LDL-C and non-HDL-C. The missing lipid data will be handled by the following principle: For subjects who have missing lipid data, the last lipid observation after randomization will be carried forward. For subjects who modify (start, stop, increase or decrease dosage) lipid-lowering therapy use during the study, the last lipid observation before modifying the lipid-lowering therapy use will be carried forward for later time points.

The percentages of subjects who modify lipid-lowering therapy during the study will be summarized by treatment group. The difference in percentages between treatment groups

**Protocol/Amendment No.:** 021-09

and the associated 95% confidence interval will be calculated using Miettinen and Nurminen's method.

In addition, the broad clinical and laboratory AE categories consisting of the percentage of subjects with any AE, with a drug-related AE, with a serious AE, with an AE which is both drug-related and serious, and who discontinued due to an AE will be considered Tier 2 endpoints. The 95% confidence intervals will be provided for between treatment differences in the percentage of subjects with events; these analyses will be performed using the Miettinen and Nurminen method.

Table 11 Analysis Strategy for Safety Parameters

| | | | 95% CI for | <b>.</b> |
|---|---|---|---|---|
| ~ ~ | | | Treatment | Descriptive |
| Safety Tier | Safety Endpoint <sup>†</sup> | p-Value | Comparison | Statistics |
| Tier 1 | Proportion of subjects with neuropsychiatric AEs | X | X | X |
| | in the following categories: | | | |
| | • Dizziness | | | |
| | Sleep disorders and disturbances | | | |
| | Altered Sensorium | | | |
| | Change from baseline in fasting LDL-C and non-HDL-C | | | |
| Tier 2 | Proportion of subjects with neuropsychiatric AEs | | X | X |
| | in the following categories: | | | |
| | Depression and suicide/self-injury | | | |
| | <ul> <li>Psychosis and psychotic disorders</li> </ul> | | | |
| | Proportion of subjects with one or more | | X | X |
| | neuropsychiatric AEs | | | |
| | Change from baseline in fasting lipids not classified as Tier 1 | | | |
| | Starting lipid-lowering therapy | | X | X |
| | Any AE | | X | X |
| | Any Serious AE | | X | X |
| | Any Drug-Related AE | | X | X |
| | Any Serious and Drug-Related AE | | X | X |
| | Discontinuation due to AE | | X | X |
| | Specific AEs, SOCs, or PDLCs <sup>‡</sup> (incidence ≥4 of | | X | X |
| | subjects in one of the treatment groups) | | | |
| Tier 3 | Specific AEs, SOCs or PDLCs <sup>‡</sup> (incidence <4 of | | | X |
| | subjects in all of the treatment groups) | | | |
| | Change from Baseline Results (Labs, Vital Signs) | | | X |

<sup>†</sup> Adverse Experience references refer to both Clinical and Laboratory AEs.

<sup>‡</sup> Includes only those endpoints not pre-specified as Tier 1 and not already pre-specified as Tier-2 endpoints. Note: SOC = System Organ Class; PDLC = Pre-Defined Limit of Change; X = results will be provided.

## 8.6.3 Summaries of Baseline Characteristics, Demographics, and Other Analyses

### **8.6.3.1** Demographic and Baseline Characteristics

The comparability of the treatment groups for each relevant characteristic will be assessed by the use of tables and/or graphs. No statistical hypothesis tests will be performed on these characteristics. The number and percentage of subjects screened, randomized, the primary reasons for screening failure, and the primary reason for discontinuation will be displayed. Demographic variables (e.g., age, gender, race, region, etc.), baseline characteristics, primary and secondary diagnoses, and prior and concomitant therapies will be summarized by treatment either by descriptive statistics or categorical tables.

#### 8.7 Interim Analyses

No interim analyses for efficacy are planned for this study. However, an external data monitoring committee will convene to review safety data approximately every 6 months during the study.

## 8.8 Multiplicity

There are no interim analyses for efficacy and no plans to stop for favorable safety in this study as part of the periodic (~every 6 months) DMC safety reviews. However, as it is customary to spend a small amount of alpha for interim analyses for safety performed by the DMC when there is a primary safety hypothesis, an alpha level of 0.00001 will be allocated for each DMC safety review through Week 48 before testing the primary safety hypothesis and subsequent safety hypotheses.

The primary efficacy hypothesis for non-inferiority will be tested at an unadjusted one-sided alpha level of 0.025 because no interim efficacy analysis will be performed. Furthermore, provided all safety hypotheses are satisfied after establishing the primary efficacy hypothesis, the superiority hypothesis for efficacy will be tested at the unadjusted alpha level of 0.025 as well.

The following hypotheses will be tested sequentially at the one-sided Type 1 error rate of 2.5% (unadjusted for the efficacy hypotheses [#1,7] and after adjusting for interim DMC safety reviews for the safety hypotheses [#2-6]) in the following order:

- 1) Primary efficacy hypothesis testing non-inferiority at Week 48
- 2) Primary safety hypothesis for dizziness
- 3) Primary safety hypothesis for sleep disorders and disturbances
- 4) Primary safety hypothesis for altered sensorium
- 5) Secondary safety hypothesis for LDL-C

**Protocol/Amendment No.:** 021-09

6) Secondary safety hypothesis for non-HDL-C

7) Secondary efficacy hypothesis testing superiority at Week 48

Testing will stop with the first of these tests failing to reach statistical significance and all subsequent tests would not be considered for statistical significance. In this way, the overall one-sided Type 1 error rate in testing these hypotheses is strongly controlled at a 2.5% level.

Note the secondary efficacy hypotheses testing non-inferiority and superiority at Week 96 are only supportive to the primary and secondary efficacy hypotheses at Week 48 and are not considered in the strong control strategy for the Type 1 error for this study.

There are no other hypotheses that will be tested and analyses associated with objectives without hypotheses will be considered supportive and/or explanatory.

### 8.9 SAMPLE SIZE AND POWER CALCULATIONS

#### 8.9.1 Sample Size and Power for Efficacy Analyses

The study will randomize 340 subjects into each treatment arm to achieve 90% power to demonstrate the primary hypothesis that MK-1439A q.d. is non-inferior to ATRIPLA<sup>TM</sup> q.d., at an overall one-sided 2.5% alpha level, as measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48. The power calculation assumes a true response rate of 80% at Week 48 for both the MK-1439A q.d. arm and the ATRIPLA™ q.d arm using the NC=F approach as defined by the FDA "snapshot" approach. A margin of 10 percentage points is used to define the non-inferiority of MK-1439A q.d. versus ATRIPLA<sup>TM</sup> q.d.; this is consistent with regulatory recommendations. Given the non-inferiority margin of 10%, the assumed response rates and the chosen sample size, non-inferiority may be established when the observed difference in response rates (MK-1439A q.d. minus ATRIPLA<sup>TM</sup> q.d.) is approximately -3.7% or larger; superiority may be concluded when the observed difference in response rates is approximately 5.7% or larger under the multiplicity testing strategy in Section 8.8. The power calculation is based on an asymptotic method proposed by Farrington and Manning (1990) [6] and is carried out using SAS v9.3. Table 12 summarizes the power for the primary comparison under various assumptions for the control response rate and underlying difference in response rates.

Table 12 Power (%) Under Various Assumptions (With 340 Subjects Randomized in Each Treatment Group)

| Response Rate (%) in | | | lying Differe<br>//K-1439A q | | , | %) | |
|---|---|---|---|---|---|---|---|
| ATRIPLA™ q.d. | -3 | -2 | -1 | 0 | 1 | 2 | 3 |
| 74 | 54 | 65 | 76 | 84 | 91 | 95 | 98 |
| 77 | 56 | 68 | 79 | 87 | 93 | 96 | 98 |
| 80 | 60 | 72 | 83 | 90 | 95 | 98 | 99 |
| 83 | 65 | 77 | 87 | 93 | 97 | 99 | >99 |
| 86 | 70 | 82 | 91 | 96 | 98 | >99 | >99 |
| Note: The power is calculate | d based on 340 | subjects expec | eted to be inclu | uded in the an | alysis for eacl | n treatment gro | oup |

## 8.9.2 Sample Size and Power for Safety Analyses

### Neuropsychiatric Adverse Experiences

MK-1439 Protocol 007 studied 4 doses of MK-1439 versus efavirenz, each in combination therapy with TRUVADATM, in HIV-1 infected treatment-naïve subjects. Based on data from Protocol 007, the expected proportions of subjects with events in each of the categories of pre-specified neuropsychiatric adverse events through Week 48 are as follows: dizziness (5% vs 24%), sleep disorders and disturbances (16% vs 29%), altered sensorium (3% vs 10%), depression and suicide/self-injury (4% vs 10%), and psychosis and psychotic disorders (2% vs 2%) in the MK-1439A group and the ATRIPLA<sup>TM</sup> group, respectively. Due to multiplicity and power considerations, only the first 3 neuropsychiatric adverse event categories (dizziness, sleep disorders and disturbances, and altered sensorium) were selected for statistical testing. If the proportions of subjects with neuropsychiatric AEs in this study are similar to those observed in Protocol 007, the power to detect a difference between MK-1439A and ATRIPLA<sup>TM</sup> in the respective Tier 1 categories (dizziness, sleep disorders and disturbances, and altered sensorium) with 340 subjects in each treatment arm is >99%, 97%, and 95%, respectively. Table 13 displays the observed percentage of subjects in each category by treatment group that would be necessary to demonstrate superiority of MK-1439A versus ATRIPLA<sup>TM</sup> assuming the efavirenz event percentages from Protocol 007 for ATRIPLATM:

Table 13 Observed Percentage in MK-1439A Necessary to Demonstrate Superiority versus ATRIPLA<sup>TM</sup>

| | MK-1439A q.d. Superiority will be achieved provided the observed % is less than or equal to | ATRIPLA <sup>TM</sup> q.d. (same as efavirenz in P007) |
|---|---|---|
| Dizziness | 17% | 24% |
| Sleep disorders and disturbances | 22% | 29% |
| Altered Sensorium | 5% | 10% |

#### Lipids

The change from baseline in fasting LDL-C and non-HDL-C at Week 48 will be analyzed using ANCOVA models adjusted by baseline lipids level and treatment group. MK-1439A q.d. will be concluded to be superior to ATRIPLA<sup>TM</sup> q.d. if the mean change from baseline in LDL-C for the MK-1439A group is significantly lower than that for the ATRIPLA<sup>TM</sup> group. If superiority for LDL-C is established, sequential testing for non-HDL-C will be conducted.

If we assume that ATRIPLA<sup>TM</sup> q.d. has an effect on lipids at least as large as efavirenz, the treatment difference in mean change from baseline in lipids observed in Protocol 007 can be used as an estimate for the power calculation for this study.

Protocol/Amendment No.: 021-09

The estimated between treatment differences in mean changes in fasting LDL-C and non-HDL-C, based on the interim data from MK-1439 Protocol 007, were 7.7 mg/dL (standard deviation of 20 mg/dL) and 20 mg/dL (standard deviation of 25 mg/dL), respectively. With 340 subjects in each treatment group, the study has >99% power to detect a between treatment difference of 7.7 mg/dL for mean change from baseline in LDL-C. The study also has >99% power to detect a between treatment difference of 20 mg/dL for mean change from baseline in non-HDL-C.

#### Adverse Experiences

The probability of observing at least one of a particular type of adverse experience in this study depends on the number of subjects treated and the underlying percentage of subjects with that adverse experience in the study population. If the underlying incidence of a particular adverse experience is 1% (1 of every 100 subjects receiving the drug), there is a 96.7% chance of observing at least one adverse experience among 340 subjects in any treatment group. If no adverse experience of that type is observed among the 340 subjects in any treatment group, this study will provide 95% confidence that the underlying percentage of subjects with that particular adverse experience is <1.1% for the treatment group.

The estimate of, and the upper bound of the 95% confidence interval for, the underlying percentage of subjects with an AE given various hypothetical observed number of subjects with the AE within each treatment group are provided in Table 14. These calculations are based on the exact binomial method proposed by Clopper and Pearson (1934) [7].

Table 14 Estimate of Incidence of AEs and 95% Upper Confidence Bound Based on Hypothetical Numbers of Subjects with AEs Among 340 Subjects Randomized in Each Treatment Group

| Hypothetical Number of Subjects With An Adverse Event | Estimate of Incidence | 95% Upper Confidence Bound <sup>†</sup> |
|---|---|---|
| 0 | 0% | 1.1 |
| 5 | 1.5% | 3.4 |
| 10 | 2.9% | 5.3 |
| 15 | 4.4% | 7.2 |
| 20 | 5.9% | 8.9 |
| 25 | 7.4% | 10.7 |
| 30 | 8.8% | 12.4 |

<sup>†</sup> Based on the two-tailed exact confidence interval for a binomial proportion (Clopper and Pearson, 1934 [7]).

Table 15 gives the difference in the incidence of adverse experiences (MK-1439A q.d. – ATRIPLA<sup>TM</sup> q.d.) that can be ruled out with different power levels and 95% confidence when there are 340 subjects in each treatment group. The underlying incidence of adverse experiences is assumed to be the same for the 2 treatment groups. For a reasonably common adverse experience which occurs in 20% of subjects either in the MK-1439A q.d. arm or

**Protocol/Amendment No.:** 021-09

ATRIPLA™ q.d. arm, the study has 90% power to declare with 95% confidence that the true difference between the treatment groups is no more than 9.9 percentage points. The calculations are based on an asymptotic method proposed by Farrington and Manning (1990) [6].

Table 15 Differences in Incidences of AEs (MK-1439A q.d. minus ATRIPLA™ q.d.) That Can Be Ruled Out With 340 Subjects in Each Treatment Group

| | Difference <sup>†</sup> in Percentage Points That Can Be Ruled Out with Target Power Assuming the Underlying Incidence of the AE is | | | | |
|---|---|---|---|---|---|
| Target Power | 10% | 20% | 30% | 40% | 50% |
| 80 | 6.4 | 8.6 | 9.8 | 10.5 | 10.7 |
| 85 | 6.9 | 9.2 | 10.5 | 11.3 | 11.5 |
| 90 | 7.5 | 9.9 | 11.4 | 12.2 | 12.4 |
| 95 | 8.3 | 11.1 | 12.7 | 13.5 | 13.8 |

<sup>†</sup>The upper bound of the two-sided 95% confidence interval (Farrington and Manning (1990) for the difference in AE incidences (MK-1439 100 mg q.d. minus darunavir/ritonavir [800 mg/100mg] q.d.) assuming the incidences are the same.

#### 8.9.3 Overall Power

The following hypotheses will be tested sequentially at the one-sided Type 1 error rate of 2.5% (unadjusted for the efficacy hypotheses [#1,7] and after adjusting for interim DMC safety reviews for the safety hypotheses [#2-6]) in the following order:

- 1) Primary efficacy hypothesis testing non-inferiority at Week 48
- 2) Primary safety hypothesis for dizziness
- 3) Primary safety hypothesis for sleep disorders and disturbances
- 4) Primary safety hypothesis for altered sensorium
- 5) Secondary safety hypothesis for LDL-C
- 6) Secondary safety hypothesis for non-HDL-C
- 7) Secondary efficacy hypothesis testing superiority at Week 48

Testing will stop with the first of these tests failing to reach statistical significance and all subsequent tests would not be considered for statistical significance. In this way, the overall one-sided Type 1 error rate in testing these hypotheses is strongly controlled at a 2.5% level. The probability to reach steps 2 through 7 for statistical testing (could also be considered the power to establish the hypotheses in steps 1 through 6) is approximately 90%, 89%, 86%, 82%, 81%, and 80%, respectively.

## 8.10 Subgroup Analyses and Effect of Baseline Factors (Base Study)

To determine whether the treatment effect is consistent across various subgroups, the estimate of the between-group treatment effect (with a nominal 95% CI unadjusted for stratification factors) for the primary endpoint will be calculated and plotted within each category of the following classification variables:

- Age category (≤median vs. >median)
- Gender (female, male)
- Region (North America, South America, Europe, Asia, Africa, etc.)
- Race (White, Black, Asian, Other)
- Ethnicity (Hispanic/Latino, not Hispanic/Latino)
- Screening HIV-1 RNA categories (HIV-1 RNA ≤100,000 copies/mL, HIV-1 RNA >100,000 copies/mL)
- Baseline HIV-1 RNA categories (HIV-1 RNA ≤100,000 copies/mL, HIV-1 RNA >100,000 copies/mL)
- Chronic Hepatitis B or C status (HBV/HCV-infected or HBV/HCV-uninfected)
- Baseline CD4 categories (<50, 50-200, and >200 cells/mm<sup>3</sup>)

The Observed Failure approach will be used to handle missing values in these subgroup analyses.

### 8.11 Compliance (Medication Adherence)

Study Medication Diary Cards will be used to ensure and document the drug compliance in the base study and study extension 1.

Subjects are to take one pill once daily from each of the 2 bottles (A & B) of study medication during the base study. For the main analysis of compliance in the base study, a day within the study will be considered an "On-Therapy" day if the subject takes at least one tablet from any bottle provided for this study.

For a subject who is followed for the entire study period, the "Number of Days Should be on Therapy" is the total number of days from Day 1 to the last scheduled day for treatment administration for that subject. For a subject who discontinued from the study permanently, the "Number of Days Should be on Therapy" is the total number of days from Day 1 to the date of the last dose of study medication.

For each subject, percent compliance will then be calculated using the following formula:

**Protocol/Amendment No.:** 021-09

Summary statistics will be provided on percent compliance by treatment group for the FAS population.

A second analysis in the base study using a different definition of compliance will also be conducted. In this analysis, a day within the study will be considered an "On-Therapy" day only if the subject takes the required number of tablets from all bottles provided for this study (as noted in Section 7.1.5.2) will also be summarized.

During the study extensions, MK-1439A will be provided as study medication by the sponsor. Compliance with MK-1439A administration will be summarized for study extension 1. A day within the study will be considered an "On-Therapy" day if the subject takes 1 tablet of MK-1439A.

Data from the study medication diary, rather than the returned pill count will serve as the primary data for compliance.

Compliance data will not be collected and analyzed for study extension 2 or for study extension 3.

## **8.12** Extent of Exposure

The extent of exposure to study therapy for all randomized and treated subjects will be summarized. The number of subjects exposed to various doses (actual total daily dose) for defined periods of time will be listed, along with a summary of the mean (range) duration subjects were exposed to various doses.

## 9.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL SUPPLIES

#### 9.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Clinical Supplies will be provided by the Sponsor as summarized in Table 16.

**Protocol/Amendment No.:** 021-09

Table 16 Product Descriptions: Base Study and Study Extensions

| Product Name & Potency | Dosage Form |
|---|---|
| Base Study | |
| MK-1439A 100 mg/ 300 mg/ 300 mg or Placebo to match MK-1439A 100 mg/ 300 mg/ 300 mg | Tablet |
| Efavirenz 600 mg / emtricitabine 200mg / tenofovir disoproxil fumarate 300 mg (which is equivalent to 245 mg of tenofovir disoproxil). (ATRIPLA <sup>TM</sup> ) or Placebo to match Efavirenz 600 mg / emtricitabine 200 mg / tenofovir disoproxil fumarate 300 mg (which is equivalent to 245 mg of tenofovir disoproxil). (ATRIPLA <sup>TM</sup> ) | Tablet |
| Study Extensions | |
| MK-1439A 100 mg/ 300 mg/ 300 mg | Tablet |

All placebos were created by the Sponsor to match the active product.

## 9.2 Packaging and Labeling Information

Clinical supplies will be affixed with a clinical label in accordance with regulatory requirements.

During the base study, subjects will receive blinded monthly bottles. No kitting is required. During the study extensions, subjects will receive open-label MK-1439A.

#### 9.3 Clinical Supplies Disclosure

The emergency unblinding call center will use the randomization schedule for the trial to unblind subjects and to unmask treatment. The emergency unblinding call center should only be used in cases of emergency (see Section 7.1.4.2). In the event that the emergency unblinding call center is not available for a given site in this trial, the central electronic randomization system (IVRS/IWRS) should be used in order to unblind subjects and to unmask treatment/vaccine identity. The Sponsor will provide random code/disclosure envelopes or lists to the emergency unblinding call center.

Treatment identification information is to be unmasked ONLY if necessary for the welfare of the subject. Every effort should be made not to unblind the subject unless necessary.

In the event that unblinding has occurred, the circumstances around the unblinding (eg, date, reason and person performing the unblinding) must be documented promptly, and the Sponsor Clinical Director notified as soon as possible. Once an emergency unblinding has

taken place, the principal investigator, site personnel, and Sponsor personnel may be unblinded so that the appropriate follow-up medical care can be provided to the subject.

## 9.4 Storage and Handling Requirements

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

### 9.5 Returns and Reconciliation

The investigator is responsible for keeping accurate records of the clinical supplies received from the Sponsor or designee, the amount dispensed to and returned, and the amount remaining at the conclusion of the trial. For all trial sites, the local country Sponsor personnel or designee will provide appropriate documentation that must be completed for drug accountability and return, or local discard and destruction if appropriate. Where local discard and destruction is appropriate, the investigator is responsible for ensuring that a local discard/destruction procedure is documented.

#### 9.6 Standard Policies

Trial site personnel will have access to a central electronic randomization system (IVRS/IWRS system) to allocate subjects, to assign treatment to subjects and to manage the distribution of clinical supplies. Each person accessing the IVRS system must be assigned an individual unique PIN. They must use only their assigned PIN to access the system, and they must not share their assigned PIN with anyone.

At the close of the trial after unblinding, a letter is to be sent by the investigator to those subjects who received placebos in the image of the competitor's product to provide the following advice:

"You have participated in a trial conducted by the Sponsor. This is to advise you that you were among those who received a look-alike tablet created by the Sponsor to resemble the drug ATRIPLA<sup>TM</sup> (efavirenz 600 mg / emtricitabine 200 mg / tenofovir disoproxil fumarate 300 mg) as much as possible. You did not receive the active drug ATRIPLA<sup>TM</sup> (efavirenz 600 mg / emtricitabine 200 mg / tenofovir disoproxil fumarate 300 mg [which is equivalent to 245 mg of tenofovir disoproxil]) as manufactured by Gilead Sciences."

Protocol/Amendment No.: 021-09

#### 10.0 ADMINISTRATIVE AND REGULATORY DETAILS

### **10.1** Confidentiality

### 10.1.1 Confidentiality of Data

By signing this protocol, the investigator affirms to the Sponsor that information furnished to the investigator by the Sponsor will be maintained in confidence, and such information will be divulged to the institutional review board, ethics review committee (IRB/ERC) or similar or expert committee; affiliated institution and employees, only under an appropriate understanding of confidentiality with such board or committee, affiliated institution and employees. Data generated by this trial will be considered confidential by the investigator, except to the extent that it is included in a publication as provided in the Publications section of this protocol.

### 10.1.2 Confidentiality of Subject Records

By signing this protocol, the investigator agrees that the Sponsor (or Sponsor representative), IRB/ERC, or regulatory authority representatives may consult and/or copy trial documents in order to verify worksheet/case report form data. By signing the consent form, the subject agrees to this process. If trial documents will be photocopied during the process of verifying worksheet/case report form information, the subject will be identified by unique code only; full names/initials will be masked prior to transmission to the Sponsor.

By signing this protocol, the investigator agrees to treat all subject data used and disclosed in connection with this trial in accordance with all applicable privacy laws, rules and regulations.

### 10.1.3 Confidentiality of Investigator Information

By signing this protocol, the investigator recognizes that certain personal identifying information with respect to the investigator, and all subinvestigators and trial site personnel, may be used and disclosed for trial management purposes, as part of a regulatory submissions, and as required by law. This information may include:

- 1. name, address, telephone number and e-mail address;
- 2. hospital or clinic address and telephone number;
- 3. curriculum vitae or other summary of qualifications and credentials; and
- 4. other professional documentation.

08K3V5

Consistent with the purposes described above, this information may be transmitted to the Sponsor, and subsidiaries, affiliates and agents of the Sponsor, in your country and other countries, including countries that do not have laws protecting such information. Additionally, the investigator's name and business contact information may be included

Protocol/Amendment No.: 021-09

when reporting certain serious adverse events to regulatory authorities or to other investigators. By signing this protocol, the investigator expressly consents to these uses and disclosures.

If this is a multicenter trial, in order to facilitate contact between investigators, the Sponsor may share an investigator's name and contact information with other participating investigators upon request.

## 10.1.4 Confidentiality of IRB/IEC Information

The Sponsor is required to record the name and address of each IRB/IEC member that reviews and approves this trial. The Sponsor is also required to document that each IRB/IEC meets regulatory and ICH GCP requirements by requesting and maintaining records of the names and qualifications of the IRB/IEC members and to make these records available for regulatory agency review upon request by those agencies.

## 10.2 Compliance with Financial Disclosure Requirements

Financial Disclosure requirements are outlined in the US Food and Drug Administration Regulations, Financial Disclosure by Clinical Investigators (21 CFR Part 54). It is the Sponsor's responsibility to determine, based on these regulations, whether a request for Financial Disclosure information is required. It is the investigator's/subinvestigator's responsibility to comply with any such request.

The investigator/subinvestigator(s) agree, if requested by the Sponsor in accordance with 21 CFR Part 54, to provide his/her financial interests in and/or arrangements with the Sponsor to allow for the submission of complete and accurate certification and disclosure statements. The investigator/subinvestigator(s) further agree to provide this information on a Certification/Disclosure Form, commonly known as a financial disclosure form, provided by the Sponsor or through a secure password-protected electronic portal provided by the The investigator/subinvestigator(s) also consent to the transmission of this information to the Sponsor in the United States for these purposes. This may involve the transmission of information to countries that do not have laws protecting personal data.

#### 10.3 Compliance with Law, Audit and Debarment

By signing this protocol, the investigator agrees to conduct the trial in an efficient and diligent manner and in conformance with this protocol; generally accepted standards of Good Clinical Practice (e.g., International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice: Consolidated Guideline and other generally accepted standards of good clinical practice); and all applicable federal, state and local laws, rules and regulations relating to the conduct of the clinical trial.

The Code of Conduct, a collection of goals and considerations that govern the ethical and scientific conduct of clinical investigations sponsored by MSD, is provided in Section 12.1 -Code of Conduct for Clinical Trials.

MK-1439A-021-09 Final Protocol 02-Nov-2022 Confidential

08K3V5

Protocol/Amendment No.: 021-09

The investigator also agrees to allow monitoring, audits, IRB/ERC review and regulatory authority inspection of trial-related documents and procedures and provide for direct access to all trial-related source data and documents.

The investigator agrees not to seek reimbursement from subjects, their insurance providers or from government programs for procedures included as part of the trial reimbursed to the investigator by the Sponsor.

The investigator shall prepare and maintain complete and accurate trial documentation in compliance with Good Clinical Practice standards and applicable federal, state and local laws, rules and regulations; and, for each subject participating in the trial, provide all data, and, upon completion or termination of the clinical trial, submit any other reports to the Sponsor as required by this protocol or as otherwise required pursuant to any agreement with the Sponsor.

Trial documentation will be promptly and fully disclosed to the Sponsor by the investigator upon request and also shall be made available at the trial site upon request for inspection, copying, review and audit at reasonable times by representatives of the Sponsor or any regulatory authorities. The investigator agrees to promptly take any reasonable steps that are requested by the Sponsor as a result of an audit to cure deficiencies in the trial documentation and worksheets/case report forms.

The investigator must maintain copies of all documentation and records relating to the conduct of the trial in compliance with all applicable legal and regulatory requirements. This documentation includes, but is not limited to, the protocol, worksheets/case report forms, advertising for subject participation, adverse event reports, subject source data, correspondence with regulatory authorities and IRBs/ERCs, consent forms, investigator's curricula vitae, monitor visit logs, laboratory reference ranges, laboratory certification or quality control procedures and laboratory director curriculum vitae. By signing this protocol, the investigator agrees that documentation shall be retained until at least 2 years after the last approval of a marketing application in an ICH region or until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. Because the clinical development and marketing application process is variable, it is anticipated that the retention period can be up to 15 years or longer after protocol database lock. The Sponsor will determine the minimum retention period and notify the investigator when documents may be destroyed. The Sponsor will determine the minimum retention period and upon request, will provide guidance to the investigator when documents no longer need to be retained. The sponsor also recognizes that documents may need to be retained for a longer period if required by local regulatory requirements. All trial documents shall be made available if required by relevant regulatory authorities. The investigator must consult with and obtain written approval by the Sponsor prior to destroying trial and/or subject files.

ICH Good Clinical Practice guidelines recommend that the investigator inform the subject's primary physician about the subject's participation in the trial if the subject has a primary physician and if the subject agrees to the primary physician being informed.

02-Nov-2022

Protocol/Amendment No.: 021-09

The investigator will promptly inform the Sponsor of any regulatory authority inspection conducted for this trial.

Persons debarred from conducting or working on clinical trials by any court or regulatory authority will not be allowed to conduct or work on this Sponsor's trials. The investigator will immediately disclose in writing to the Sponsor if any person who is involved in conducting the trial is debarred or if any proceeding for debarment is pending or, to the best of the investigator's knowledge, threatened.

In the event the Sponsor prematurely terminates a particular trial site, the Sponsor will promptly notify that trial site's IRB/IEC.

According to European legislation, a Sponsor must designate an overall coordinating investigator for a multi-center trial (including multinational). When more than one trial site is open in an EU country, MSD, as the Sponsor, will designate, per country, a national principal coordinator (Protocol CI), responsible for coordinating the work of the principal investigators at the different trial sites in that Member State, according to national regulations. For a single-center trial, the Protocol CI is the principal investigator. In addition, the Sponsor must designate a principal or coordinating investigator to review the trial report that summarizes the trial results and confirm that, to the best of his/her knowledge, the report accurately describes the conduct and results of the trial [Clinical Study Report (CSR) CI]. The Sponsor may consider one or more factors in the selection of the individual to serve as the Protocol CI and or CSR CI (e.g., availability of the CI during the anticipated review process, thorough understanding of clinical trial methods, appropriate enrollment of subject cohort, timely achievement of trial milestones). The Protocol CI must be a participating trial investigator.

## 10.4 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Amendments Act (FDAAA) of 2007 and the European Medicines Agency (EMA) clinical trial Directive 2001/20/EC, the Sponsor of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to http://www.clinicaltrials.gov, www.clinicaltrialsregister.eu or other local registries. MSD, as Sponsor of this trial, will review this protocol and submit the information necessary to fulfill these requirements. MSD entries are not limited to FDAAA or the EMA clinical trial directive mandated trials. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

By signing this protocol, the investigator acknowledges that the statutory obligations under FDAAA, the EMA clinical trials directive or other locally mandated registries are that of the Sponsor and agrees not to submit any information about this trial or its results to those registries.

Protocol/Amendment No.: 021-09

## 10.5 Quality Management System

By signing this protocol, the Sponsor agrees to be responsible for implementing and maintaining a quality management system with written development procedures and functional area standard operating procedures (SOPs) to ensure that trials are conducted and data are generated, documented, and reported in compliance with the protocol, accepted standards of Good Clinical Practice, and all applicable federal, state, and local laws, rules and regulations relating to the conduct of the clinical trial.

## 10.6 Data Management

The investigator or qualified designee is responsible for recording and verifying the accuracy By signing this protocol, the investigator acknowledges that his/her of subject data. electronic signature is the legally binding equivalent of a written signature. By entering his/her electronic signature, the investigator confirms that all recorded data have been verified as accurate.

Detailed information regarding Data Management procedures for this protocol will be provided separately.

#### 10.7 Publications

This trial is intended for publication, even if terminated prematurely. Publication may include any or all of the following: posting of a synopsis online, abstract and/or presentation at a scientific conference, or publication of a full manuscript. The Sponsor will work with the authors to submit a manuscript describing trial results within 12 months after the last data become available, which may take up to several months after the last subject visit in some cases such as vaccine trials. However, manuscript submission timelines may be extended on OTC trials. For trials intended for pediatric-related regulatory filings, the investigator agrees to delay publication of the trial results until the Sponsor notifies the investigator that all relevant regulatory authority decisions on the trial drug have been made with regard to pediatric-related regulatory filings. MSD will post a synopsis of trial results for approved products on www.clinicaltrials.gov by 12 months after the last subject's last visit for the primary outcome, 12 months after the decision to discontinue development, or product marketing (dispensed, administered, delivered or promoted), whichever is later.

These timelines may be extended for products that are not yet marketed, if additional time is needed for analysis, to protect intellectual property, or to comply with confidentiality agreements with other parties. Authors of the primary results manuscript will be provided the complete results from the Clinical Study Report, subject to the confidentiality agreement. When a manuscript is submitted to a biomedical journal, the Sponsor's policy is to also include the protocol and statistical analysis plan to facilitate the peer and editorial review of the manuscript. If the manuscript is subsequently accepted for publication, the Sponsor will allow the journal, if it so desires, to post on its website the key sections of the protocol that are relevant to evaluating the trial, specifically those sections describing the trial objectives and hypotheses, the subject inclusion and exclusion criteria, the trial design and procedures,
Protocol/Amendment No.: 021-09

the efficacy and safety measures, the statistical analysis plan, and any amendments relating to those sections. The Sponsor reserves the right to redact proprietary information.

For multicenter trials, subsequent to the multicenter publication (or after public disclosure of the results online at www.clinicaltrials.gov if a multicenter manuscript is not planned), an investigator and his/her colleagues may publish their data independently. In most cases, publication of individual trial site data does not add value to complete multicenter results, due to statistical concerns. In rare cases, publication of single trial site data prior to the main paper may be of value. Limitations of single trial site observations in a multicenter trial should always be described in such a manuscript.

Authorship credit should be based on 1) substantial contributions to conception and design, or acquisition of data, or analysis and interpretation of data; 2) drafting the article or revising it critically for important intellectual content; and 3) final approval of the version to be published. Authors must meet conditions 1, 2 and 3. Significant contributions to trial execution may also be taken into account to determine authorship, provided that contributions have also been made to all three of the preceding authorship criteria. Although publication planning may begin before conducting the trial, final decisions on authorship and the order of authors' names will be made based on participation and actual contributions to the trial and writing, as discussed above. The first author is responsible for defending the integrity of the data, method(s) of data analysis and the scientific content of the manuscript.

The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

#### 11.0 LIST OF REFERENCES

- 1. Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. Department of Health and Human Services. November 3, 2008; 1-139. Available at <a href="http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL">http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL</a>.
- 2. Consolidated guidelines on the use of antiretroviral drugs for treating and preventing HIV infection recommendations for a public health approach.
- 3. Anderson M, Gilmartin J, Cilissen C, etc., Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of MK-1439, a Novel HIV Non-Nucleoside Reverse Transcriptase Inhibitor, in Healthy Subjects, Abstract presented at Conference on Retroviruses and Opportunistic Infections, March 3 6, 2014, Boston, MA

**Protocol/Amendment No.:** 021-09

4. Gatell1 JM, Morales-Ramirez JO, Hagins DP, Thompson M, Arastéh K, Hoffmann C, Rugina S, Osiyemi O, Erscoiu S, Dretler R, Harvey C, Xu X, Teppler H. 48 week Efficacy and Safety and Early CNS tolerability of Doravirine, a novel NNRTI, with TDF/FTC in ART-Naïve HIV Infected patients. Presented at the Conference on HIV Drug Therapy, Glasgow, Nov. 2 – 6, 2014.

- 5. Miettinen OS, Nurminen M. Comparative analysis of two rates. Statistics in Medicine 1985; 4:213-226.
- 6. Farrington CP, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Statistics in Medicine 1990; 9: 1447-54.
- 7. Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. Biometrika 1934; 26: 404-13.

**Protocol/Amendment No.:** 021-09

## 12.0 APPENDICES

#### 12.1 Code of Conduct for Clinical Trials

#### Merck Sharp & Dohme LLC, Rahway, NJ, USA (MSD) Code of Conduct for Interventional Clinical Trials

#### I. Introduction

#### A. Purpose

MSD, through its subsidiaries, conducts clinical trials worldwide to evaluate the safety and effectiveness of our products. As such, we are committed to designing, implementing, conducting, analyzing, and reporting these trials in compliance with the highest ethical and scientific standards. Protection of participants in clinical trials is the overriding concern in the design and conduct of clinical trials. In all cases, MSD clinical trials will be conducted in compliance with local and/or national regulations (including all applicable data protection laws and regulations), and International Council for Harmonisation Good Clinical Practice (ICH-GCP), and also in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

#### B. Scope

Highest ethical and scientific standards shall be endorsed for all clinical interventional investigations sponsored by MSD irrespective of the party (parties) employed for their execution (e.g., contract research organizations, collaborative research efforts). This Code is not intended to apply to trials that are observational in nature, or which are retrospective. Further, this Code does not apply to investigator-initiated trials, which are not under the full control of MSD.

#### II. Scientific Issues

#### A. Trial Conduct

#### 1. Trial Design

Except for pilot or estimation trials, clinical trial protocols will be hypothesis-driven to assess safety, efficacy and/or pharmacokinetic or pharmacodynamic indices of MSD or comparator products. Alternatively, MSD may conduct outcomes research trials, trials to assess or validate various endpoint measures, or trials to determine patient preferences, etc.

The design (i.e., participant population, duration, statistical power) must be adequate to address the specific purpose of the trial and shall respect the data protection rights of all participants, trial site staff and, where applicable, third parties. All trial protocols are and will be assessed for the need and capability to enroll underrepresented groups. Participants must meet protocol entry criteria to be enrolled in the trial.

#### 2. Site Selection

MSD's clinical trials are conducted globally in many different countries and in diverse populations, including people of varying age, race, ethnicity, gender, and accounting for other potential disease related factors. MSD selects investigative sites based on medical expertise, access to appropriate participants, adequacy of facilities and staff, previous performance in clinical trials, as well as budgetary considerations. Prior to trial initiation, sites are evaluated by MSD personnel (or individuals acting on behalf of MSD) to assess the ability to successfully conduct the trial.

Where appropriate, and in accordance with regulatory authority guidance, MSD will make concerted efforts to raise awareness of clinical trial opportunities in various communities. MSD will seek to engage underrepresented groups and those disproportionately impacted by the disease under study. MSD will support clinical trial investigators to enroll underrepresented groups and expand access to those who will ultimately use the products under investigation.

#### 3. Site Monitoring/Scientific Integrity

Investigative trial sites are monitored to assess compliance with the trial protocol and Good Clinical Practice (GCP). MSD reviews clinical data for accuracy, completeness, and consistency. Data are verified versus source documentation according to standard operating procedures. Per MSD policies and procedures, if potential fraud, scientific/research misconduct, privacy incidents/breaches or Clinical Trial-related Significant Quality Issues are reported, such matters are investigated. When necessary, appropriate corrective and/or preventative actions are defined and regulatory authorities and/or ethics review committees are notified.

#### B. Publication and Authorship

Regardless of trial outcome, MSD commits to publish the primary and secondary results of its registered trials of marketed products in which treatment is assigned, according to the pre-specified plans for data analysis. To the extent scientifically appropriate, MSD seeks to publish the results of other analyses it conducts that are important to patients, physicians, and payers. Some early phase or pilot trials are intended to be hypothesis-generating rather than hypothesis testing; in such cases, publication of results may not be appropriate since the trial may be underpowered and the analyses complicated by statistical issues such as multiplicity.

MSD's policy on authorship is consistent with the recommendations published by the International Committee of Medical Journal Editors (ICMJE). In summary, authorship should reflect significant contribution to the design and conduct of the trial, performance or interpretation of the analysis, and/or writing of the manuscript. All named authors must be able to defend the trial results and conclusions. MSD funding of a trial will be acknowledged in publications.

#### III. Participant Protection

# A. Regulatory Authority and Ethics Committee Review (Institutional Review Board [IRB]/Independent Ethics Committee [IEC])

All protocols and protocol amendments will be submitted by MSD for regulatory authority acceptance/authorization prior to implementation of the trial or amendment, in compliance with local and/or national regulations.

The protocol, protocol amendment(s), informed consent form, investigator's brochure, and other relevant trial documents must be reviewed and approved by an IRB/IEC before being implemented at each site, in compliance with local and/or national regulations. Changes to the protocol that are required urgently to eliminate an immediate hazard and to protect participant safety may be enacted in anticipation of ethics committee approval. MSD will inform regulatory authorities of such new measures to protect participant safety, in compliance with local and/or national regulations.

#### B. Safety

The guiding principle in decision-making in clinical trials is that participant welfare is of primary importance. Potential participants will be informed of the risks and benefits of, as well as alternatives to, trial participation. At a minimum, trial designs will take into account the local standard of care.

All participation in MSD clinical trials is voluntary. Participants enter the trial only after informed consent is obtained. Participants may withdraw from an MSD trial at any time, without any influence on their access to, or receipt of, medical care that may otherwise be available to them.

#### C. Confidentiality

MSD is committed to safeguarding participant confidentiality, to the greatest extent possible, as well as all applicable data protection rights. Unless required by law, only the investigator, Sponsor (or individuals acting on behalf of MSD), ethics committee, and/or regulatory authorities will have access to confidential medical records that might identify the participant by name.

#### D. Genomic Research

Genomic research will only be conducted in accordance with a protocol and informed consent authorized by an ethics committee

#### IV. Financial Considerations

#### A. Payments to Investigators

Clinical trials are time- and labor-intensive. It is MSD's policy to compensate investigators (or the sponsoring institution) in a fair manner for the work performed in support of MSD trials. MSD does not pay incentives to enroll participants in its trials. However, when enrollment is particularly challenging, additional payments may be made to compensate for the time spent in extra recruiting efforts.

MSD does not pay for participant referrals. However, MSD may compensate referring physicians for time spent on chart review and medical evaluation to identify potentially eligible participants.

#### **B.** Clinical Research Funding

Informed consent forms will disclose that the trial is sponsored by MSD, and that the investigator or sponsoring institution is being paid or provided a grant for performing the trial. However, the local ethics committee may wish to alter the wording of the disclosure statement to be consistent with financial practices at that institution. As noted above, all publications resulting from MSD trials will indicate MSD as a source of funding.

**Protocol/Amendment No.:** 021-09

## C. Funding for Travel and Other Requests

Funding of travel by investigators and support staff (e.g., to scientific meetings, investigator meetings, etc.) will be consistent with local guidelines and practices.

## V. Investigator Commitment

Investigators will be expected to review MSD's Code of Conduct as an appendix to the trial protocol, and in signing the protocol, agree to support these ethical and scientific standards.

# 12.2 Collection and Management of Specimens for Future Biomedical Research

#### 1. Definitions

- a. Biomarker: A biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition.<sup>1</sup>
- b. Pharmacogenomics: The investigation of variations of DNA and RNA characteristics as related to drug/vaccine response.<sup>2</sup>
- c. Pharmacogenetics: A subset of pharmacogenomics, pharmacogenetics is the influence of variations in DNA sequence on drug/vaccine response.<sup>2</sup>
- d. DNA: Deoxyribonucleic acid.
- e. RNA: Ribonucleic acid.

## 2. Scope of Future Biomedical Research

The specimens collected in this trial as outlined in Section 7.1.3.8 – Future Biomedical Research will be used to study various causes for how subjects may respond to a drug/vaccine. Future biomedical research specimen(s) will be stored to provide a resource for future trials conducted by MSD focused on the study of biomarkers responsible for how a drug/vaccine enters and is removed by the body, how a drug/vaccine works, other pathways a drug/vaccine may interact with, or other aspects of disease. The specimen(s) may be used for future assay development and/or drug/vaccine development.

It is now well recognized that information obtained from studying and testing clinical specimens offers unique opportunities to enhance our understanding of how individuals respond to drugs/vaccines, enhance our understanding of human disease and ultimately improve public health through development of novel treatments targeted to populations with the greatest need. All specimens will be used by MSD or designees and research will be monitored and reviewed by a committee of our scientists and clinicians.

## 3. Summary of Procedures for Future Biomedical Research

a. Subjects for Enrollment

All subjects enrolled in the clinical trial will be considered for enrollment in future biomedical research.

## b. Informed Consent

Informed consent for specimens (i.e., DNA, RNA, protein, etc.) will be obtained during screening for protocol enrollment from all subjects or legal guardians, at a trial visit by the investigator or his or her designate. Informed consent for Future Biomedical Research should be presented to the subjects on Visit 1. If delayed, present consent at next possible Subject Visit. Informed consent must be obtained prior to collection of all Future Biomedical Research specimens. Consent forms signed by the subject will be kept at the clinical trial site under secure storage for regulatory reasons. Information contained on the consent form alone cannot be traced

Protocol/Amendment No.: 021-09

to any specimens, test results, or medical information once the specimens have been rendered de-identified

A template of each trial site's approved informed consent will be stored in the Sponsor's clinical document repository. Each consent will be assessed for appropriate specimen permissions.

Each informed consent approved by an ethics committee is assigned a unique tracking number. The tracking number on this document will be used to assign specimen permissions for each specimen into the Entrusted Keyholder's Specimen Database.

# c. eCRF Documentation for Future Biomedical Research Specimens

Documentation of participant consent for future biomedical research will be captured in the eCRFs. Any specimens for which such an informed consent cannot be verified will be destroyed.

## d. Future Biomedical Research Specimen Collections

Blood specimens for DNA or RNA isolation will usually be obtained at a time when the subject is having blood drawn for other trial purposes. Specimens like tissue and bone marrow will usually be obtained at a time when the subject is having such a procedure for clinical purposes.

Specimens will be collected and sent to the laboratory designated for the trial where they will be processed (e.g., DNA or RNA extraction, etc) following the MSD approved policies and procedures for specimen handling and preparation.

# 4. Confidential Subject Information for Future Biomedical Research

In order to optimize the research that can be conducted with Future Biomedical Research specimens, it is critical to link subject' clinical information with future test results. In fact little or no research can be conducted without connecting the clinical trial data to the specimen. The clinical data allow specific analyses to be conducted. Knowing subject characteristics like gender, age, medical history and treatment outcomes are critical to understanding clinical context of analytical results.

To maintain privacy of information collected from specimens obtained for Future Biomedical Research, MSD has developed secure policies and procedures. specimens will be de-identified as described below.

At the clinical trial site, unique codes will be placed on the Future Biomedical Research specimens for transfer to the storage facility. This first code is a random number which does not contain any personally identifying information embedded within it. The link (or key) between subject identifiers and this first unique code will be held at the trial site. No personal identifiers will appear on the specimen tube.

This first code will be replaced with a second code at a MSD designated storage/lab facility. The second code is linked to the first code via a second key. The specimen is now double coded. Specimens with the second code are sometimes referred to as deidentified specimens. The use of the second code provides additional confidentiality and


08K3V5

Protocol/Amendment No.: 021-09

privacy protection for subjects over the use of a single code. Access to both keys would be needed to link any data or specimens back to the subject's identification.

The second code is stored separately from the first code and all associated personal specimen identifiers. A secure link, the second key, will be utilized to match the second code to the first code to allow clinical information collected during the course of the trial to be associated with the specimen. This second key will be transferred under secure procedures by the MSD designated facility to an Entrusted Keyholder at MSD. The second code will be logged into the primary biorepository database at MSD and, in this database, this identifier will not have identifying demographic data or identifying clinical information (i.e., race, sex, age, diagnosis, lab values) associated with it. The specimen will be stored in a designated biorepository site with secure policies and procedures for specimen storage and usage.

The second key can be utilized to reconstruct the link between the results of future biomedical research and the clinical information, at the time of analysis. This linkage would not be possible for the scientist conducting the analysis, but can only be done by the MSD Entrusted Keyholder under strict security policies and procedures. The MSD Entrusted Keyholder will link the information and then issue a de-identified data set for analysis. The only other circumstance by which future biomedical research data would be directly linked to the full clinical data set would be those situations mandated by regulatory authorities (e.g., EMEA, FDA), whereby this information would be directly transferred to the regulatory authority.

# 5. Biorepository Specimen Usage

Specimens obtained for the Sponsor will be used for analyses using good scientific practices. Analyses utilizing the future biomedical research specimens may be performed by the Sponsor, or an additional third party (eg, a university investigator) designated by the Sponsor. The investigator conducting the analysis will follow the Sponsor's privacy and confidentiality requirements. Any contracted third party analyses will conform to the specific scope of analysis outlined in future biomedical research protocol and consent. Future biomedical research specimens remaining with the third party after specific analysis is performed will be reported to the Sponsor.

## 6. Withdrawal From Future Biomedical Research

Subjects may withdraw their consent for Future Biomedical Research and have their specimens and all derivatives destroyed. Subjects may withdraw consent at any time by contacting the principal investigator for the main trial. If medical records for the main trial are still available, the investigator will contact MSD using the designated mailbox (clinical.specimen.management@MSD.com) and a form will be provided by MSD to obtain appropriate information to complete specimen withdrawal. Subsequently, the subject's specimens will be removed from the biorepository and be destroyed. A letter will be sent from MSD to the investigator confirming the destruction. It is the responsibility of the investigator to inform the subject of completion of destruction. Any analyses in progress at the time of request for destruction or already performed prior to the request being received by the Sponsor will continue to be used as part of the overall

Confidential

08K3V5

Protocol/Amendment No.: 021-09

research trial data and results. No new analyses would be generated after the request is received.

In the event that the medical records for the main trial are no longer available (e.g., if the investigator is no longer required by regulatory authorities to retain the main trial records) or the specimens have been completely anonymized, there will no longer be a link between the subject's personal information and their specimens. In this situation, the request for specimen destruction can not be processed.

# 7. Retention of Specimens

Future Biomedical Research specimens will be stored in the biorepository for potential analysis for up to 20 years from acquisition. Specimens may be stored for longer if a regulatory or governmental authority has active questions that are being answered. In this special circumstance, specimens will be stored until these questions have been adequately addressed.

Specimens from the trial site will be shipped to a central laboratory and then shipped to the MSD designated biorepository. The specimens will be stored under strict supervision in a limited access facility which operates to assure the integrity of the specimens. Specimens will be destroyed according to MSD policies and procedures and this destruction will be documented in the biorepository database.

## 8. Data Security

Databases containing specimen information and test results are accessible only to the authorized Sponsor representatives and the designated study administrator research personnel and/or collaborators. Database user authentication is highly secure, and is accomplished using network security policies and practices based on international standards to protect against unauthorized access.

## 9. Reporting of Future Biomedical Research Data to Subjects

There is no definitive requirement in either authoritative ethical guidelines or in relevant laws/regulations globally that research results have to be, in all circumstances, returned to the trial participant. Some guidelines advocate a proactive return of data in certain instances. No information obtained from exploratory laboratory studies will be reported to the subject or family, and this information will not be entered into the clinical database maintained by MSD on subjects. Principle reasons not to inform or return results to the subject include: lack of relevance to subject health, limitations of predictive capability, concerns of misinterpretation and absence of good clinical practice standards in exploratory research typically used for diagnostic testing.

If any exploratory results are definitively associated with clinical significance for subjects while the clinical trial is still ongoing, investigators will be contacted with information as to how to offer clinical diagnostic testing (paid for by MSD) to subjects enrolled and will be advised that counseling should be made available for all who choose to participate in this diagnostic testing.

If any exploratory results are definitively associated with clinical significance after completion of a clinical trial, MSD will publish the results without revealing specific

Protocol/Amendment No.: 021-09

subject information, inform all trial sites who participated in the MSD clinical trial and post anonymized results on our website or other accredited website(s) that allow for public access (e.g., disease societies who have primary interest in the results) in order that physicians and patients may pursue clinical diagnostic testing if they wish to do so.

# 10. Gender, Ethnicity and Minorities

Although many diagnoses differ in terms of frequency by ethnic population and gender, every effort will be made to recruit all subjects diagnosed and treated on MSD clinical trials for future biomedical research. When trials with specimens are conducted and subjects identified to serve as controls, every effort will be made to group specimens from subjects and controls to represent the ethnic and gender population representative of the disease under current investigation.

## 11. Risks Versus Benefits of Future Biomedical Research

For future biomedical research, risks to the subject have been minimized. Risks include those associated with venipuncture to obtain the whole blood specimen. This specimen will be obtained at the time of routine blood specimens drawn in the main trial.

MSD has developed strict security, policies and procedures to address subject data privacy concerns. Data privacy risks are largely limited to rare situations involving possible breach of confidentiality. In this highly unlikely situation there is risk that the information, like all medical information, may be misused.

It is necessary for subject-related data (i.e., ethnicity, diagnosis, drug therapy and dosage, age, toxicities, etc.) to be re-associated to double coded specimens at the time of data analysis. These subject data will be kept in a separate, secure MSD database, and all specimens will be stripped of subject identifiers. No information concerning results obtained from future biomedical research will be entered into clinical records, nor will it be released to outside persons or agencies, in any way that could be tied to an individual subject.

## 12. Self-Reported Ethnicity

Subjects who participate in future biomedical research will be asked to provide selfreported ethnicity. Subjects who do not wish to provide this data may still participate in future biomedical research.

## 13. Questions

Any questions related to the future biomedical research should be e-mailed directly to clinical.specimen.management@MSD.com.

## 14. References

- 1. National Cancer Institute: http://www.cancer.gov/dictionary/?searchTxt=biomarker
- 2. International Conference on Harmonization: DEFINITIONS FOR GENOMIC BIOMARKERS, PHARMACOGENOMICS, PHARMACOGENETICS, GENOMIC AND **SAMPLE** CODING **CATEGORIES** E15; http://www.ich.org/LOB/media/MEDIA3383.pdf

02-Nov-2022 Confidential 08K3V5

**Protocol/Amendment No.:** 021-09

12.3 Understanding the Intent, Scope and Public Health Benefits of Exploratory Biomarker Research: A Guide for IRBs/IECs and Investigational Site Staff



08K3V5

This informational brochure is intended for IRBs/IECs and Investigational Site Staff. The brochure addresses issues relevant to specimen collection for biomarker research in the context of pharmaceutical drug and vaccine development.

Developed by The Industry Pharmacogenomics Working Group (I-PWG) www.i-pwg.org

# 1. What is a Biomarker and What is Biomarker Research?

A biomarker is a "characteristic that is objectively measured and evaluated as an indicator of normal biological processes, pathogenic processes, or pharmacologic responses to a therapeutic intervention". !

Biomarker research, including research on pharmacogenomic biomarkers, is a tool used to improve the development of pharmaceuticals and understanding of disease. It involves the analysis of biomolecules (such as DNA, RNA, proteins, and lipids), or other measurements (such as blood pressure or brain images) in relation to clinical endpoints of interest. Biomarker research can be influential across all phases of drug development, from drug discovery and preclinical evaluations to clinical development and post-marketing studies. This brochure focuses on biomarker research involving analysis of biomolecules from biological samples collected in clinical trials. Please refer to I-PWG Pharmacogenomic Informational Brochure<sup>2</sup> and ICH Guidance E153 for additional information specific to pharmacogenomic biomarkers.

# 2. Why is Biomarker Research Important?

#### Importance to Patients and Public Health

Biomarker research is helping to improve our ability to predict, detect, and monitor diseases and improve our understanding of how individuals respond to drugs. This research underlies personalized medicine: a tailored approach to patient treatment based on the molecular analysis of genes, proteins, and metabolites.4 The goal of biomarker research is to aid clinical decision-making toward safer and more efficacious courses of treatment, improved patient outcomes, and overall cost-savings. It also allows for the continued development and availability of drugs that are effective in certain sub-populations when they otherwise might not have been developed due to insufficient efficacy in the broader population.

Recent advances in biomedical technology, including genetic and molecular medicine, have greatly increased the power and precision of analytical tools used in health research and have accelerated the drive toward personalized medicine. In some countries, highly focused initiatives have been created to promote biomarker research (e.g., in the US: www.fda.gov/oc/initiatives/criticalpath/; in the EU: www.imi.europa.eu/index en.html).

#### Importance to Drug Development

Biomarker research is being used by the pharmaceutical industry to streamline the drug development process. Some biomarkers are used as substitutes or "surrogates" for safety or efficacy endpoints in clinical trials particularly where clinical outcomes or events cannot practically or ethically be measured (e.g., cholesterol as a surrogate for cardiovascular disease). By using biomarkers to assess patient response, ineffective drug candidates may be terminated earlier in the development process in favor of more promising drug candidates. Biomarkers are being used to optimize clinical trial designs and outcomes by identifying patient populations that are more likely to respond to a drug therapy or to avoid specific adverse events.

**Protocol/Amendment No.:** 021-09

Biomarker research is also being used to enhance scientific understanding of the mechanisms of both treatment response and disease processes, which can help to identify future targets for drug development. Depending on the clinical endpoints in a clinical trial, biomarker sample collection may either be a required or optional component of the trial. However, both mandatory and optional sample collections are important for drug development.

# Importance of Biomarkers to Regulatory Authorities

Regulatory health authorities are increasingly aware of the benefits of biomarkers and how they may be used for drug approval, clinical trial design, and clinical care. Biomarkers have been used to establish risk:benefit profiles. For example, the FDA has modified the US warfarin (Coumadin®) label to include the analysis of CYP2C9 and VKORC1 genes to guide dosing regimens. Health authorities such as the FDA (USA), EMEA (European Union), MHLW (Japan), and ICH (International) are playing a key role in advancing this scientific field as it applies to pharmaceutical development by creating the regulatory infrastructure to facilitate this research. Numerous regulatory guidances and concept papers have already been issued, many of which are available through www.i-pwg.org. Global regulatory authorities have highlighted the importance of biomarker research and the need for the pharmaceutical industry to take the lead in this arena.3,6-24

# 4. How are Biomarkers Being Used in Drug/Vaccine Development?

Biomarker research is currently being used in drug/vaccine development to:

- Explain variability in response among participants in clinical trials
- Better understand the mechanism of action or metabolism of investigational drugs
- Obtain evidence of pharmacodynamic activity (i.e., how the drug affects the body) at the molecular level
- Address emerging clinical issues such as unexpected adverse events
- Determine eligibility for clinical trials to optimize trial design
- Optimize dosing regimens to minimize adverse reactions and maximize efficacy
- Develop drug-linked diagnostic tests to identify patients who are more likely or less likely to benefit from treatment or who may be at risk of experiencing adverse events
- · Provide better understanding of mechanisms of disease
- Monitor clinical trial participant response to medical interventions

Biomarker research, including research on banked samples, should be recognized as an important public health endeavor for the overall benefit of society, whether by means of advancement of medical science or by development of safer and more effective therapies. Since the value of collected samples may increase over time as scientific discoveries are made, investment in long-term sample repositories is a key component of biomarker research.

2



## 5. Biomarkers are Already a Reality in Health Care

A number of drugs now have biomarker information included in their labels.26 Biomarker tests are already being used in clinical practice to serve various purposes:

Predictive biomarkers (efficacy) - In clinical practice, predictive efficacy biomarkers are used to predict which patients are most likely to respond, or not respond, to a particular drug. Examples include: i) Her2/neu overexpression analysis required for prescribing trastuzumab (Herceptin®) to breast cancer patients, ii) c-kit expression analysis prior to prescribing imatinib mesylate (Gleevec®) to gastrointestinal stromal tumor patients, and iii) KRAS mutational status testing prior to prescribing panitumumab (Vectibix®) or cetuximab (Erbitux®) to metastatic colorectal cancer patients.

Predictive biomarkers (safety) - In clinical practice, predictive safety biomarkers are used to select the proper drug dose or to evaluate the appropriateness of continued therapy in the event of a safety concern. Examples include: i) monitoring of blood potassium levels in patients receiving drospirenone and ethinyl estradiol (Yasmin®) together with daily long-term drug regimens that may increase serum potassium, and ii) prospective HLA-B\*5701 screening to identify those at increased risk for hypersensitivity to abacavir (Ziagen®).

Surrogate biomarkers - In clinical practice, surrogate biomarkers may be used as alternatives to measures such as survival or irreversible morbidity. Surrogate biomarkers are measures that are reasonably likely, based on epidemiologic, therapeutic, pathophysiologic, or other evidence, to predict clinical benefit. Examples include: i) LDL level as a surrogate for risk of cardiovascular diseases in patients taking lipid-lowering agents such as atorvastatin calcium (Lipitor®), ii) blood glucose as a surrogate for clinical outcomes in patients taking anti-diabetic agents, and iii) HIV plasma viral load and CD4 cell counts as surrogates for time-to-clinical-events and overall survival in patients receiving antiretroviral therapy for HIV disease.

Prognostic biomarkers - Biomarkers can also help predict clinical outcomes independent of any treatment modality. Examples of prognostic biomarkers used in clinical practice include: i) CellSearch<sup>TM</sup> to predict progressionfree survival in breast cancer, ii) anti-CCP (cyclic citrullinated protein) for the severity of rheumatoid arthritis, iii) estrogen receptor status for breast cancer, and iv) antidsDNA for the severity of systemic lupus erythematosus.

# 6. Biomarker Samples from Clinical Trials: An Invaluable Resource

Adequate sample sizes and high-quality data from controlled clinical trials are key to advancements in biomarker research. Samples collected in clinical trials create the opportunity for investigation of biomarkers related to specific drugs, drug classes, and disease areas. Clinical drug development programs are therefore an invaluable resource and a unique opportunity for highly productive biomarker research. In addition to conducting independent research, pharmaceutical companies are increasingly contributing to consortia efforts by pooling samples, data, and expertise in an effort to conduct rigorous and efficient biomarker research and to maximize the probability of success. 26-27

# 7. Informed Consent for Collection & Banking of Biomarker Samples

Collection of biological samples in clinical trials must be undertaken with voluntary informed consent of the participant (or legally-acceptable representative). Policies

3

and regulations for legally-appropriate informed consent vary on national, state, and local levels, but are generally based on internationally recognized pillars of ethical conduct for research on human subjects. 28-31

Optional vs. Required Subject Participation Depending on the relevance of biomarker research to a clinical development program at the time of protocol development, the biomarker research may be a core required component of a trial (e.g., key to elucidating the drug mechanism of action or confirming that the drug is interacting with the target) or may be optional (e.g., to gain valuable knowledge that enhances the understanding of diseases and drugs). Informed consent for the collection of biomarker samples may be presented either in the main clinical informed consent form or as a separate informed consent form, with approaches varying somewhat across pharmaceutical companies. The relevance of biomarker research to a clinical development program may change over time as the science evolves. The samples may therefore increase in value after a protocol is developed.

Consent for Future Research Use While it can be a challenge to specify the details of the research that will be conducted in the future. the I-PWG holds the view that future use of samples collected for exploratory biomarker research in clinical trials should be permissible when i) the research is scientifically sound, ii) participants are informed of the scope of the intended future research, even if this is broadly defined (see potential uses in Section 4 above), iii) autonomy is respected by providing the option to consent separately to future use of samples or by providing the option to terminate further use of samples upon request (consent withdrawal / sample destruction), and iv) industry standards for confidentiality protection per Good Clinical Practice guidelines are met.3, 31 Importantly, any research using banked samples should be consistent with the original informed consent, except where otherwise permitted by local law or regulation.

Important elements of informed consent for future use of samples include, but are not limited to:29

The scope of research - Where the scope of the potential future research is broad, participants should be informed of the boundaries of the research. While it may not be possible to describe the exact analytical techniques that will be used, or specific molecules that will be analyzed. it is possible to clearly articulate in reasonable detail the type of research to be conducted and its purpose. Information regarding whether stored samples may be shared with other parties or utilized for commercialization purposes should also be addressed.

Withdrawal of consent / sample destruction - The informed consent form should inform participants of their right to withdraw their consent / request destruction of their samples. This should include the mechanisms for exercising that right and any limitations to exercising that right. For example, participants should be informed that it is not possible to destroy samples that have been anonymized.3 In addition, according to industry standards and regulatory guidance, participants should be informed that data already generated prior to a consent withdrawal request are to be maintained as part of the study data. 38

The duration of storage - The permissible duration of storage may vary according to the nature and uses of the samples and may also vary on national, state, and local levels. The intended duration of storage, including indefinite storage, should be specified.



# Biomarker Sample Collection in Different Countries

Collection of biological samples for biomarker research is straightforward in most jurisdictions. Some countries have specific laws and regulations regarding collection, labeling, storage, export, and/or use of exploratory samples. In addition, some regulations distinguish between DNA and non-DNA samples or between samples used for diagnostic purposes and samples collected for scientific research. Processes for the collection, labeling, storage, export, and/or use of biomarker samples should always adhere to the laws and regulations of the country/region in which those samples are collected.

# Return of Research Results to Study Participants

Policies for the return of biomarker research results to study participants who request them vary among pharmaceutical companies. There are many considerations that pharmaceutical companies weigh when determining their policy regarding the return of biomarker research results to study participants. These include:

- i) the conditions under which biomarker research results were generated (i.e., exploratory research laboratory versus accredited diagnostic laboratory)
- ii) whether the results will have an impact on the medical care of the participant or on a related person, if applicable
- iii) whether genetic counseling is recommended (for genetic results)
- iv) the ability to accurately link the result to the individual from whom the sample was collected
- v) international, national, and local guidelines, policies, legislation, and regulations regarding participants' rights to access data generated on them

Renegar et al. 2006 and Article 29 Data Protection Working Party (an advisory committee to the European Commission on the European Data Protection Directive) have addressed these considerations in detail in relation to pharmacogenomic research data and provided a list of documents addressing the general issue of return of research results. 34-36

# Benefits and Risks Associated with Biomarker Research

#### Benefits

While it may not always directly benefit the study participant who is providing the samples, biomarker research can improve overall understanding of disease and treatment of future patients receiving therapies developed from such research. Patients are now benefiting from retrospective biomarker research conducted on samples collected from clinical trials and stored for exploratory research. One example is the recent label update to the EGFR antibody drugs cetuximab (Erbitux®) and panitumumab (Vectibix®) which highlights the value of KRAS status as a predictive biomarker for treatment of metastatic colorectal cancer with this class of drug.

The humanitarian benefit of human research is recognized by the Nuremberg Code, <sup>28,23</sup> Provided that the degree of risk does not exceed that determined by the humanitarian importance of the problem to be solved, research participants should not be denied the right to contribute to the greater common good. <sup>26,32</sup>

#### Risks

Risks associated with biomarker research are primarily related to the physical aspects of obtaining the sample and to patient privacy concerns.

Physical risks associated with biomarker sample collection in clinical trials can be characterized in two ways: i) negligible additional risk when the biomarker sample is collected as part of a procedure conducted to support

I-PWG

8

Protocol/Amendment No.: 021-09

other core trial objectives, and ii) some added risk where the sampling procedure would otherwise have not been performed as a core component of a trial. Risks are also determined by the invasiveness of the sample collection procedure.

Privacy risks are generally those associated with the inappropriate disclosure and misuse of data. Pharmaceutical companies have policies and procedures for confidentiality protection to minimize this risk for all data collected and generated in clinical trials. These may vary across companies, but are based on industry standards of confidentiality and privacy protection highlighted in the following section. Importantly, privacy risks inherent to biomarker data are no greater than other data collected in a clinical trial.

# 11. Privacy, Confidentiality, and Patient Rights

Maintaining the privacy of study participants and the confidentiality of information relating to them is of paramount concern to industry researchers, regulators, and patients. Good Clinical Practice (GCP), the standard adhered to in pharmaceutical clinical research, is a standard that

"... provides assurance that the data and reported results are credible and accurate, and that the rights, integrity, and confidentiality of trial subjects are protected",

where confidentiality is defined as, "The prevention of disclosure, to other than authorized individuals, of a sponsor's proprietary information or of a subject's identity."

This standard dictates that "the confidentiality of records that could identify subjects should be protected, respecting the privacy and confidentiality rules in accordance with applicable regulatory requirements."

Exploratory biomarker research in pharmaceutical development is commonly conducted in research laboratories that are not accredited to perform diagnostic tests used for healthcare decision-making. Therefore, results from exploratory biomarker research usually are not appropriate for use in making decisions about a trial participant's health. In addition, exploratory research data should not be included as part of a participant's medical record accessible for use by insurance companies. Legislation and policies to protect individuals against discrimination based on genetic information continually evolve based on social, ethical, and legal considerations. Examples of such legislation include the Human Tissue Act 2004 (UK) and the Genetic Information Nondiscrimination Act (GINA) 2008 (USA).36-33

#### 12. Where to Get More Information?

Educational resources related to biomarker and pharmacogenomic research that caters to health care professionals, IRBs/IECs, scientists, and patients are continually being created and are publicly available. Links to many of these resources are available through the I-PWG website: www.i-pwg.org.

#### 13. What is I-PWG?

The Industry Pharmacogenomics Working Group (I-PWG) (formerly the Pharmacogenetics Working Group) is a voluntary association of pharmaceutical companies engaged in pharmacogenomic research. The Group's activities focus on non-competitive educational, informational, ethical, legal, and regulatory topics. The Group provides information and expert opinions on these topics and sponsors educational/ informational programs to promote better understanding of pharmacogenomic and other biomarker research for key stakeholders. The I-PWG interacts with regulatory author-

**Protocol/Amendment No.:** 021-09

ities and policy groups to ensure alignment. More information about the I-PWG is available at: www.i-pwg.org.

## 14. Contributing authors

Monique A. Franc, Teresa Hesley, Feng Hong, Ronenn Roubenoff, Jasjit Sarang, Andrea Tyukody Renninger, Amelia Warner

#### 15. References

- Afkinson AJ, Colbum WA, DeGruttola VG, et al. Biomarkers and surrogate endpoints: Preferred definitions and conceptual framework. Clinical Pharmacology & Therapeutics 2001; 69(3): 89-95. (Accessed at: www.ncbl.nim.nih.gov/pubmed/11240971)
- I PWG Pharmacogenomics Informational Brochure, 2008. (Accessed at: http://www.i-pwg.org/cms/index.php?option=com\_docman&task=doc\_domioad&gd=77&itemid=118)
- ICH E15 Definitions for Genomic Biomarkers, Pharmacogenemics, Pharmacogenetics, Genomic Data and Sample Coding Categories. April 2008. (Accessed at: www.fda.gov/OHRMS/DOCKETS/98ft/FDA-2008-D-0199-gdl.pdf and at: http://www.ich.org/LOB/media/MEDIA3383.pdf)
- Davis JC, Furstenthal L, Desal AA, et al. The microeconomics of personalized medicine: today's challenge and tomorrow's promise. Nature Reviews Drug Discovery, 2009; 8: 279. (Accessed at:http://www.nature.com/nrd/journaliv8/n4/abs/hrd2825.html)
- Bems B, Démoils P, Scheulen ME. How can biomarkers become surrogate endpoints? European Journal of Cancer Supplements 2007; 5: 37-40.
   (Accessed at: www.journalis.eisevierhealth.com/periodicals/ejcsup/issues/ contents?issue\_key=\$1359-6349%2807%29X0031-4)
- Lesko LJ, Woodcock J. Translation of pharmacogenomics and pharmacogenetics: a regulatory perspective. Nature Reviews Drug Discovery, 2004; 3: 763-769. (Accessed at: www.nature.com/mrd/journal/v3/n9/abs/mrd/1499.html)
- Lesko LJ, Woodcock J. Pharmacogenomic-guided drug development: regulatory perspective. The Pharmacogenomics Journal, 2002; 2: 20-24. (Accessed at www.ncbi.nlm.nlh.gov/pubmed/11990376)
- Petricoin EF, Hackett JL, Lesko LJ, et al. Medical applications of microarray technologies: a regulatory science perspective. Nat Genet., 2002; 32: 474-479.

(Accessed at: www.nature.com/ng/journal/v32/n4s/abs/ng1029.html)

- Lesko LJ, Salemo RA, Spear BB, et al. Pharmacogenetics and pharmacogenomics in drug development and regulatory decision making: report of the first FDA-PWG-PhRIMA-DruSafe Workshop. J Clin Pharmacol., 2003; 43: 342-358. (Accessed at: http://jcp.sagepub.com/cgi/content/abstract/43/4/342)
- Salemo RA, Lesko LJ. Pharmacogenomics in Drug Development and Regulatory Decision-making: the Genomic Data Submission (GDS) Proposal. Pharmacogenomics, 2004; 5: 25-30. (Accessed at: www.futuremedicine.com/doi/pdt/10.2217/14622416.5.1.25)
- Frueh FW, Goodsald F, Rudman A, et al. The need for education in pharmacogenomics: a regulatory perspective. The Pharmacogenomics Journal, 2005; 5: 218-220. (Accessed at: www.hature.com/tp/journal/v5/h4/ abs/6500316a.html)
- Genomic Biomarkers Related to Drug Response: Context, Structure and Format of Qualification Submissions. ICH E16 Step 3 draft. (Accessed at: www.emea.europa.eurpdfs/human/lch/35053609endraft.pdf)
- Guiding principles Processing Joint FDA EMEA Voluntary Genomic Data Submissions (VGDSs) within the framework of the Confidentiality Arrangement. May 19, 2006. (Accessed at:

www.fds.gov/downloads/Drugs/Science/Research/Research/Areas/Pharmacogenetics/ucm085378.pdf)

 Guidance for Industry Pharmacogenomic Data Submissions. FDA. March 2005. (Accessed at:

www.tb.gov/downcode/Duge/OuderorComplance/Cogustorynformation/Ouderces/Lon079649.pdf)
15. Pharmacogenomic Data Submissions - Companion Guidance. FDA Draft Guidance. August 2007. (Accessed at:

www.tls.gov/sowicada/Druga/Outlanos/Compleme/Regulator/information/Outlances/unit/1995.pdf)
16. Reflection Paper on Pharmacogenomics in Oncology. EMEA 2008.

www.emea.europa.eu/pdfs/human/pharmacogenetics/12843506endraft.pdf)

- Position paper on Terminology in Pharmacogenetics. EMEA. 2002. (Accessed at: www.emea.europa.eu/pdfs/human/press/pp/307001en.pdf)
- Concept paper on the development of a Guideline on the use of pharmacogenomic methodologies in the pharmacokinetic evaluation of medicinal products. EMEA 2009. (Accessed at:

www.emea.europa.eu/pdfs/human/pharmacogenetics/6327009en.pdf}

 Reflection paper on Pharmacogenomic samples, testing and data handling. EMEA. 2007. (Accessed at:

www.emea.europa.eu/pdfs/human/pharmacogenetics/20191406en.pdf)

- Ishiguro A, Toyoshima S, Uyama Y. Current Japanese regulatory situations of pharmacogenomics in drug administration. Expert Review of Clinical Pharmacology, 2008;1: 505-514. (Accessed at: www.ingentaconnect.com/ contentritdecp/2008/00000001/00000004/art00007)
- 21. Amur S, Frueh FW, Lesko LJ, et al. Integration and use of

I-PWG

8

Protocol/Amendment No.: 021-09

blomarkers in drug development, regulation and clinical practice: A US http://hwetgate.access.gov.gov/cgi-bingetdoc.og/?ibname=115\_cong\_public\_laws6dock=fpub/255.110.pdf) regulatory practice. Biomarkers Med. 2008; 2, 305-311. (Accessed at: 38. Guidance for Sponsors, Clinical Investigators, and IRBs. Data Retention. www.ingentaconnect.com/content/fm/bmm/2008/00000002/00000003/ When Subjects Withdraw from FDA-Requiated Clinical Trials. FDA October 2008. www.fda.gov/OHRMS/DOCKETS/96ft/FDA-2008-D-0576-gdl.pdf art00010?crawler=true) 39. Anderson C, Gomez-Mandilla B, Spear BB, Barnes DM, Cheeseman 22. Mendrick DL, Brazell C, Mansfield EA, et al. Pharmacogenomics and regulatory decision making: an international perspective. The Pharmacogenomics K, Shaw P, Friedman J, McCarthy A, Brazell C, Ray SC, McHale D, Journal, 2006; 6(3), 154-157, (Accessed at: Hashimoto L. Sandbrink R. Watson ML. Salemo RA. on behalf of The www.nature.com/tpi/fournal/v6/n3/abs/6500364a.html) Pharmacogenetics Working Group, Elements of Informed Consent for 23. Pendergast MK. Regulatory agency consideration of pharmacogenomics. Pharmacogenetic Research; Perspective of the Pharmacogenetics Exp Bloi Med (Maywood). 2008; 233:1498-503. (Accessed at: Working Group. Pharmacogenomics Journal 2002;2:284-92. (Accessed at: www.nature.com/tpl/journal/v2/n5/abs/6500131a.html) www.ebmonline.org/cgi/content/abstract/233/12/1498) 24. Goodsald F, Frueh F. Process map proposal for the validation of genomic biomarkers. Pharmacogenomics., 2006; 7(5):773-82 (Accessed at: www.futuremedicine.com/dol/abs/10.2217/14622416.7.5.773) 25. FDA Table of Valid Genomic Biomarkers in the Context of Approved Drug Labels. (Accessed at: www.fda.gov/Drugs/ScienceResearch/ResearchAreas/Pharmacogenetics/ ucm083378.htm) 26. International Serious Adverse Event Consortium. (Accessed at: www.saeconsortium.org) 27. Predictive Safety Testing Consortium. (Appeased at: www.c-path.org/pstc.cfm) 28. Nuremberg code. (Accessed al: http://ohsr.od.nih.gov/guidelines/nuremberg.html) 29. Declaration of Heisinki. (Accessed at: http://ahsr.od.nlh.gov/guidelines/heisinki.html) 30. Belmont report. (Accessed at: http://ohsr.od.nih.gov/guidelines/belmont.html) 31. ICH E6(R1) - Guideline for Good Clinical Practice, June 1995. (Accessed at: www.ich.org/LOB/media/MEDIA482.pdf) 32. Barnes M, Heffernan K. The "Future Uses" Dilemma: Secondary Uses of Data and Materials by Researchers for Commercial Research Sponsors, Medical Research Law & Policy, 2004; 3: 440-450. 33. Eriksson S, Heigesson G. Potential harms, anonymization, and the right to withdraw consent to blobank research. Eur J Hum Genet., 2005; 13:1071-1076. (Accessed at: www.nature.com/ejhg/journal/v13/n9/pdf/5201458a.pdf) 34. Renegar G, Webster CJ, Stuerzebecher S, et al. Returning genetic research results to Individuals: points-to-consider. Bioethics 2006; 20: 24-36. (Accessed at: http://www3.interscience.wiley.com/cgi-bin/fulltext/118562753/PDFSTART) 35. Article 29 Data Protection Working Party. (Accessed at: www.ec.europa.eu/justice home/fsj/privacy/workinggroup/index en.htm) 36. Human Tissue Act 2004 (UK). (Accessed at: www.opsl.gov.uk/acts/acts2004/en/ukpgaen\_20040030\_en\_1) 37. Genetic Information Nondiscrimination Act. (Accessed at: 9

MK-1439A-021-09 Final Protocol 02-Nov-2022 Confidential



# 12.4 Approximate Blood Volumes Drawn/Collected by Trial Visit and by Sample Types

# 12.4.1 Base Study

| Visit Number/Title: | 1 | 2<br>Random-<br>ization | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | U (Virologic<br>Failure<br>Confirmation) | U (Early<br>Discon-<br>tinuation | 99 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen- | | | | | | | | | | | | | | Post | |
| Trial Period | ing | | | 1 | | | atment | | 1 | 1 | 1 | | | | treatment | |
| | | | | | | Fast- | | Fast- | | | | Fast- | | | Post- | |
| | | F .: 2 | 33777 | 33777 | 11777 | inga | 33.77 | inga | 33.77.7 | 33777 | 33717 | inga | >1week after | | study | |
| T 1 D 1 | C | Fastinga | WK | WK | WK | WK | WK | | WK | WK | WK<br>84 | WK | initial virologic | At time | 14-day | |
| Trial Procedures | Screen | Day 1 <sup>a</sup> | 4 | 8 | 16 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | failure | of Discon | follow-up | Total |
| Laboratory<br>Procedures/Assessments | | | | | | | | | | | | | | | | Volume |
| Hematology | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | | 2 | 2 | 28 |
| Serum Pregnancy Test <sup>c</sup> | | | | | | | | | | | | | | _ | _ | |
| Collect Blood for Safety Laboratory | 20 | 70 | _ | _ | _ | 70 | _ | _ | _ | _ | | 70 | 2 5h | - | _ | 100.5 |
| Tests (Chemistry) | 29 | 7ª | 7 | 7 | 1 | 7 <sup>a</sup> | 7 | 7 | 7 | 1 | 7 | 7ª | 3.5 <sup>h</sup> | 7 | 7 | 123.5 |
| HIV/Hepatitis Screen <sup>b</sup> | | | | | | | | | | | | | | | | |
| Hemostatic Function Test <sup>d</sup> | 4.5 | | | | | | | | | | | | | | | 4.5 |
| Virology Test Plasma HIV viral | | | | | | | | | | | | | | | | |
| RNA quantification test (Abbott | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 150 |
| Real Time HIV-1) | | | | | | | | | | | | | | | | |
| Collect Blood for CD4 Cell Count | 2 | 2 | | 2 | | 2 | | 2 | | 2 | | 2 | | | | 14 |
| Collect Blood for MK-1439 PK <sup>e</sup> | | 4 | 4 | 4 | | 8 | | 8 | | | | | | | | 28 |
| Collect Plasma for Viral Resistance | 14 | | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 <sup>g</sup> | | 182 |
| Test | 17 | | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | | | | |
| Collect Blood (DNA) for Genetic<br>Analysis <sup>b</sup> | | 8.5 | | | | | | | | | | | | | | 8.5 |
| Collect Plasma for Future<br>Biomedical Research <sup>b</sup> | | 10 | | | | | | 10 | | | | 10 | | | | 30 |
| Total (mL) | 61.5 | 43.5 | 37 | 39 | 33 | 43 | 33 | 53 | 33 | 35 | 33 | 45 | 27.5 | 33 | 19 | 568.5 |
| Total (tablespoons) | 4.1 | 2.9 | 2.5 | 2.6 | 2.2 | 2.9 | 2.2 | 3.5 | 2.2 | 2.3 | 2.2 | 3.0 | 1.8 | 2.2 | 1.3 | ~37.9 |

| Visit Number/Title: | 1 | 2<br>Random-<br>ization | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | U (Virologic<br>Failure<br>Confirmation) | U (Early<br>Discon-<br>tinuation | 99 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen- | | | | | | | | | | | | | Post | |
| Trial Period | ing | | | | | Tre | atment | , | | | | | | | treatment |
| | | | | | | Fast- | | Fast- | | | | Fast- | | | Post- |
| | | | | | | inga | | inga | | | | inga | >1week after | | study |
| | | Fasting <sup>a</sup> | WK | WK | WK | WK | WK | WK | WK | WK | WK | WK | initial virologic | At time | 14-day |
| Trial Procedures | Screen | Day 1 <sup>a</sup> | 4 | 8 | 16 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | failure | of Discon | follow-up |

a. Fasting is required at these visits for lipids measurement.

- c. For women of childbearing potential.
- d. Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) and International Normalized Ratio (INR).
- e. At Study Day 1 and Study Week 4, sample must be collected predose. At Study Week 12, the sample may be collected irrespective of time of dose. At Study Weeks 24 and 48, samples must be collected predose, and within 0.5 to 2 hours postdose (subjects should remain fasting until postdose PK sample is collected).
- f. One Tablespoon = 15 mL.
- g. If viral failure or relapse is confirmed (with a confirmatory HIV-1 RNA at least one week later), and the decision is made to discontinue the subject, plasma for resistance needs not be collected again at the discontinuation visit.
- h. For creatinine clearance only.

b. Includes Enzyme Immunoassay HIV Antibody Screen, Serum Hepatitis B Surface Antigen, Serum Hepatitis B Surface Antibody, Serum Hepatitis B e-Antigen and Serum Hepatitis C Antibody. A plasma Hepatitis C virus PCR quantitative test (an additional ~6 ml= 0.4 tablespoon of blood) will be performed if the Hepatitis C antibody test is positive.

# 12.4.2 Week 100 Through Week 192 Including Post-Study 14-Day Follow-up (Study Extension 1)

| Week (Visit) | 100<br>(V13) | 116<br>(V14) | 132<br>(V15) | Fasting 148 (V16) <sup>a</sup> | 164<br>(V17) | 180<br>(V18) | Fasting 192 (V19) <sup>a</sup> | Viral Failure<br>Confirmation<br>(U) | Early<br>Discontinuation<br>(U) | Post-Study<br>14-Day<br>Follow-up<br>(99) | Total Vol.<br>in Study<br>Extension 1 <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Hematology | 2 | 2 | 2 | 2 | 2 | 2 | 2 | | 2 | 2 | 18 |
| Collect Blood for CD4<br>Cell Count | 2 | | | 2 | | | 2 | | | | 6 |
| Collect Blood for Safety<br>Laboratory Tests<br>(Chemistry) | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 3.5° | 7 | 7 | 66.5 |
| Virology Test Plasma<br>HIV viral RNA<br>quantification test<br>(Abbott Real Time<br>HIV-1) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 100 |
| Collect Plasma for Viral<br>Resistance | | | | | | | | 14 | 14 <sup>d</sup> | | 28 |
| TOTAL for visit (mL) | 21 | 19 | 19 | 21 | 19 | 19 | 21 | 27.5 | 33 | 19 | 218.5 |
| Total (tablespoons) <sup>e</sup> | 1.4 | 1.3 | 1.3 | 1.4 | 1.3 | 1.3 | 1.4 | 1.8 | 2.2 | 1.2 | ~14.5 |

<sup>&</sup>lt;sup>a</sup> Fasting is required at these visits for lipids measurement.

b These samples are in addition to those collected during the base study. Because an early discontinuation visit could potentially happen during the base study or study extension 1, but not both, and because there is no post-study follow-up visit after the base study for subjects who continue into study extension 1, the total volume for the base study and study extension 1 could be less than the sum.

<sup>&</sup>lt;sup>c</sup> For creatinine clearance only.

d Early Discontinuation Visit sample should be collected only if not done at Viral Failure Confirmation Visit.

e One tablespoon = 15 mL.

**Protocol/Amendment No.:** 021-09

12.5 Plasma Assay—Sample Collection, Handling, Labeling, Storage, and Shipment

See Laboratory Manual.

**Protocol/Amendment No.:** 021-09

# 12.6 List of Preferred Neuropsychiatric Adverse Events

| Category | Active PTs in MedDRA version 17.0 |
|---|---|
| Dizziness | |
| | Dizziness |
| Sleep Disorders and Disturbances | |
| 2.000 2.001 00.00 00.00 | Behavioural insomnia of childhood |
| | Hyposomnia |
| | Initial insomnia |
| | Insomnia |
| | Middle insomnia |
| | Terminal insomnia |
| | Breathing-related sleep disorder |
| | Dyssomnia |
| | Hypnagogic hallucination |
| | Hypnopompic hallucination |
| | Sleep attacks |
| | * |
| | Abnormal dreams |
| | Abnormal sleep-related event Confusional arousal |
| | Loss of dreaming |
| | Nightmare |
| | Parasomnia |
| | Rapid eye movements sleep abnormal |
| | Sleep inertia |
| | Sleep sex |
| | Sleep talking |
| | Sleep terror |
| | Sleep-related eating disorder |
| | Somnambulism |
| | Sleep disorder due to a general medical condition |
| | Sleep disorder due to general medical condition, hypersomnia type |
| | Sleep disorder due to general medical condition, insomnia type |
| | Sleep disorder due to general medical condition, mixed type |
| | Sleep disorder due to general medical condition, parasomnia type |
| | Hypersomnia-bulimia syndrome |
| | Sleep disorder |
| | Sopor |
| | Hypersomnia related to another mental condition |
| | Insomnia related to another mental condition |
| Altered Sensorium | |
| | Altered state of consciousness |
| | Apallic syndrome |
| | Consciousness fluctuating |
| | Depressed level of consciousness |
| | Hyperglycaemic unconsciousness |
| | Lethargy |
| | Loss of consciousness |
| | Neonatal oversedation |
| | Post-injection delirium sedation syndrome |
| | Postictal state |
| | Preictal state |
| | 1 releast state |

| Category | Active PTs in MedDRA version 17.0 |
|---|---|
| | Sedation |
| | Somnolence |
| | Somnolence neonatal |
| | Stupor |
| | Syncope |
| Depression and suicide/self-injury | |
| | Activation syndrome |
| | Adjustment disorder with depressed mood |
| | Adjustment disorder with mixed anxiety and depressed mood |
| | Agitated depression |
| | Anhedonia |
| | Antidepressant therapy |
| | Childhood depression |
| | Decreased interest |
| | Depressed mood |
| | Depression |
| | Depression postoperative |
| | Depressive symptom |
| | Dysphoria |
| | Dysthymic disorder |
| | Electroconvulsive therapy |
| | Feeling guilty |
| | Feeling of despair |
| | Feelings of worthlessness |
| | Major depression |
| | Menopausal depression |
| | Post stroke depression |
| | Postictal depression |
| | Postpartum depression |
| | Completed suicide |
| | Depression suicidal |
| | Intentional overdose |
| | Intentional self-injury |
| | Poisoning deliberate |
| | Self-injurious behaviour |
| | Self-injurious ideation |
| | Suicidal behaviour |
| | Suicidal ideation |
| | Suicide attempt |
| Psychosis and psychotic disorders | Acute psychosis |
| | Alcoholic psychosis |
| | Alice in wonderland syndrome |
| | Brief psychotic disorder with marked stressors |
| | Brief psychotic disorder without marked stressors |
| | Brief psychotic disorder, with postpartum onset |
| | Charles Bonnet syndrome |
| | Childhood psychosis |
| | Clang associations |
| | Cotard's syndrome |
| | Delusion |
| | Delusion of grandeur |

| Category | Active PTs in MedDRA version 17.0 |
|---|---|
| | Delusion of reference |
| | Delusion of replacement |
| | Delusional disorder, erotomanic type |
| | Delusional disorder, grandiose type |
| | Delusional disorder, jealous type |
| | Delusional disorder, mixed type |
| | Delusional disorder, persecutory type |
| | Delusional disorder, somatic type |
| | Delusional disorder, unspecified type |
| | Delusional perception |
| | Delusions, mixed |
| | Dementia of the Alzheimer's type, with delusions |
| | Depressive delusion |
| | Derailment |
| | Epileptic psychosis |
| | Erotomanic delusion |
| | Flight of ideas |
| | Hallucination |
| | Hallucination, auditory |
| | Hallucination, gustatory |
| | Hallucination, olfactory |
| | Hallucination, synaesthetic |
| | Hallucination, tactile |
| | Hallucination, visual |
| | Hallucinations, mixed |
| | Hypnagogic hallucination |
| | Hypnopompic hallucination |
| | Hysterical psychosis |
| | Ideas of reference |
| | Illusion |
| | Jealous delusion |
| | Loose associations |
| | Neologism |
| | Paranoia |
| | Paranoid personality disorder |
| | Parkinson's disease psychosis |
| | Paroxysmal perceptual alteration |
| | Persecutory delusion |
| | Postictal psychosis |
| | Post-injection delirium sedation syndrome |
| | Posturing |
| | Psychosis postoperative |
| | Psychotic behaviour |
| | Psychotic disorder |
| | Psychotic disorder due to a general medical condition |
| | Reactive psychosis |
| | Rebound psychosis |
| | Schizoaffective disorder |
| | Schizoaffective disorder bipolar type |
| | Schizoaffective disorder depressive type Schizoaffective disorder depressive type |
| | Schizophrenia |
| | Бенгоринена |

| Category | Active PTs in MedDRA version 17.0 |
|----------|--------------------------------------|
| | Schizophrenia simple |
| | Schizophrenia, catatonic type |
| | Schizophrenia, disorganised type |
| | Schizophrenia, paranoid type |
| | Schizophrenia, residual type |
| | Schizophrenia, undifferentiated type |
| | Schizophreniform disorder |
| | Schizotypal personality disorder |
| | Senile psychosis |
| | Shared psychotic disorder |
| | Somatic delusion |
| | Somatic hallucination |
| | Substance-induced psychotic disorder |
| | Tangentiality |
| | Thought blocking |
| | Thought broadcasting |
| | Thought insertion |
| | Thought withdrawal |
| | Transient psychosis |
| | Waxy flexibility |

**Protocol/Amendment No.:** 021-09

# 12.7 List of Abbreviations and Acronyms

| Abbreviation | Definition |
|---|---|
| 3TC | Lamivudine |
| AE | Adverse event / adverse experience |
| AIDS | Acquired Immune Deficiency Syndrome |
| ALT | Serum alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| ART | Antiretroviral therapy |
| ASaT | All Subjects as Treated |
| AST | Serum aspartate aminotransferase |
| BLoQ | Below the limit of quantification |
| cART | Combination antiretroviral therapy |
| CCR5 | Chemokine Receptor Type 5 |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval; or (as in section 10.3 only) Coordinating Investigator |
| Cl <sub>cr</sub> | Creatinine Clearance |
| CPT | Child-Pugh Class C score or Pugh-Turcotte |
| CSR | Clinical Study Report |
| CYP | Cytochrome |
| DAIDS | Division of Acquired Immunodeficiency Syndrome |
| DMC | Data Monitoring Committee |
| DNA | Deoxyribonucleic Acid |
| ECG | Electrocardiogram |
| ECI | Event of clinical interest |
| eCRF | Electronic case report form |
| eDMC | External Data Monitoring Committee |
| EFV | Efavirenz |
| EOC | Executive Oversight Committee |
| ERC | Ethical Review Committee |
| EU | European Union |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FDR | Fixed Dose Regimen |
| FTC | Emtricitabine |
| GCP | Good Clinical Practice |
| HAART | Highly Active Antiretroviral Therapy |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HDL-C | High Density Lipoprotein Cholesterol |
| HIV | Human Immunodeficiency Virus |
| HIV-1 | Human Immunodeficiency Virus Type I |
| IB | Investigator Brochure |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| INR | International Normalized Ratio |
| InSTI | Integrase Strand Inhibitors |
| IRB | Institutional Review Board |
| IRIS | Immune Reconstitution Syndrome |
| IUD | Intrauterine Device |
| IVRS/IWRS | Interactive voice response system/Integrated web response system |
| LDL-C | Low-Density Lipoprotein Cholesterol |
| | 20. 2 thong Dipoprotein Choresteror |

| Abbreviation | Definition |
|---|---|
| MedDRA | Medical Dictionary for Regulatory Activities |
| MK-1439 | Doravirine |
| MK-1439A | Doravirine/ Lamivudine/ Tenofovir disoproxil fumarate |
| N(t)RTI | Nucleotide Reverse transcriptase inhibitor |
| NC=F | Non-Completer = Failure |
| NNRTI | Non-Nucleoside Reverse transcriptase inhibitor |
| NRTI | Nucleoside Reverse transcriptase inhibitor |
| OF | Observed Failure |
| PCR | Polymerase Chain Reaction |
| PDLC | Pre-Defined Limit of Change |
| PDVF | Protocol-Defined Virologic Failure |
| PI | Protease Inhibitor |
| PK | Pharmacokinetic |
| PK/PD | Pharmacokinetic/Pharmacodynamic |
| PO | Per os |
| PT | Prothrombin Time |
| q.d. | Once Daily |
| RNA | Ribonucleic acid |
| SAC | Scientific Advisory Committee |
| SAE | Serious adverse event |
| (s)SAP | (supplemental) Statistical Analysis Plan |
| SAP | Statistical Analysis Plan |
| SGOT | serum glutamic-oxaloacetic transaminase |
| SGPT | serum glutamic-pyruvic transaminase |
| SOC | System Organ Class |
| TDF | Tenofovir disoproxil fumarate |
| TDF/FTC | Tenofovir disoproxil fumarate/ Emtricitabine (TRUVADA <sup>TM</sup> ) |
| TLOVR | Time to Loss of Virologic Response |
| U | Unscheduled |
| ULN | Upper Limit of Normal |
| US | United States |
| WPAI | Work Productivity and Activity Impairment Questionnaire |

# 12.8 DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS **VERSION 1.0, DECEMBER, 2004; CLARIFICATION AUGUST 2009**

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| HEMATOLOGY Standard International Units are listed | HEMATOLOGY Standard International Units are listed in italics | | | |
| Absolute CD4+ count – Adult and Pediatric >13 years (HIV NEGATIVE ONLY) | 300 – 400/mm3<br>300 – 400/μL | 200 – 299/mm3<br>200 – 299/μL | 100 – 199/mm3<br>100 – 199/μL | <100/mm <sub>3</sub><br><100/μL |
| Absolute lymphocyte count – Adult and Pediatric >13 years (HIV NEGATIVE ONLY) | 600 – 650/mm3<br>0.600 x 109 – 0.650 x<br>109/L | 500 – 599/mm3<br>0.500 x 109 – 0.599 x<br>109/L | 350 – 499/mm3<br>0.350 x 109 – 0.499 x<br>109/L | <350/mm3<br><0.350 x 109/L |
| <b>Comment:</b> Values in children ≤13 years are not given for the 2 pa | rameters above because t | the absolute counts are var | iable. | |
| Absolute neutrophil count (ANC) | | | | |
| Adult and Pediatric, >7 days | 1,000 – 1,300/mms<br>1.000 x 109 – 1.300 x<br>109/L | 750 – 999/mm3<br>0.750 x 109 – 0.999 x<br>109/L | 500 – 749/mms<br>0.500 x 109 – 0.749 x<br>109/L | <500/mm3<br><0.500 x 109/L |
| Fibrinogen, decreased | 100 – 200 mg/dL<br>1.00 – 2.00 g/L OR<br>0.75 – 0.99 x LLN | 75 – 99 mg/dL<br>0.75 – 0.99 g/L OR<br>0.50 – 0.74 x LLN | 50 – 74 mg/dL<br>0.50 – 0.74 g/L OR<br>0.25 – 0.49 x LLN | <50 mg/dL<br><0.50 g/L OR<br><0.25 x LLN OR<br>Associated with gross bleeding |
| † Use age and sex appropriate values (e.g., bilirubin). | | • | | |

| | LABORATORY | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Hemoglobin (Hgb) | <u> </u> | | | |
| <b>Comment:</b> The Hgb values in mmol/l used conversion factor). For grading lappropriate conversion factor for that | Hgb results obtained by an analytic m | on factor used to convert g/dL to<br>nethod with a conversion factor o | mmol/L has been changed from 0. ther than 0.6206, the result must be | 155 to 0.6206 (the most commonly e converted to g/dL using the |
| Adult and Pediatric ≥57 days<br>(HIV POSITIVE ONLY) | 8.5 – 10.0 g/dL<br>5.24 – 6.23 mmol/L | 7.5 – 8.4 g/dL<br>4.62–5.23 mmol/L | 6.50 – 7.4 g/dL<br>4.03–4.61 mmol/L | <6.5 g/dL<br><4.03 mmol/L |
| Adult and Pediatric ≥57 days<br>(HIV NEGATIVE ONLY) | 10.0 – 10.9 g/dL<br>6.18 – 6.79 mmol/L OR<br>Any decrease 2.5 - 3.4 g/dL<br>1.58 – 2.13 mmol/L | 9.0 – 9.9 g/dL<br>5.55 - 6.17 mmol/L OR<br>Any decrease 3.5 - 4.4 g/dL<br>2.14 – 2.78 mmol/L | 7.0 – 8.9 g/dL<br>4.34 - 5.54 mmol/L OR<br>Any decrease ≥4.5 g/dL<br>>2.79 mmol/L | <7.0 g/dL<br><4.34 mmol/L |
| Comment: The decrease is a decrease | from baseline | | | |
| International Normalized Ratio of prothrombin time (INR) | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.1 – 3.0 x ULN | >3.0 x ULN |
| Methemoglobin | 5.0 – 10.0% | 10.1 – 15.0% | 15.1 – 20.0% | >20.0% |
| Prothrombin Time (PT) | 1.1 – 1.25 x ULN | 1.26 – 1.50 x ULN | 1.51 – 3.00 x ULN | >3.00 x ULN |
| Partial Thromboplastin Time (PTT) | 1.1 – 1.66 x ULN | 1.67 – 2.33 x ULN | 2.34 – 3.00 x ULN | >3.00 x ULN |
| Platelets, decreased | 100,000 – 124,999/mm3<br>100.000 x 109 – 124.999 x 109/L | 50,000 – 99,999/mm3<br>50.000 x 109 – 99.999 x 109/L | 25,000 – 49,999/mm3<br>25.000 x 109 - 49.999 x 109/L | <25,000/mm <sup>3</sup><br><25.000 x 109/L |
| WBC, decreased | 2,000 – 2,500/mm <sup>3</sup><br>2.000 x 109 – 2.500 x 109/L | 1,500 – 1,999/mm3<br>1.500 x 109 – 1.999 x 109/L | 1,000 – 1,499/mm3<br>1.000 x 109 – 1.499 x 109/L | <1,000/mm3<br><1.000 x 109/L |
| * Values are for term infants. Pretern | infants should be assessed using loc | al normal ranges. | · | • |

<sup>†</sup> Use age and sex appropriate values (e.g., bilirubin).

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1 PARAMETER MILD | | | |
| CHEMISTRIES Standard In | ternational Units are | listed in italics | | |
| Acidosis | NA | pH <normal, but="" td="" ≥7.3<=""><td>pH &lt;7.3 without life-threatening consequences</td><td>pH &lt;7.3 with life-threatening consequences</td></normal,> | pH <7.3 without life-threatening consequences | pH <7.3 with life-threatening consequences |
| Albumin, serum, low | 3.0 g/dL – <lln<br>30 g/L – &lt;<i>LLN</i></lln<br> | 2.0 – 2.9 g/dL<br>20 – 29 g/L | <2.0 g/dL<br><20 g/L | NA |
| Alkaline Phosphatase | 1.25 – 2.5 x ULN† | 2.6 – 5.0 x ULN† | 5.1 − 10.0 x ULN† | >10.0 x ULN† |
| Alkalosis | NA | pH >normal, but ≤7.5 | pH >7.5 without life-threatening consequences | pH >7.5 with life-threatening consequences |
| ALT (SGPT) | 1.25 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10.0 x ULN | >10.0 x ULN |
| AST (SGOT) | 1.25 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10.0 x ULN | >10.0 x ULN |
| Bicarbonate, serum, low | 16.0 mEq/L - <lln<br>16.0 mmol/L - <lln< td=""><td>11.0 – 15.9 mEq/L<br/>11.0 – 15.9 mmol/L</td><td>8.0 – 10.9 mEq/L<br/>8.0 – 10.9 mmol/L</td><td>&lt;8.0 mEq/L<br/>&lt;<i>8.0 mmol/L</i></td></lln<></lln<br> | 11.0 – 15.9 mEq/L<br>11.0 – 15.9 mmol/L | 8.0 – 10.9 mEq/L<br>8.0 – 10.9 mmol/L | <8.0 mEq/L<br>< <i>8.0 mmol/L</i> |
| <b>Comment:</b> Some laboratories will according to the ranges for Bicarb | • | arbonate (HCO3) and other | ers as Total Carbon Dioxide (CO <sub>2</sub> ). These are the | same tests; values should be graded |
| Bilirubin (Total) | | | | |
| Adult and Pediatric >14 days | 1.1 – 1.5 x ULN | 1.6 – 2.5 x ULN | 2.6 – 5.0 x ULN | >5.0 x ULN |
| Calcium, serum, high | | | | |
| Adult and Pediatric ≥7 days | 10.6 – 11.5 mg/dL<br>2.65 – 2.88 mmol/L | 11.6 – 12.5 mg/dL<br>2.89 – 3.13 mmol/L | 12.6 – 13.5 mg/dL<br>3.14 – 3.38 mmol/L | >13.5 mg/dL<br>>3.38 mmol/L |
| Calcium, serum, low | | | | |
| Adult and Pediatric ≥7 days | 7.8 – 8.4 mg/dL<br>1.95 – 2.10 mmol/L | 7.0 – 7.7 mg/dL<br>1.75 – 1.94 mmol/L | 6.1 – 6.9 mg/dL<br>1.53 – 1.74 mmol/L | <6.1 mg/dL<br><1.53 mmol/L |
| Comment: Do not adjust Calcium | n, serum, low or Calciun | n, serum, high for albumin | 1 | |
| † Use age and sex appropriate va | lues (e.g., bilirubin). | | | |

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Cardiac troponin I (cTnI) | NA | NA | NA | Levels consistent with myocardial infarction or unstable angina as defined by the manufacturer |
| Cardiac troponin T (cTnT) | NA | NA | NA | $\geq$ 0.20 ng/mL OR Levels consistent with myocardial infarction or unstable angina as defined by the manufacturer |
| Cholesterol (fasting) | | | | |
| Adult ≥18 years | 200 – 239 mg/dL<br>5.18- 6.19 mmol/L | 240 – 300 mg/dL<br>6.20 - 7.77 mmol/L | >300 mg/dL<br>>7.77 mmol/L | NA |
| Pediatric <18 years | 170 – 199 mg/dL<br>4.40 - 5.15 mmol/L | 200 – 300 mg/dL<br>5.16 - 7.77 mmol/L | >300 mg/dL<br>>7.77 mmol/L | NA |
| Creatine Kinase | 3.0 - 5.9 x ULN† | 6.0 – 9.9 x ULN† | 10.0 - 19.9 x ULN† | ≥ 20.0 x ULN† |
| Creatinine | 1.1 – 1.3 x ULN† | 1.4 – 1.8 x ULN† | 1.9 – 3.4 x ULN† | ≥ 3.5 x ULN† |

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Glucose, serum, high | | | | |
| Nonfasting | 116 – 160 mg/dL<br>6.44 – 8.88 mmol/L | 161 – 250 mg/dL<br>8.89 – 13.88 mmol/L | 251 – 500 mg/dL<br>13.89 – 27.75 mmol/L | >500 mg/dL<br>>27.75 mmol/L |
| Fasting | 110 – 125 mg/dL<br>6.11 – 6.94 mmol/L | 126 – 250 mg/dL<br>6.95 – 13.88 mmol/L | 251 – 500 mg/dL<br>13.89 – 27.75 mmol/L | >500 mg/dL<br>>27.75 mmol/L |
| Glucose, serum, low | | | | |
| Adult and Pediatric ≥1 month | 55 – 64 mg/dL<br>3.05 – 3.55 mmol/L | 40 – 54 mg/dL<br>2.22 – 3.06 mmol/L | 30 – 39 mg/dL<br>1.67 – 2.23 mmol/L | <30 mg/dL<br><1.67 mmol/L |
| Infant*†, <1 month | 50 – 54 mg/dL<br>2.78 – 3.00 mmol/L | 40 – 49 mg/dL<br>2.22 – 2.77 mmol/L | 30 – 39 mg/dL<br>1.67 – 2.21 mmol/L | <30 mg/dL<br><1.67 mmol/L |
| Lactate | ULN - <2.0 x ULN without acidosis | ≥2.0 x ULN without acidosis | Increased lactate with pH <7.3 without life-threatening consequences | Increased lactate with pH <7.3 with life-threatening consequences |
| Comment: Added ULN to Grade | Comment: Added ULN to Grade 1 parameter | | | |
| LDL cholesterol (fasting) | | | | |
| Adult ≥18 years | 130 – 159 mg/dL<br>3.37 – 4.12 mmol/L | 160 – 190 mg/dL<br>4.13 – 4.90 mmol/L | ≥190 mg/dL<br>≥4.91 mmol/L | NA |
| Pediatric >2 - <18 years | 110 – 129 mg/dL<br>2.85 – 3.34 mmol/L | 130 – 189 mg/dL<br>3.35 – 4.90 mmol/L | ≥190 mg/dL<br>≥4.91 mmol/L | NA |
| Lipase | 1.1 – 1.5 x ULN | 1.6 – 3.0 x ULN | 3.1 – 5.0 x ULN | >5.0 x ULN |
| Magnesium, serum, low | 1.2 – 1.4 mEq/L<br>0.60 – 0.70 mmol/L | 0.9 – 1.1 mEq/L<br>0.45 – 0.59 mmol/L | 0.6 – 0.8 mEq/L<br>0.30 – 0.44 mmol/L | <0.60 mEq/L<br><0.30 mmol/L |
| Pancreatic amylase | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.1 – 5.0 x ULN | >5.0 x ULN |

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Phosphate, serum, low | | | | · |
| Adult and Pediatric >14 years | 2.5 mg/dL – <lln< td=""><td>2.0 – 2.4 mg/dL</td><td>1.0 – 1.9 mg/dL</td><td>&lt;1.00 mg/dL</td></lln<> | 2.0 – 2.4 mg/dL | 1.0 – 1.9 mg/dL | <1.00 mg/dL |
| | 0.81 mmol/L – <lln< td=""><td>0.65 – 0.80 mmol/L</td><td>0.32 – 0.64 mmol/L</td><td>&lt;0.32 mmol/L</td></lln<> | 0.65 – 0.80 mmol/L | 0.32 – 0.64 mmol/L | <0.32 mmol/L |
| Pediatric 1 year – 14 years | 3.0 – 3.5 mg/dL | 2.5 – 2.9 mg/dL | 1.5 – 2.4 mg/dL | <1.50 mg/dL |
| | 0.97 – 1.13 mmol/L | 0.81 – 0.96 mmol/L | 0.48 – 0.80 mmol/L | <0.48 mmol/L |
| Pediatric <1 year | 3.5 – 4.5 mg/dL | 2.5 – 3.4 mg/dL | 1.5 – 2.4 mg/dL | <1.50 mg/dL |
| | 1.13 – 1.45 mmol/L | 0.81 – 1.12 mmol/L | 0.48 – 0.80 mmol/L | <0.48 mmol/L |
| Potassium, serum, high | 5.6 – 6.0 mEq/L | 6.1 – 6.5 mEq/L | 6.6 – 7.0 mEq/L | >7.0 mEq/L |
| | 5.6 – 6.0 mmol/L | 6.1 – 6.5 mmol/L | 6.6 – 7.0 mmol/L | >7.0 mmol/L |
| Potassium, serum, low | 3.0 – 3.4 mEq/L | 2.5 – 2.9 mEq/L | 2.0 – 2.4 mEq/L | <2.0 mEq/L |
| | 3.0 – 3.4 mmol/L | 2.5 – 2.9 mmol/L | 2.0 – 2.4 mmol/L | <2.0 mmol/L |
| Sodium, serum, high | 146 – 150 mEq/L | 151 – 154 mEq/L | 155 – 159 mEq/L | ≥160 mEq/L |
| | 146 – 150 mmol/L | 151 – 154 mmol/L | 155 – 159 mmol/L | ≥160 mmol/L |
| Sodium, serum, low | 130 – 135 mEq/L<br>130 – 135 mmol/L | 125 – 129 mEq/L<br>125 – 129 mmol/L | 121 – 124 mEq/L<br>121 – 124 mmol/L | $\leq$ 120 mEq/L $\leq$ 120 mmol/L |
| Triglycerides (fasting) | NA | 500 – 750 mg/dL<br>5.65 – 8.48 mmol/L | 751 – 1,200 mg/dL<br>8.49 – 13.56 mmol/L | >1,200 mg/dL<br>>13.56 mmol/L |
| † Use age and sex appropriate va | lues (e.g., bilirubin). | 5.65 – 8.48 mmol/L | 8.49 – 13.56 mmol/L | >13.56 mmol/L |

**Protocol/Amendment No.:** 021-09

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Uric acid | 7.5 – 10.0 mg/dL<br>0.45 – 0.59 mmol/L | 10.1 – 12.0 mg/dL<br>0.60 – 0.71 mmol/L | 12.1 – 15.0 mg/dL<br>0.72 – 0.89 mmol/L | >15.0 mg/dL<br>>0.89 mmol/L |
| URINALYSIS Standard International & | URINALYSIS Standard International Units are listed in italics | | | |
| Hematuria (microscopie) | 6 – 10 Red Blood Cell/HPF | >10 RBC/HPF | Gross, with or without clots OR with RBC casts | Transfusion indicated |
| Proteinuria, random collection | 1+ | 2-3+ | 4+ | NA |
| Proteinuria, 24 hour collection | | | | |
| Adult and Pediatric ≥ 10 years | 200 – 999 mg/24 h<br>0.200 – 0.999 g/d | 1,000 - 1,999 mg/24 h<br>1.000 – 1.999 g/d | 2,000 – 3,500 mg/24 h<br>2.000 – 3.500 g/d | >3,500 mg/24 h<br>>3.500 g/d |
| Pediatric >3 mo - <10 years | 201 - 499 mg/m2/24 h<br>0.201 – 0.499 g/d | 500 - 799 mg/m2/24 h<br>0.500 - 0.799 g/d | 800 – 1,000 mg/m2/24 h<br>0.800 – 1.000 g/d | >1,000 mg/ m2/24 h<br>>1.000 g/d |
| † Use age and sex appropriate values (e.g | g., bilirubin). | | | |

Adapted from DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS, PUBLISH DATE: 28 Dec-04/Clarification Aug 09 DECEMBER.

Protocol/Amendment No.: 021-09

#### 13.0 SIGNATURES

## 13.1 Sponsor's Representative

| TYPED NAME |
|-------------|
| TITLE |
| SIGNATURE |
| DATE SIGNED |

# 13.2 Investigator

I agree to conduct this clinical trial in accordance with the design outlined in this protocol and to abide by all provisions of this protocol (including other manuals and documents referenced from this protocol). I agree to conduct the trial in accordance with generally accepted standards of Good Clinical Practice. I also agree to report all information or data in accordance with the protocol and, in particular, I agree to report any serious adverse events as defined in Section 7.0 – Assessing and Recording Adverse Events. I also agree to handle all clinical supplies provided by the Sponsor and collect and handle all clinical specimens in accordance with the protocol. I understand that information that identifies me will be used and disclosed as described in the protocol, and that such information may be transferred to countries that do not have laws protecting such information. Since the information in this protocol and the referenced Investigator's Brochure is confidential, I understand that its disclosure to any third parties, other than those involved in approval, supervision, or conduct of the trial is prohibited. I will ensure that the necessary precautions are taken to protect such information from loss, inadvertent disclosure or access by third parties.

| TYPED NAME |
|-------------|
| TITLE |
| SIGNATURE |
| DATE SIGNED |